Version Date: August 1, 2025

**To:** CTEP Protocol and Information Office

From: Adel Mandl, MD

**Date:** August 1, 2025

**Protocol:** 10315 A Phase 2 Study of XL184 (Cabozantinib) in Combination with Nivolumab

and Ipilimumab for the Treatment of Poorly Differentiated Neuroendocrine

Carcinomas

**Re:** Amendment #8 to address PIO's comment from their review of amendment 7.

## **SUMMARY OF CHANGES – Protocol**

# I. Comments Requiring a Response – Major Issues:

| # | Section | Comments |
|---|---|---|
| 1. | 1.2.5,<br>1.2.6, | This amendment (A07) included edits to remove the biomarker-related objectives from the protocol. Please remove the related language in the listed sections. |
| | 1.3, 5.8,<br>5.9,<br>9.4.5 | Instead, it is suggested to report the following for each relevant objective to ClinicalTrials.gov: |
| | 9.4.5 | The number of patients with data collected for this outcome measure is zero: <i>insert objective</i> . <i>Insert reason</i> . Accordingly, no results will be reported. |
| | | Example reason - This biomarker assay was not performed as there were insufficient samples available to interpret the planned correlative studies |
| | | PI Response: Comments related to removing some of the correlative objectives have been removed. Corrected subsection numbering within section 5.9. |

## **SUMMARY OF CHANGES – Consent Form**

| # | Section | Comments |
|----|---------|--------------------------------|
| 1. | Header | Updated Protocol Version Date. |


**To:** CTEP Protocol and Information Office

From: Adel Mandl, MD

**Date:** June 3, 2025

**Protocol:** 10315 A Phase 2 Study of XL184 (Cabozantinib) in Combination with Nivolumab

and Ipilimumab for the Treatment of Poorly Differentiated Neuroendocrine

Carcinomas

**Re:** Amendment to address PIO's recommendations from their review of

amendment 6, replace the Study PI, and update the objectives and correlatives

that the NCI has determined will not be performed.

### **SUMMARY OF CHANGES - Protocol**

## **I.** Recommendations from PIO's review of Amendment 6:

| # | Section | Comments |
|---|---|---|
| 2. | Cover Page | Please revise the excerpt below as indicated. |
| | | LAO-PA015 / UPMC Hillman University of Pittsburgh Cancer Center Institute LAO |
| | | PI Response: This site has been updated. |
| 3. | Page 2 of cover page | Please delete IND #: on page 2 of cover page and replace with IND #: |
| | | PI Response: The IND number has been updated. |
| 4. | <u>8.1.1</u> | Please replace the Storage with the following: |
| | | <b>Storage:</b> Store intact bottles at controlled room temperature 20 <sup>o</sup> C to 25 <sup>o</sup> C (68 <sup>o</sup> F to 77 <sup>o</sup> F); temperature excursions are permitted between 15 <sup>o</sup> C and 30 <sup>o</sup> C (59 <sup>o</sup> F to 86 <sup>o</sup> F) [see USP Controlled Room Temperature]. |
| | | If a storage temperature excursion outside of 15°C and 30°C (59°F to 86°F) is identified, promptly return XL184 (Cabozantinib) to 20° to 25°C (68° to 77°F) and quarantine the supplies. Provide a detailed report of the excursion (including documentation of temperature monitoring and duration of the excursion) to <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> for determination of suitability. |
| | | PI Response: This information has been updated. |


| # | Section | Comments |
|---|---|---|
| 5. | 8.1.1 | Please replace the <u>Stability</u> with the following: |
| | | <b>Stability:</b> Refer to the drug label for expiration date. Dispense XL184 (Cabozantinib) in original bottles. |
| | | However, if dispensing the exact quantity of cabozantinib tablets is an institutional guideline: |
| | | <ul> <li>Removing the extra tablets from the original bottle is allowed, and it must be used within 30 days of the preparation date. Document the extra tablets as waste in Oral DARF.</li> <li>Adding additional cabozantinib tablets into the original bottle in which the original bottle is exceeding its 30 Count bottle, is Not Allowed.</li> </ul> |
| | | Repackaging XL184 (Cabozantinib) for a short period of time is acceptable and limited to: |
| | | <ul> <li>Up to 24 hours when dispensed in an open container such as a pill cup.</li> <li>Up to 7 days when dispensed in a closed container (e.g., a pharmacy dispensing bottle).</li> </ul> |
| | | PI Response: This information has been updated. |

# II. Requested changes by the PI

| # | Section | Comments |
|---|---|---|
| 6. | Header, | Update protocol version date. |
| | Title Page | |
| 7. | Title Page | Removed Dr. Tesfaye as Study PI since he is no longer affiliated as a CTEP investigator. Adding Dr. Mandl as the Study PI. |
| | | Removed Dr. Chen as the Translational PI. Funds were not established for his work and then the study closed early for futility. |
| 8. | 1.2.5, 1.2.6,<br>1.3, 5.8, 5.9.1,<br>5.9.2, 5.10.1,<br>5.10.2, 5.10.3,<br>5.10.4, 9.4.5 | After discussion with the NCI in April 2025, it was agreed to remove WES and RNAseq as secondary objectives and all exploratory correlative analyses. The study closed early due to futility and as a result there are insufficient samples to provide meaningful interpretation of the data. |
| 9. | 3.3 | Per the Executive Order, the use of 'gender' has been removed. |


# **SUMMARY OF CHANGES – Consent Form**

| # | Section | Comments |
|----|---------|--------------------------------|
| 2. | Header | Updated Protocol Version Date. |


NCI Protocol #: P10315

**Local Protocol #:** TBD

ClinicalTrials.gov Identifier: NCT04079712

**TITLE:** A Phase 2 Study of XL184 (Cabozantinib) in Combination with Nivolumab and Ipilimumab for the Treatment of Poorly Differentiated Neuroendocrine Carcinomas

Corresponding Organization: LAO-MD017 / JHU Sidney Kimmel Comprehensive Cancer

Center LAO

## **Principal Investigator:**

Adel Mandl, MD Johns Hopkins University 201 N. Broadway Street, Viragh, Box 7 Baltimore, MD 21287 410-955-8827 amandl1@jhu.edu

# **Participating Organizations**

| LAO-11030 / University Health Network Princess Margaret Cancer Center LAO |
|---------------------------------------------------------------------------|
| LAO-CA043 / City of Hope Comprehensive Cancer Center LAO |
| LAO-CT018 / Yale University Cancer Center LAO |
| LAO-MA036 / Dana-Farber - Harvard Cancer Center LAO |
| LAO-MD017 / JHU Sidney Kimmel Comprehensive Cancer Center LAO |
| LAO-OH007 / Ohio State University Comprehensive Cancer Center LAO |
| LAO-PA015 / UPMC Hillman Cancer Center LAO |
| LAO-TX035 / University of Texas MD Anderson Cancer Center LAO |
| LAO-NCI / National Cancer Institute LAO |

### Statistician:

Ruizhe Chen, PhD Johns Hopkins University 550 N. Broadway Street, Suite 1103 Baltimore, MD 21205

Phone: 410-955-4884 Email: rzchen@jhu.edu

### **Study Contact:**

Judy Murray, CCRC Johns Hopkins University 201 N. Broadway Street, Viragh, Box 1 Baltimore, MD 21287

Phone: 443-927-3568 Email: jmurra33@jhmi.edu


NCI-Supplied Agents: XL184 (Cabozantinib) (NSC761968)

Nivolumab (BMS-936558, MDX-1106) (NSC748726) Ipilimumab (BMS-734016, MDX-010) (NSC732442)

IND #:

IND Sponsor: DCTD, NCI

### **Protocol Type / Version # / Version Date:**

Original / May 1, 2019

Revision 1 / July 22, 2019

Revision 2 / August 15, 2019

Revision 3a / September 30, 2019

Revision 4 / October 18, 2019

Revision 5 / September 4, 2020

Revision 6 / September 18, 2020

Revision 7 / October 20, 2020 (CIRB Approved, CTEP Disapproved)

Revision 8 / February 22, 2021

Amendment 4 / August 23, 2024

Amendment 5 / November 5, 2024 RRA

Amendment 6 / November 25, 2024

Amendment 7 / June 3, 2025 Disapproved

Amendment 8 / August 1, 2025


### **SCHEMA**

This study is a multicenter phase 2 study of XL184 (cabozantinib) in combination with nivolumab and ipilimumab in patients with advanced/metastatic poorly differentiated neuroendocrine neoplasms after the failure of at least one line of systemic cancer treatment.

| Regimen Description | | | | | | |
|---|---|---|---|---|---|---|
| Cycles | Agent | Premedications; Precautions | Dose | Route | Schedule | Cycle<br>Length |
| | XL184<br>(cabozantinib) | XL184 (cabozantinib) should be taken on an empty stomach. Patients should not eat for at least 2 hours before, and 1 hour after each dose. | 40 mg | PO | Days 1-21 | 21 days |
| 1-4 | Nivolumab | N/A | 3 mg/kg | IV | Day 1 of Cycles<br>1-4<br>(4 total doses) | (3 weeks) |
| | Ipilimumab | N/A | 1 mg/kg | IV | Day 1 of Cycles<br>1-4<br>(4 total doses) | |
| 5+ | XL184<br>(cabozantinib) | XL184 (cabozantinib) should be taken on an empty stomach. Patients should not eat for at least 2 hours before, and 1 hour after each dose. | 40 mg | РО | Days 1-28 | 28 days<br>(4 weeks) |
| | Nivolumab | N/A | 480 mg | IV | Day 1of Cycles<br>5+ | |

PO = Oral: IV = Intravenous

Treatment will be continued until criteria for removal from the study are met (See Section 6.5 Duration of Therapy)

Treatment will be given on an outpatient basis and includes continuous daily administration of XL184 (cabozantinib) 40 mg by mouth (PO). Nivolumab will be given at a dose of 3 mg/kg on Day 1 (±3 days) of each 3-week cycle for the first 4 cycles (12 weeks). Ipilimumab is to be administered at a dose of 1 mg/kg immediately following nivolumab administration on Day 1 of each 3-week cycle for the first 4 cycles. No more than four doses of ipilimumab should be administered.

Starting Cycle 5, patients will continue to take cabozantinib 40 mg PO daily and receive IV infusion of nivolumab 480 mg every 4 weeks. Treatment will be continued until criteria for removal from the study is met.

# TABLE OF CONTENTS

| SCH | EMA | | 2 |
|---|---|---|---|
| 1. | OBJE | ECTIVES | 6 |
| | 1.1 | Primary Objectives | |
| | 1.2 | Secondary Objectives | |
| | 1.3 | Exploratory Objectives | |
| 2. | BAC | KGROUND | 7 |
| | 2.1 | Study Disease | 7 |
| | 2.2 | CTEP IND Agents | 9 |
| | 2.3 | Rationale | 23 |
| | 2.4 | Correlative Studies Background | 24 |
| 3. | PATI | ENT SELECTION | 27 |
| | 3.1 | Eligibility Criteria | 27 |
| | 3.2 | Exclusion Criteria | 29 |
| | 3.3 | Inclusion of Women and Minorities | 33 |
| 4. | REGISTRATION PROCEDURES | | |
| | 4.1 | Investigator and Research Associate Registration with CTEP | |
| | 4.2 | Site Registration | 35 |
| | 4.3 | Patient Registration | 37 |
| | 4.4 | General Guidelines | 39 |
| 5. | BION | MARKER, CORRELATIVE, AND SPECIAL STUDIES | |
| | 5.1 | Summary Table for Specimen Collection. | |
| | 5.2 | Summary Table(s) for Interventional Radiologist for Research Biopsies | 40 |
| | 5.3 | Specimen Procurement Kits and Scheduling | 41 |
| | 5.4 | Specimen Tracking System Instructions | 42 |
| | 5.5 | Specimen Collection | |
| | 5.6 | Shipping Specimens from Clinical Site to the ETCTN Biorepository | |
| | 5.7 | Shipping of Specimens from Clinical Site to Other Laboratories | 48 |
| | 5.8 | Biomarker Plan | |
| | 5.9 | Integrated Correlative Studies | 51 |
| | 5.10 | Exploratory/Ancillary Correlative Studies | 52 |
| 6. | TREA | TREATMENT PLAN | |
| | 6.1 | Agent Administration | 55 |
| | 6.2 | General Concomitant Medication and Supportive Care Guidelines | 57 |
| | 6.3 | Duration of Therapy | |
| | 6.4 | Duration of Follow-Up | |
| 7. | DOSI | ING DELAYS/DOSE MODIFICATIONS | 61 |
| | 7.1 | XL184 (Cabozantinib) | 61 |

| | 7.2 | Nivolumab and Ipilimumab | 79 |
|---|---|---|---|
| 8. | PHARMACEUTICAL INFORMATION | | |
| • | 8.1 | CTEP IND Agents | |
| 9. | STATISTICAL CONSIDERATIONS | | |
| | 9.1 | Study Design/Endpoints | 102 |
| | 9.2 | Sample Size/Accrual Rate | |
| | 9.3 | | |
| | 9.4 | | |
| | 9.5 | Reporting and Exclusions | 106 |
| 10. | | ERSE EVENTS: LIST AND REPORTING REQUIREMENTS | |
| | 10.1 | Comprehensive Adverse Events and Potential Risks Lists (CAEPRs) | |
| | 10.2 | Adverse Event Characteristics | |
| | 10.3 | Expedited Adverse Event Reporting | |
| | 10.4 | Routine Adverse Event Reporting | |
| | 10.5 | Pregnancy | |
| | 10.6 | Secondary Malignancy | |
| | 10.7 | Second Malignancy | 127 |
| 11. | STUI | DY CALENDAR | 128 |
| 12. | MEASUREMENT OF EFFECT | | |
| | 12.1 | | |
| | 12.2 | Other Response Parameters | 137 |
| 13. | | STUDY OVERSIGHT AND DATA REPORTING / REGULATORY | |
| | REQU | JIREMENTS | |
| | 13.1 | Study Oversight | |
| | 13.2 | Data Reporting | |
| | 13.3 | Data Quality Portal | |
| | 13.4 | CTEP Multicenter Guidelines | |
| | | 13.5 Collaborative Agreements Language | |
| | | 13.6 Genomic Data Sharing Plan | |
| | 13.7 | Incidental/Secondary Findings Disclosure Procedure Error! Book defined. | mark not |
| 14. | REFE | RENCES | 144 |
| APPI | ENDIX . | A PERFORMANCE STATUS CRITERIA | 151 |
| APPI | ENDIX | | 1.50 |
| | SEKU | JM CREATININE | |
| APPI | ENDIX | C PATIENT CLINICAL TRIAL WALLET CARD | 153 |
| A PPI | ENDIX | D PRE-BIOPSY ASSESSMENT | 154 |

| NCI Protocol #: 10315<br>Version Date: August 1, 2025 | | |
|---|---|---|
| APPENDIX E | PATIENT MEDICATION DIARY | 155 |
| ALGORITHN<br>HEPATIC, N | NIVOLUMAB AND IPILIMUMAB MANAGEMENT<br>MS FOR ENDOCRINOPATHY, GASTROINTESTINAL,<br>EUROLOGICAL, PULMONARY, RENAL, AND SKIN<br>VEN <b>ts</b> | 158 |


#### 1. OBJECTIVES

### 1.1 Primary Objectives

1.1.1 To evaluate the overall response rate (ORR) associated with the combination of XL184 (cabozantinib), nivolumab, and ipilimumab in patients with advanced poorly-differentiated neuroendocrine carcinomas (NECs), after the failure of at least one line of prior therapy.

## 1.2 Secondary Objectives

- 1.2.1 To evaluate progression-free survival (PFS).
- 1.2.2 To measure the safety and tolerability of the combination of XL184 (cabozantinib), nivolumab, and ipilimumab in patients with advanced, poorly-differentiated NECs.
- 1.2.3 To evaluate disease control rate (DCR).
- 1.2.4 To measure duration of response (DOR).
- 1.2.5 To describe the tumor molecular profile using whole exome sequencing (WES) and correlate it with treatment outcome.
- 1.2.6 To describe the tumor molecular profile using RNA sequencing (RNAseq) and correlate it with treatment outcome.

### 1.3 Exploratory Objectives

- 1.3.1 To measure the tumor-infiltrating CD8+ T lymphocytes in pre- and on-treatment biopsies.
- 1.3.2 To measure tumor-infiltrating myeloid derived suppressor cells (MDSCs) in pre- and ontreatment biopsies.
- 1.3.3 To measure tumor-infiltrating tumor-associated macrophages (TAM) in the pre and ontreatment biopsies.
- 1.3.4 To measure the expression of programmed death-ligand 1 (PD-L1) in tumor cells and infiltrating immune cells.


#### 2. BACKGROUND

### 2.1 Study Disease

Neuroendocrine neoplasms (NENs) are rare cancers contributing to 1-2% of cancers diagnosed in the western hemisphere (Taal *et al.*, 2004; Basu *et al.*, 2010; Dasari *et al.*, 2017). Studies show a rise in their incidence in the United States (US), from 1.09/100,000 population in 1973 to 6.98/100,000 in 2012 (Dasari *et al.*, 2017). This is mostly attributed to increased use of better diagnostic imaging. There are regional reports indicating an incidence of 10.3 per 100,000 population (Chauhan *et al.*, 2018). Given the mostly indolent nature of the disease, the prevalence is much higher than its incidence. The gastrointestinal tract is the most common site of origin (55-60%), followed by the bronchopulmonary tract (20-30%). Other sites include genitourinary, biliary, soft tissue, and head and neck (Taal *et al.*, 2004; Maggard *et al.*, 2004).

The 2018 WHO classification system reclassified NENs into well differentiated NETs and poorly differentiated neuroendocrine carcinomas (NECs) on a morphologic basis (Rindi *et al.*, 2018). Based on Ki-67 index or mitotic index, well-differentiated NETs are further classified into low-grade (G1, Ki-67 index <3%, mitotic index <2 per 2 mm²); intermediate-grade (G2, Ki-67 index 3-20%, mitotic index 2-20 per 2 mm²); and high-grade (G3, Ki-67 index >20%, mitotic index >20 per 2 mm²). This reclassification highlights the better understanding of the histological subtypes and their importance in the prognosis and treatment of these patients (Bosman *et al.*, 2010; Kim *et al.*, 2017). Tumor grade corresponds to disease virulence in the well differentiated NETs. Median overall survival (OS) is reported to be 16.2 years, 8.3 years, and 10 months in low-, intermediate-, and high-grade disease, respectively (Dasari *et al.*, 2017).

Poorly-differentiated NECs can have small cell, large cell, or mixed phenotypes. It is estimated that poorly-differentiated NECs contribute to about 10-20% of all the cases of NENs (Dasari *et al.*, 2017; Kang *et al.*, 2017; Yao *et al.*, 2008). Poorly-differentiated NECs have an aggressive clinical course, marked by presentation at a late stage and dismal median overall survival. A report from the Nordic NEC study showed the median OS of patients with gastrointestinal NEC to be 11 months with palliative chemotherapy and only 1 month with best supportive care alone (Sorbye *et al.*, 2013).

## 2.1.1 Currently accepted treatment strategies for poorly-differentiated NECs

Poorly-differentiated NECs with small cell phenotype outside of the thorax are generally labelled as extra pulmonary small cell carcinomas. Other phenotypes, large cell, or mixed NECs are also seen. Regardless of the heterogeneity in origin, poorly-differentiated NECs are uniformly fatal and are traditionally treated with a platinum and etoposide combination, a regimen used to treat small cell carcinoma of the lungs, the efficacy of which was shown in small single-arm studies (Mitry *et al.*, 1999; Moertel *et al.*, 1991).

Smaller studies have shown response rates to platinum etoposide combination chemotherapy ranging from 40-67% and median OS ranging from 15 to 19 months (Mitry *et al.*, 1999; Moertel *et al.*, 1991; Imai *et al.*, 2016; Iwasa *et al.*, 2010; Patta *et al.*, 2011). Second line treatment options reported include reintroduction of platinum-etoposide, temozolomide-based regimens,


topotecan, FOLFOX, and FOLFIRI. Response rates with these regimens in the second line varies from 0-40%, with a median OS ranging from 3.2 to 18 months (Sorbye *et al.*, 2013; Olsen *et al.*, 201; Hentic *et al.*, 2012; Hadoux *et al.*, 2015). Overall, there is a paucity of effective treatment options for patients with high-grade NENs, which follow a very aggressive clinical course, beyond these traditional chemotherapy regimens tried based on pure empiricism.

### 2.1.2 Immunotherapy and NENs

Immunotherapy has been explored for the treatment of NENs in the era of interferon (IFN)-based therapy. Although there was clinical benefit shown from IFN-based therapy, because of difficulty of administration and resulting increased toxicity, such treatment has not been adopted into a routine clinical practice (Oberg *et al.*, 1991; Oberg *et al.*, 1986). Findings from small studies have shown that NENs are responsive to immune modulation. In metastatic pancreatic NETs, the efficacy of IFN was demonstrated after failure to first-line chemotherapy showing a biochemical response of 63% (20/32) with a median DOR of 20.5 months (Eriksson *et al.*, 1990). Oberg *et al.* treated 9 NET patients, including six with carcinoid syndrome, with daily intramuscular IFN for three months (Oberg *et al.*, 1983). All six syndromic patients experienced temporary relief in carcinoid syndrome symptoms and concomitant decline in urinary 5-hydroxyindoleacetic acid (5-HIAA) levels.

The role of IFNα-2b in combination with continuous fluorouracil infusion was studied in 24 patients with rapidly progressive NETs, 9 of which were confirmed high-grade NECs (Andreyev *et al.*, 1995). An ORR of 41.6% and a median DOR of 20 months were seen in all patients, with a response rate of 33% and median DOR of 6 months. The median OS of patients with the high-grade NECs was 8 months. Moertel *et al.* treated 27 of their NET patients with IFN, twenty-four of whom had carcinoid syndrome (Moertel *et al.*, 1989). Objective response (OR) was seen in 20% of the patients, while 39% of functional NET patients experienced reduction in urinary 5-HIAA (>50%) levels. In a prospective randomized clinical trial of octreotide (n=35) *versus* octreotide with IFN (n=33) for metastatic midgut carcinoid tumor patients, a superior PFS was evident for the combination arm (Kolby *et al.*, 2003).

## 2.1.2.1 Immune-Checkpoint inhibitors and high-grade NECs

On analysis of 37 cases of poorly differentiated NEC of the digestive tract, programmed cell death protein-1 (PD-1) expression on tumor cells and tumor-associated immune cells was seen in 16% and 63%, respectively (Roberts *et al.*, 2017). The expression of PD-L1 was seen on tumor cells and tumor associated immune cells in 14% and 27% respectively. There was no difference in PD-1 and PD-L1 expression between small cell and large cell NECs. The expression of PD-1 and PD-L1 in small cell NECs was studied in 94 patient-derived samples (61 pulmonary, 33 extrapulmonary) (Schultheis *et al.*, 2015). PD-L1 and PD-1 expression was seen in the stroma and not on the carcinoma cells themselves. On immunohistochemistry, 18.5% of the samples had expression of PD-L1 on their tumor-infiltrating macrophages, while 48% showed PD-1 expression on tumor-infiltrating lymphocytes. On RNA sequencing, there was moderate PD-L1 gene expression in 37.2 %, while PD-L2 was expressed in 27.9%.


There is scarcity of completed study of checkpoint inhibitors in high-grade neuroendocrine neoplasms, with the exception of Merkel-cell carcinoma and small cell lung carcinoma. The SWOG DART study has 19 patients with high grade neuroendocrine tumors, with a good number of poorly differentiated NEC. There was a very good response rate (>40%) to nivolumab/ipilimumab in this cohort as presented at the American Association for Cancer Research (AACR) 2019 annual meeting (AACR Press Release, 31 March 2019).

In patients with chemotherapy-refractory Merkel-cell carcinoma, avelumab showed an ORR of 32%, with a complete response of 9% (Kaufman *et al.*, 2016). Pembrolizumab had an ORR of 56%, of which 16% were complete responses (CRs) in treatment-naïve patients with advanced Merkle-cell carcinoma (Nghiem *et al.*, 2016).

In patients with chemotherapy-resistant extensive stage small cell lung cancer with PD-L1 expression, pembrolizumab showed an ORR of 33% (Ott *et al.*, 2017). The median time to response was 2 months (range 1.7-3.7) and the median DOR was 19.4 months (range: 3.6-20). The median PFS was 1.9 months (95% confidence interval [CI], 1.7-5.9). The median OS was 9.7 months (95% CI, 4.1 to NR).

A multicenter phase 1/2 study was conducted in patients with small cell lung cancer after the failure of at least one prior platinum-based chemotherapy regimen, using nivolumab alone or nivolumab and ipilimumab combination (Antonia *et al.*, 2016). Confirmed OR was seen in 10% of patients treated with nivolumab 3 mg/kg (n=98), in 23% of patients treated with nivolumab 1 mg/kg plus ipilimumab 3 mg/kg (n=61), and 19% of patients treated with nivolumab 3 mg/kg plus ipilimumab 1mg/kg (n=54). The median OS was 4.4 months (95% CI, 3.0–9.3) in the nivolumab 3 mg/kg cohort, 7.7 months (3.6–18.0) in the nivolumab 1 mg/kg plus ipilimumab 3 mg/kg cohort, and 6.0 months (3.6–11.0) in the nivolumab 3 mg/kg plus ipilimumab 1 mg/kg cohort. Time to OR was 2 months for nivolumab alone, while it was 1.4 months in patients treated with nivolumab 3 mg/kg and ipilimumab 1 mg/kg. The median PFS was 1.4 months (95% CI, 1.4-1.9), 2.6 months (95% CI, 1.4-4.1), and 1.4 months (95% CI, 1.3-2.2) in the nivolumab alone, nivolumab 1 mg/kg plus ipilimumab 3 mg/kg and nivolumab 3 mg/kg plus ipilimumab 1 mg/kg cohorts respectively. PD-L1 expression was checked in 148 patients, of whom 17% had PD-L1 expression of 1% or more. There was tumor response irrespective of PD-L1 expression status.

### 2.2 CTEP IND Agents

#### 2.2.1 XL184 (cabozantinib)

XL184 (cabozantinib, Cabometyx®, Cometriq®) is an oral multi-targeted inhibitor of receptor tyrosine kinases (RTKs) with half-maximal inhibitory concentrations (IC50) ranging from 2 to 101 nM (XL184 [cabozantinib] Investigator's Brochure, 2018). The targets of XL184 (cabozantinib) include several RTKs known to play important roles in tumor cell proliferation and/or tumor neovascularization, namely VEGFR2, MET, AXL, and RET. Other recognized targets of XL184 (cabozantinib) include ROS1, TRKA, TRKB, TIE2, TYRO3, and MER, two additional members of the VEGFR family (VEGFR1, VEGFR3), and the closely related RTKs KIT and FLT-3. The mode of action for XL184 (cabozantinib) is similar to other drugs targeting


RTKs: binding in a fully reversible manner to a region of the kinase domain (including the ATP-binding site) which forces the kinase activation loop into a pseudo-inactive conformation, thereby inhibiting subsequent catalytic activity. Both MET and VEGFR2 are important mediators of tumor growth and tumor angiogenesis, and *in vivo* pharmacodynamic activity of XL184 (cabozantinib) against MET and VEGFR2 has been demonstrated in both preclinical and clinical studies.

RTKs regulate many processes including cell growth and survival, organ morphogenesis, neovascularization, and tissue repair (Christensen *et al.*, 2005). Dysregulation of RTKs by mutation, gene rearrangement, gene amplification, or overexpression of the receptor or its ligands have been implicated as causative factors in the development and progression of numerous cancers.

The proto-oncogene *MET* encodes the high-affinity receptor for hepatocyte growth factor (HGF) (also known as scatter factor [SF]) (Christensen *et al.*, 2005). MET and HGF are each required for normal mammalian development and have been shown to be important in cell migration, morphogenic differentiation, and organization of three-dimensional tubular structures (*e.g.*, renal tubular cells, gland formation, *etc.*), as well as cell growth, angiogenesis, and tumor invasiveness and metastasis. Upregulation of MET is found in a wide range of malignancies including thyroid, prostate, ovarian, lung, and breast cancers, and is associated with more aggressive and invasive phenotypes of cancer cells *in vitro* and metastases *in vivo* (XL184 [cabozantinib] Investigator's Brochure, 2018). MET-driven metastasis may be exacerbated by a number of factors, including tumor hypoxia caused by selective inhibition of the VEGF pathway.

Evidence linking MET and HGF as causative or progression factors in human cancers includes the overexpression of both receptors and ligands in neoplasms relative to surrounding tissues, the correlation of receptor and ligand overexpression with disease severity and outcome, and genetic alteration of *MET* by mutation or gene amplification in multiple cancer types (Christensen *et al.*, 2005). Introduction of MET and HGF, or mutant MET into cell lines conferred the properties of tumorgenicity and metastatic propensity on engineered cells and introduction of MET or HGF as transgenes into the germline of mice resulted in primary and secondary neoplasms. The inhibition of MET or HGF function with dominant-negative receptors, antibody antagonists (both MET and HGF), or biologic antagonists (*e.g.*, NK4) have reversed cancer-associated phenotypes such as motility, invasion and proliferation of tumor cells, and tumor growth and dissemination in vivo.

A wide variety of human cancers, including brain, colorectal, gastric, and lung, demonstrate dysregulated MET activity (Liu *et al.*, 2010), either by means of MET kinase overexpression (Comoglio *et al.*, 2008), activating MET gene mutations and/or amplification (Comoglio *et al.*, 2008; Jeffers *et al.*, 1997; Schmidt *et al.*, 1997), or increased autocrine and/or paracrine secretion of the MET ligand, HGF/SF (Birchmeier *et al.*, 2003; Boccaccio and Comoglio, 2006). These alterations have been implicated in tumor progression and metastasis, and high constitutive activation of MET has been correlated with poor clinical prognosis (Birchmeier *et al.*, 2003).

VEGFR2 is the predominant mediator of VEGF-stimulated endothelial cell migration, proliferation, survival, and enhanced vascular permeability (Roskoski, 2008). Increased


expression of VEGFR2, often in combination with VEGFR3, has been observed in the tumor vascular endothelium in most common human solid tumor types, on tumor cells in melanoma and hematological malignancies, and in colitis-associated colon cancer (Tugues *et al.*, 2011). High VEGFR2 expression is an unfavorable prognostic biomarker in hepatocellular carcinoma (HCC), and correlated with triple-negative (*i.e.*, therapy-resistant) breast cancer (TNBC) and poor survival.

# 2.2.1.1 Nonclinical Development of XL184 (cabozantinib)

### 2.2.1.1.1 Nonclinical *In Vivo* Activity

Data from pharmacodynamic experiments have shown that XL184 (cabozantinib) inhibits MET and VEGFR2 *in vivo*. Oral administration of XL184 (cabozantinib) resulted in blockade of MET phosphorylation in human lung tumor xenografts grown in nude mice, blockade of MET phosphorylation in livers of mice, and blockade of VEGFR2 phosphorylation in mouse lung tissue. For both targets, the duration of action for XL184 (cabozantinib) was sustained, with >50% inhibition observed for >8 hours post-dose at a single dose level of 100 mg/kg (Yakes *et al.*, 2011). In addition, oral administration of XL184 (cabozantinib) resulted in blockade of phosphorylation of mutationally activated RET in TT human MTC xenografts grown in nude mice (Bentzien *et al.* 2013).

Treatment with XL184 (cabozantinib) results in anti-angiogenic effects in xenograft tumors, with disruption of the vasculature beginning within 24 hours after administration, and is associated with pro-apoptotic effects (Yakes *et al.* 2011). These effects translate into significant tumor growth inhibition or tumor regression after XL184 (cabozantinib) treatment in multiple tumor models including MTC, breast cancer, lung carcinoma, and glioblastoma.

Inhibition of the VEGF signaling pathway alone was previously shown to result in more invasive tumors in the transgenic RIP-Tag2 mouse model of neuroendocrine pancreatic cancer that spontaneously develops aggressive tumors (Pàez-Ribes *et al.* 2009). Treatment with XL184 (cabozantinib) for 3 weeks, from age 14 to 17 weeks, significantly prevented formation of liver metastases in the RIP-Tag2 model compared with anti-VEGF treatment or vehicle alone (P<0.05 vs. vehicle and anti-VEGF antibody). The number of liver metastases was 5-fold greater in anti-VEGF antibody-treated animals compared with vehicle-treated animals, and no liver metastases were detected in XL184 (cabozantinib)-treated animals. In addition, treatment with XL184 (cabozantinib) from age 14 to 20 weeks improved survival. Median survival was 14.7 weeks for vehicle-treated animals (n=12) and 16.4 weeks for anti-VEGF antibody-treated animals (n=7; P<0.05 vs. vehicle), and all XL184 (cabozantinib)-treated animals survived for the full 20 weeks of observation (n=6; P<0.05 vs. vehicle and anti-VEGF antibody).

### 2.2.1.1.2 Nonclinical Pharmacokinetics

Nonclinical pharmacokinetics (PK) of XL184 (cabozantinib) was studied in mice, rats, dogs, and monkeys (XL184 [cabozantinib] Investigator's Brochure, 2018). Oral bioavailability was comparably high in rats (80-86%), dogs (87%) and monkeys (73%) and moderately high in mice (42-51%) when XL184 (cabozantinib) was formulated with an aqueous vehicle. In rats, systemic


drug exposure parameters (maximum plasma concentration  $[C_{max}]$  and area under the concentration-time curve [AUC] from 0 hours to a specific post-dose time [AUC<sub>0-t</sub>]) increased less than dose-proportionally in association with single XL184 (cabozantinib) oral doses, and generally dose-proportionally with moderate accumulation ( $\leq$ 4-fold) following repeat daily oral dosing. In dogs, systemic drug exposure parameters increased less than dose-proportionally with increasing single XL184 (cabozantinib) oral doses, and generally dose-proportionally with little or no accumulation ( $\leq$ 2-fold increase) following repeat daily dosing.

### 2.2.1.1.3 Toxicology

Toxicity associated with oral administration of XL184 (cabozantinib) was characterized in definitive (Good Laboratory Practice [GLP]-compliant) single-dose and repeat-dose studies in mice, rats, and dogs; a fertility study in rats; embryotoxicity/teratogenicity studies in rats and rabbits; juvenile toxicity studies in rats; in vitro and in vivo genotoxicity bioassays; and an in vitro phototoxicity study (XL184 [cabozantinib] Investigator's Brochure, 2018). Target tissues for XL184 (cabozantinib)-related toxicity identified in these studies include gastrointestinal (GI) tract, bone marrow, lymphoid tissues, reproductive tract tissues, endocrine tissues, kidney, and skin. Histopathologic changes were also present in bone, central nervous system (CNS) tissues and liver/gall bladder. Adverse findings associated with XL184 (cabozantinib) administration were observed in both rodent and non-rodent species and were generally dose-related and often correlative with clinical signs and/or clinical pathology parameter changes reflective of associated target tissue histopathologic findings. Adverse findings were generally reversible upon discontinuation of treatment. In definitive reproductive and developmental toxicity studies, XL184 (cabozantinib) reduced fertility in male and female rats, was embryotoxic in rats, produced a fetal soft-tissue malformation (small spleen) in rabbits, and produced fetal external malformations (cleft palate/lip, dermal aplasia and kinked or rudimentary tail) in rats. XL184 (cabozantinib) was negative in *in vitro* bacterial and mammalian genotoxicity, clastogenicity, and phototoxicity bioassays. The metabolite present at highest plasma concentrations in humans administered XL184 (cabozantinib), EXEL-1644, was negative in an in vitro bacterial genotoxicity bioassay and caused no systemic tissue toxicity in rats dosed subcutaneously with EXEL-1644 for 2 weeks.

#### 2.2.1.2 Clinical Development of XL184 (Cabozantinib)

Patients have received XL184 (cabozantinib) in 18 Exelixis-sponsored clinical trials, 35 investigator-sponsored studies, and 19 NCI Cancer Therapy Evaluation Program (CTEP)-sponsored studies (XL184 [cabozantinib] Investigator's Brochure, 2018). The maximum tolerated dose (MTD) on once daily oral (PO) dosing schedule was determined to be 175 mg L-malate salt (or approximately 138 mg freebase equivalent by weight). Detailed information for each of these studies, including pharmacokinetic data, can be found in the XL184 (cabozantinib) Investigator's Brochure (2018). Safety and efficacy information from the 2018 XL184 (cabozantinib) Investigator's Brochure is summarized below.


### 2.2.1.2.1 Safety

Across Exelixis-sponsored studies with single-agent XL184 (cabozantinib), the most frequently observed adverse events (AEs) (≥20% of patients), regardless of causality, were diarrhea, fatigue, decreased appetite, nausea, palmar-plantar erythrodysaesthesia syndrome (PPES), vomiting, weight loss, constipation, hypertension, dysgeusia, dysphonia, and asthenia (Investigator's Brochure, 2018). The most frequently observed serious AEs (SAEs) (≥2% of patients), regardless of causality, were pulmonary embolism (PE), pneumonia, general physical health deterioration, vomiting, nausea, dehydration, anemia, and diarrhea. In these single-agent studies, 42 patients had grade 5 AEs that were assessed as related to study treatment. The only related grade 5 AEs that occurred more than once were PE (n=5), hepatic failure (n=3); death (unspecified; n=3), hemorrhage (n=2), respiratory failure (n=2), sudden death (n=2), and GI perforation (n=2). In investigator-sponsored and CTEP-sponsored trials, the most frequent SAEs were embolism, nausea, dyspnea, dehydration, fatigue, and hypophosphatemia.

# 2.2.1.2.2 Efficacy

The clinical activity of XL184 (cabozantinib) has been evaluated in pivotal trials in renal cell cancer (RCC), hepatocellular carcinoma (HCC), MTC, and castrate-resistant prostate cancer (CRPC) (XL184 [cabozantinib] Investigator's Brochure, 2018). In phase 1 and 2 studies, XL184 (cabozantinib) has also demonstrated findings consistent with broad clinical antitumor activity in multiple tumor types.

Phase 3, randomized, open-label, active-controlled Study XL184-308 was conducted in 658 patients (330 XL184 [cabozantinib], 328 everolimus) with advanced RCC who had received prior treatment with at least one VEGFR-tyrosine kinase inhibitor (TKI) (XL184 [cabozantinib] Investigator's Brochure, 2018). XL184 (cabozantinib) demonstrated statistically significant improvements in the primary endpoint (PFS) and both secondary endpoints (ORR and OS) compared with the standard-of-care control treatment (everolimus). In the primary PFS analysis performed in the first 375 patients randomized, the hazard ratio (HR) adjusted for stratification factors was 0.58 (95% CI, 0.45-0.74; stratified logrank P<0.0001), and the Kaplan-Meier estimates for median PFS were 7.4 months in the XL184 (cabozantinib) arm vs. 3.8 months in the everolimus arm. The PFS analysis was repeated in all 658 patients, and the results (stratified HR = 0.51 [95% CI, 0.41-0.62]) were similar to those obtained from the initial analysis. In the primary analysis of ORR, the ORRs for the XL184 (cabozantinib) and everolimus arms were 17% (95% CI, 13%-22%) and 3% (95% CI, 2%-6%), respectively (unstratified *P*<0.0001). Kaplan-Meier estimates for median OS were 21.4 months in the XL184 (cabozantinib) arm and 16.5 months in the everolimus arm. Results for extensive subgroup analyses of PFS, OS, and ORR showed a consistent benefit for XL184 (cabozantinib) treatment versus everolimus.

Phase 2, randomized, open-label, active-controlled Study A031203 (CABOSUN), was sponsored by CTEP and conducted by The Alliance for Clinical Trials in Oncology (Alliance) in 157 patients (79 XL184 (cabozantinib), 78 sunitinib) with untreated clear cell locally advanced or metastatic RCC of intermediate or poor risk (XL184 [cabozantinib] Investigator's Brochure, 2018). Compared with the standard-of-care control treatment, sunitinib, XL184 (cabozantinib) demonstrated statistically significant improvements in the primary endpoint of PFS and the


secondary endpoint of ORR as well as a non-significant trend of improvement in the secondary endpoint of OS. In the primary analysis performed by the Alliance, a benefit in PFS per investigator assessment was demonstrated for XL184 (cabozantinib) compared with sunitinib. In Exelixis-initiated retrospective primary PFS and secondary ORR analyses based on blinded assessments, there was a statistically significant improvement in PFS for patients in the XL184 (cabozantinib) arm compared with the sunitinib arm (HR=0.48 [95% CI, 0.31-0.74]; stratified 2-sided logrank P=0.0008); median PFS was 8.6 months in the XL184 (cabozantinib) arm and 5.3 months in the sunitinib arm. Further, ORR (secondary endpoint) per IRC in the XL184 (cabozantinib) arm was improved compared with the sunitinib arm: 20% vs. 9% (stratified 2-sided P=0.0406). In an OS (secondary endpoint) analysis of data, the Kaplan-Meier estimates for median OS were 30.3 months in the XL184 (cabozantinib) arm vs. 21.0 months in the sunitinib arm (stratified HR adjusted for stratification factors was 0.74 [95% CI, 0.47-1.14]; stratified 2-sided logrank P=0.1700).

A total of 707 patients (470 XL184 (cabozantinib), 237 placebo) with advanced HCC who had received prior treatment with sorafenib were enrolled in phase 3, randomized, double-blinded, placebo-controlled Study XL184-309 through the 01 June 2017 database cutoff date (XL184 [cabozantinib] Investigator's Brochure, 2018). In the study, XL184 (cabozantinib) demonstrated a robust and statistically significant improvement in OS, PFS, and ORR. The analysis of duration of OS (primary endpoint) demonstrated a statistically significant improvement for patients in the XL184 (cabozantinib) arm compared with the placebo arm: the HR, adjusted for stratification factors was 0.76 (95% CI, 0.63-0.92; stratified logrank P=0.0049). The Kaplan-Meier estimates for median OS were 10.2 months in the XL184 (cabozantinib) arm vs. 8.0 months in the placebo arm. A statistically significant improvement in PFS for patients in the XL184 (cabozantinib) arm compared with the placebo arm was also observed. The HR, adjusted for stratification factors was 0.44 (95% CI, 0.36-0.52; stratified logrank P<0.0001). The Kaplan-Meier estimates for median PFS were 5.2 months in the XL184 (cabozantinib) arm vs. 1.9 months in the placebo arm. The ORR was 4% and 0.4% for patients in the XL184 (cabozantinib) and placebo arms, respectively (stratified Cochran-Mantel-Haenszel [CMH] test P=0.0086).

Phase 3, randomized, double-blind, placebo-controlled study XL184-301 was conducted in 330 MTC patients (219 XL184 (cabozantinib), 111 placebo) (XL184 [cabozantinib] Investigator's Brochure, 2018). An increase in PFS (primary endpoint) was seen, with a median PFS of 11.2 months in the XL184 (cabozantinib) arm compared with 4.0 months for placebo (HR=0.28 [95 CI, 0.19-0.40]). For the secondary endpoint of ORR, confirmed PRs occurred in 28% of XL184 (cabozantinib)-treated patients and no placebo-treated patients and responses were durable (median DOR=14.6 months). The final analysis of the secondary endpoint of OS included 218 deaths and showed a non-significant trend for improved median OS in the XL184 (cabozantinib) arm compared with the placebo arm (26.6 months *vs.* 21.1 months; HR=0.85 [95% CI, 0.64-1.12]; *P*=0.2409). Because MTC is a relatively rare disease, the study was not designed to be large enough to provide high power to detect the minimum clinically significant difference in the secondary endpoint of OS. The subgroup analysis of patients with a RET M918T mutation revealed a larger improvement in OS for the XL184 (cabozantinib) arm: the median OS was 44.3 months for the XL184 (cabozantinib) arm *versus* 18.9 months for the placebo arm (HR=0.60 [95% CI, 0.38-0.94]; *P*=0.0255, not adjusted for multiple subgroup analyses). In all


patients, the median duration of XL184 (cabozantinib) treatment was 10.8 months, and the 75th percentile for duration of treatment was 24.8 months. The maximum duration of treatment was 59.4 months at the data cutoff of the final OS analysis.

In addition to RCC, HCC, and MTC, XL184 (cabozantinib) has demonstrated findings consistent with broad clinical antitumor activity in multiple other tumor types (XL184 [cabozantinib] Investigator's Brochure, 2018). Observations of clinical activity have included decrease of soft tissue tumor lesions including visceral metastases, reduction in serum markers of bone resorption and formation, and reduction in circulating tumor cells (CTCs) in patients with prostate cancer. Though they failed to meet their respective primary endpoints of OS and pain response, phase 3 studies XL184-307 and XL184-306 demonstrated clinical activity in CRPC including effects on PFS (XL184-307) and bone scan response (both studies). Clinical antitumor activity has also been observed in company-sponsored phase 1 and 2 studies across indications including non-small cell lung cancer (NSCLC), breast cancer, melanoma, ovarian cancer, glioblastoma (GB), and differentiated thyroid cancer (DTC).

### 2.2.1.3 Marketing Experience

XL184 (cabozantinib) is approved in the United States as Cometriq<sup>®</sup> for the treatment of progressive, metastatic MTC and as Cabometyx<sup>®</sup> for advanced RCC (XL184 [cabozantinib] Investigator's Brochure, 2018). As of February 2018, commercial exposure in the post-marketing setting to Cometriq<sup>®</sup> was estimated as >2000 patients and exposure to Cabometyx<sup>®</sup> was estimated as >12000 patients. No new safety signals associated with Cometriq<sup>®</sup> or Cabometyx<sup>®</sup> were observed in post-marketing.

### 2.2.2 Nivolumab

Nivolumab (BMS-936558, MDX-1106, ONO-4538, Opdivo®) is a fully human monoclonal immunoglobulin G4 (IgG4) antibody (HuMAb) that is specific for human PD-1, cluster of differentiation 279 (CD279) cell surface membrane receptor (Nivolumab Investigator's Brochure, 2018). PD-1 is a negative regulatory molecule that is expressed transiently following T-cell activation and on chronically stimulated T-cells characterized by an "exhausted" phenotype. Nivolumab binds to cynomolgus monkey PD-1 but not mouse, rat, or rabbit molecules. Clinical activity of nivolumab has been observed in patients with a variety of cancers. The combination of nivolumab and ipilimumab, an anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) agent, in a phase 1/2 trial showed markedly enhanced clinical activity with an acceptable safety profile in patients with melanoma (Wolchok *et al.*, 2013). See Section 2.2.3 for more information about ipilimumab.

The clinical use of monoclonal antibodies to T-cell inhibitory receptors has provided transformative information on the nature of the immune system and cancer (Nivolumab Investigator's Brochure, 2018). An emerging picture suggests that endogenous immune responses can mediate effective tumor regression and/or improved survival even in patients with large volume tumors resistant to other forms of therapy. Some of the unique features of this type of therapy, based largely on experience in advanced melanoma, include: improved OS with or without radiographic responses or improved PFS; responses that may be delayed or occur after


radiographic disease progression; combinations of immune modulators with enhanced or novel activities (in the example of ipilimumab and nivolumab); and toxicity that is almost exclusively immune or inflammatory in nature. It is not yet clear what factors determine responses and which components of the immune system are needed for this to occur. It seems likely that both memory helper and effector cells would be needed to sustain long-term responses. Increasing emphasis has been placed on understanding the relationships of the tumor, cellular infiltrate, and immunologic milieu surrounding each tumor.

PD-1, a 55-kDa type 1 transmembrane protein, is a member of the CD28 family of T-cell costimulatory receptors that include Ig super family member CD28, CTLA-4, inducible costimulator (ICOS), and B and T lymphocyte attenuator (BTLA) (Nivolumab Investigator's Brochure, 2018). PD-1 is transiently, but highly expressed on activated T-cells and functions to limit immune effectors at the site of activation. Chronic stimulation may prevent the remethylation of the PD-1 gene leading to continuous expression and characterizes a state of "exhausted" T-cells that lose function and proliferative capacity while enhancing a suppressive tumor microenvironment. PD-1 may act together with other T-cell modulating molecules, including CTLA-4, TIM-3 (T-cell immunoglobulin mucin 3), lymphocyte-activation gene 3 (LAG-3) as well as indoleamine-pyrrole 2,3-dioxygenase 1 (IDO-1), cytokines, and transforming growth factor beta (TGF-β).

Two ligands specific for PD-1 have been identified: PD-L1, (also known as B7-H1 or CD274, expressed on tumor, antigen-presenting cells [APCs], and dendritic cells [DCs]) and PD-L2 (also known as B7-DC or CD273, expressed on endothelial cells). The interaction of PD-1 with PD-L1 and PD-L2 results in negative regulatory stimuli that down-modulate the activated T-cell immune response through SHP-1 phosphatase.

PD-1 knockout mice develop strain-specific lupus-like glomerulonephritis (C57BL/6) and cardiomyopathy (BALB/c). In transplantable tumor models that expressed PD-1 and LAG-3 on tumor-infiltrating CD4+ and CD8+ T-cells dual anti-LAG-3/anti-PD-1 antibody treatment cured most mice of established tumors that were largely resistant to single antibody treatment (Woo *et al.*, 2012). Despite minimal immunopathologic sequelae in PD-1 and LAG-3 single knockout mice, dual knockout mice abrogated self-tolerance with resultant autoimmune infiltrates in multiple organs, leading to eventual lethality.

PD-L1 expression is found on a number of tumors, and is associated with poor prognoses based on OS in many tumors, including melanoma (Taube *et al.*, 2012), renal (Thompson *et al.*, 2004; Thompson *et al.*, 2005; Thompson *et al.*, 2006), esophageal (Ohigashi *et al.*, 2005), gastric (Wu *et al.*, 2006), ovarian (Dong *et al.*, 2003), pancreatic (Nomi *et al.*, 2007), lung (Zitvogel *et al.*, 2006), and other cancers (Nivolumab Investigator's Brochure, 2018).

The PD-1/PD-L1 axis plays a role in human infections, particularly in hepatitis C virus (HCV) and human immunodeficiency virus (HIV). In these cases, high expression levels of PD-1 were found in viral-specific CD8+ T-cells that also display a non-responsive or exhausted phenotype. Non-responsive PD-1-high T-cells were observed in simian immunodeficiency virus (SIV) infection in rhesus macaques. Treatment of SIV-infected macaques with an anti-PD-1 mAb (3


 $mg/kg \times 4$ ) resulted in decreased viral loads and increased survival along with expanded T-cells with increased T-cell functionality.

## 2.2.2.1 Nonclinical Development of Nivolumab

In intravenous (IV) repeat-dose toxicology studies in cynomolgus monkeys, nivolumab alone was well tolerated (Nivolumab Investigator's Brochure, 2018). Combination studies have highlighted the potential for toxicity when combined with ipilimumab, MDX-1408, and BMS-986016. Nivolumab bound specifically to PD-1 (and not to related members of the CD28 family such as CD28, ICOS, CTLA-4, and BTLA) with a dissociation constant (K<sub>d</sub>) of 3.06 nM. A surrogate rat anti-mouse PD-1 antibody (4H2) was derived and expressed as chimeric IgG1 murine antibody. Antitumor activity was seen for several tumor models, including colon carcinoma and fibrosarcoma.

### 2.2.2.2 Clinical Development of Nivolumab

Nivolumab has demonstrated clinical activity, and has been approved for use in NSCLC, melanoma, RCC, classical Hodgkin's Lymphoma (cHL), squamous cell carcinoma (SCC) of the head and neck, and urothelial carcinoma as monotherapy and in combination with ipilimumab and other therapeutics (Nivolumab Investigator's Brochure, 2018). It has also demonstrated activity in other tumor types. The majority of responses were durable and exceeded 6 months. In randomized, controlled studies, nivolumab monotherapy demonstrated statistically significant improvement in OS over standard of care in patients with advanced or metastatic melanoma, patients with advanced or metastatic squamous cell carcinoma of the head and neck (SCCHN). In randomized, controlled studies, nivolumab in combination with ipilimumab demonstrated statistically significant improvement in PFS and ORR over ipilimumab monotherapy in patients with advanced or metastatic melanoma.

Nivolumab is also being evaluated in several other cancers, including small cell lung cancer (SCLC), gastric and esophageal cancer, hepatocellular carcinoma, colorectal cancer, GB, and Merkel cell carcinoma (MCC).

#### 2.2.2.2.1 Pharmacokinetics

PK of nivolumab was linear in the range of 0.3 to 10 mg/kg, with dose-proportional increases in  $C_{max}$  and AUC from time zero to infinity (AUC<sub>0-∞</sub>), with low to moderate inter-patient variability observed at each dose level (Nivolumab Investigator's Brochure, 2018). Clearance of nivolumab is independent of dose in the dose range (0.1 to 10 mg/kg) and tumor types studied. Body weight normalized dosing showed approximately constant trough concentrations over a wide range of body weights. The mean terminal elimination half-life of nivolumab is 17 to 25 days consistent with the half-life of endogenous IgG4.


### 2.2.2.2.2 Efficacy

In a randomized, open-label, phase 3 trial, patients with unresectable or metastatic melanoma who had progressed after treatment with ipilimumab were given either IV nivolumab (3 mg/kg every 2 weeks) or investigator's choice chemotherapy (ICC): dacarbazine 1000 mg/m² every 3 weeks or paclitaxel 175 mg/m² combined with carboplatin AUC=6 every 3 weeks) (Weber *et al.*, 2015). Of the first 120 patients treated with nivolumab, objective responses (CR or PR) were seen in 38 (31.7%) versus 5 (10.6%) out of 47 patients in the ICC arm. Grade 3-4 AEs related to nivolumab included increased lipase, increased alanine aminotransferase, anemia, and fatigue. Grade 3-4 drug-related SAEs were noted in 12 (5%) nivolumab-treated patients. No treatment-related deaths occurred.

In a phase 1/2 trial, patients with virus-positive and -negative solid tumors, including MCC, were given 240 mg nivolumab IV every 2 weeks (Nivolumab Investigator's Brochure, 2018). As of the February 16, 2017 data cutoff, of 25 patients with MCC who had received nivolumab, objective responses (PR or CR) were seen in 16 patients (64%, 95% CI 42.5%-82%). Median DOR, PFS, and OS have not been reached.

In a randomized, open-label, phase 3 trial, patients with recurrent SCCHN were given either IV nivolumab (3 mg/kg every 2 weeks) or standard systemic therapy (methotrexate, docetaxel, or cetuximab) (Ferris *et al.*, 2016). The median OS was 7.5 months (95% CI, 5.5-9.1 months) in the nivolumab group versus 5.1 months (95% CI, 4-6 months) in the group that received standard therapy. OS was significantly longer with nivolumab than with standard therapy (HR, 0.70 [97.73% CI, 0.51-0.96]; *P*=0.01), and the estimates of the 1-year survival rate were approximately 19% higher with nivolumab than with standard therapy (36.0% *vs.* 16.6%). The median PFS was 2 months (95% CI, 1.9-2.1 months) with nivolumab versus 2.3 months (95% CI, 1.9-3.1 months) with standard therapy (HR for disease progression or death, 0.89 [95% CI, 0.70-1.13]; *P*=0.32). The PFS rate at 6 months was 19.7% with nivolumab versus 9.9% with standard therapy. The response rate was 13.3% in the nivolumab group versus 5.8% in the standard-therapy group. Treatment-related AEs of grade 3 or 4 occurred in 13.1% of the patients in the nivolumab group versus 35.1% of those in the standard-therapy group. Physical, role, and social functioning was stable in the nivolumab group, whereas it was meaningfully worse in the standard-therapy group.

In an open-label, phase 2 trial, patients with recurrent or metastatic colorectal cancer assessed as MSI-high were given 3 mg/kg IV nivolumab every 2 weeks as monotherapy, or in combination with 1 mg/kg IV ipilimumab every 3 weeks for 4 doses followed by 3 mg/kg IV nivolumab every 2 weeks (Nivolumab Investigator's Brochure, 2018; Overman *et al.*, 2017). As of the September 19, 2016 data cut-off, 74 patients had received nivolumab monotherapy and 30 had received combination nivolumab/ipilimumab therapy. At a median follow-up of 12 months, 23 of 74 nivolumab-treated patients (31.1% [95% CI, 20.8%-42.9%]) achieved an objective response and 51 patients (69% [95% CI, 57%-79%]) had disease control for 12 weeks or longer. As of the data cut-off, median DOR had not yet been reached; all responders were alive, and eight had responses lasting 12 months or longer (Kaplan-Meier 12-month estimate, 86% [95% CI, 62%-95%]). Median PFS was 7.6 months (95% CI, 3 months-not reached [NR]). The 6- and 12-month PFS rates were 51.5% (95% CI, 38.9%-62.8%) and 45.6% (95% CI, 32.2%-58.1%),


respectively. The 6- and 12-month OS rates were 83.4% (95% CI, 72.5%-90.2%) and 73.8% (95% CI, 59.8%-83.5%), respectively. The most common grade 3 or 4 drug-related AEs were increased concentrations of lipase (six patients, 8%) and amylase (two patients, 3%). Twenty-three patients (31%) died during the study; none of these deaths were deemed to be treatment related by the investigator. Out of 30 patients who had received nivolumab and ipilimumab combination therapy, 27 were evaluable for response (Nivolumab Investigator's Brochure, 2018). Of these, objective responses were seen in 9 patients (33.3%, 95% CI, 18.6%-50.9%). The 6-month PFS rate was 66.6% (95% CI, 45.5%-81.1%) and the 6-month OS rate was 85.1% (95% CI, 65.0%-94.2%).

### 2.2.2.2.3 Toxicology

An MTD of nivolumab was not reached at any dose up to 10 mg/kg (Topalian *et al.*, 2012; Nivolumab Investigator's Brochure, 2018). There was no pattern in the incidence, severity, or causality of AEs to nivolumab dose level. Most AEs were low-grade (Grade 1-2) with relatively few drug-related high-grade (Grade 3-4) AEs. The safety profile of nivolumab combination therapy varies with the agent combined with nivolumab but is generally consistent with the safety profiles observed with either agent alone and, in some cases, both frequency and severity of AEs were greater than that observed with either agent alone. The safety profile of nivolumab + ipilimumab combination therapy was consistent with the mechanisms of action of nivolumab and ipilimumab (Nivolumab Investigator's Brochure, 2018). A dose of 3 mg/kg nivolumab/3 mg/kg ipilimumab exceeded the MTD, and both 1 mg/kg nivolumab/3 mg/kg ipilimumab and 3 mg/kg nivolumab/1 mg/kg ipilimumab were identified as the MTD. For nivolumab monotherapy and combination therapy, most high-grade events were manageable with use of corticosteroids or hormone replacement therapy (endocrinopathies).

The overall safety experience with nivolumab is based on experience in approximately 16,900 patients who received either nivolumab alone or in combination with other therapeutics (Nivolumab Investigator's Brochure, 2018). In general, for monotherapy, the safety profile is similar across tumor types. The only exception is pulmonary inflammation AEs, which may be numerically greater in patients with NSCLC, possibly because in some cases, it can be difficult to distinguish between nivolumab-related and unrelated causes of pulmonary symptoms and radiographic changes. The most frequently reported treatment-related AE is fatigue, which is almost always of low grade.

# 2.2.2.4 Pharmacodynamics/Biomarkers

Tumor-cell expression (melanoma) of PD-L1 was characterized in combination with ipilimumab with the use of immunohistochemistry (IHC) staining and pharmacodynamics changes in the peripheral-blood absolute lymphocyte count (Wolchok *et al.*, 2013). With PD-L1 positivity defined as expression in at least 5% of tumor cells, biopsy specimens from 21 of 56 patients (38%) were PD-L1 positive. Among patients treated with the concurrent regimen of nivolumab and ipilimumab, ORs were observed in patients with either PD-L1–positive tumor samples (6 of 13 patients) or PD-L1–negative tumor samples (9 of 22). In the sequenced regimen cohorts, a higher number of overall responses was seen among patients with PD-L1–positive tumor samples (4 of 8 patients) than among patients with PD-L1–negative tumor samples (1 of 13)


suggesting the possibility that these tumors have higher response rates to the combination. The relationship between PDL-1 expression and responses may not be present in patients treated with the combination. Tissue expression of PDL-2, interferon-gamma (IFN- $\gamma$ ), indoleamine 2,3 dioxygenase (IDO), and T-cell CD8+ are of current interest. Until more reliable data based on standardized procedures for tissue collection and assays are available, PD-L1 status cannot be used to select patients for treatment at this time.

## 2.2.2.3 Marketing Experience

Nivolumab monotherapy (Opdivo®) was first approved in July 2014 in Japan for unresectable melanoma (Nivolumab Investigator's Brochure, 2018). Since then, it has been approved in multiple countries, including the US, and has been approved for several other indications, including metastatic NSCLC, advanced RCC, cHL, SCCHN, urothelial carcinoma, HCC, RCC, and adjuvant treatment of melanoma. Nivolumab is also approved in combination with ipilimumab for unresectable or metastatic melanoma in multiple countries, including the US, and for previously untreated advanced RCC in the US. Qualitative and quantitative safety data has been consistent with the established safety profile as observed in clinical trials. No new safety concerns have been identified based on global post-marketing reports.

### 2.2.3 Ipilimumab

Ipilimumab (BMS-734016, MDX010, MDX-CTLA4, Yervoy®) is an Ig-G1κ HuMAb specific for human cytotoxic T lymphocyte antigen 4 (CTLA-4, CD152), which is expressed on a subset of activated T-cells (Ipilimumab Investigator's Brochure, 2018). CTLA-4 is a negative regulator of T-cell activation. Ipilimumab binds to CTLA-4 and inhibits its interaction with ligands on APCs. Blockade of CTLA-4 has been shown to augment T cell activation and proliferation, including the activation and proliferation of tumor-infiltrating T-effector cells. Inhibition of CTLA-4 signaling can also reduce Treg function, which may contribute to a general increase in T-cell responsiveness, including the anti-tumor response.

#### 2.2.3.1 Nonclinical Development of Ipilimumab

Ipilimumab has specificity and high affinity for human CTLA-4 (Ipilimumab Investigator's Brochure, 2018). The calculated dissociation constant value (K<sub>D</sub>) from an average of several studies was 5.25 nM. Binding of ipilimumab to purified, recombinant human CTLA-4 antigen was also demonstrated by enzyme-linked immunosorbent assay with half-maximal binding at 15 ng/mL, while saturation was observed at approximately 0.1 mcg/mL. No cross-reactivity was observed against human CD28. Ipilimumab completely blocked binding of the CTLA-4 ligands B7-1 and B7-2 to human CTLA-4 at concentrations higher than 6 mcg/mL and 1 mcg/mL, respectively.

*In vivo*, blockade of CTLA-4, utilizing anti-CTLA-4 mAb, induced regression of established tumors and enhanced antitumor immune responses in several murine tumor models (Ipilimumab Investigator's Brochure, 2018). Blockade of CTLA-4-mediated signals is effective in inducing rejection of immunogenic cancers in mice. Moreover, when anti-CTLA-4 mAb is used in conjunction with granulocyte macrophage-colony stimulating factor (GM-CSF)-secreting tumor


vaccines, poorly immunogenic cancers in mice are rejected. These findings suggest that CTLA-4 blockade, alone or in combination with antigenic stimulation and other immune modulating agents can induce a potent antitumor response. Complete information on pre-clinical studies can be found in the ipilimumab Investigator's Brochure (2018).

# 2.2.3.2 Clinical Development of Ipilimumab

Bristol-Myers Squibb (BMS) and Medarex (acquired by BMS in September 2009) have cosponsored an extensive clinical development program for ipilimumab, encompassing >22,571 patients in several cancer types in completed and ongoing studies, including a compassionate use program (Ipilimumab Investigator Brochure, 2018). The focus of the clinical program is in melanoma, prostate cancer, and lung cancer, with advanced melanoma being the most comprehensively studied indication. Ipilimumab is being investigated both as monotherapy and in combination with other modalities such as chemotherapy, radiation therapy, and other immunotherapies.

CTEP's clinical development of ipilimumab focuses on cervical, GI, ovarian, prostate cancer, chronic lymphocytic leukemia, head and neck squamous cell carcinoma, solid tumors, Hodgkin and non-Hodgkin lymphomas, melanoma, and myelodysplastic syndrome. While the toxicity and clinical responses overlap, mechanisms of immune activation and range of responses appear to be different for each of the single agents.

#### 2.2.3.2.1 Clinical Pharmacokinetics

The PK of ipilimumab was studied in 499 patients with unresectable or metastatic melanoma who received doses of 0.3, 3, or 10 mg/kg administered once every 3 weeks (q3w) for four doses (Ipilimumab Investigator's Brochure, 2018). C<sub>max</sub>, trough concentration (C<sub>min</sub>), and AUC of ipilimumab were found to be dose proportional within the dose range examined. Upon repeated dosing of ipilimumab administered q3w, ipilimumab clearance was found to be time-invariant, and minimal systemic accumulation was observed as evident by an accumulation index of 1.5-fold or less. Ipilimumab steady-state concentration was reached by the third dose. The mean terminal half-life was 14.7 days, systemic clearance (CL) was 15.3 mL/h, and the volume of distribution at steady-state (V<sub>ss</sub>) was 7.21 L. The mean ipilimumab C<sub>min</sub> achieved at steady-state with the 3-mg/kg regimen was 21.8 mcg/mL.

# 2.2.3.2.2 Safety

The immune-based mechanism of action is reflected in the safety profile of ipilimumab (Ipilimumab Investigator's Brochure, 2018). The most common treatment-related AEs are inflammatory in nature, consistent with the mechanism of action of the drug and generally medically manageable with topical and/or systemic immunosuppressants. Such immunological safety events are described as immune-related adverse events (irAEs) or immune mediated adverse reactions (imARs). The irAEs are described as AEs of unknown etiology, which were consistent with an immune phenomenon and considered causally related to drug exposure by the investigators. The irAEs primarily involve the GI tract and skin. Immune-related AEs in the liver were also observed, particularly in patients receiving 10 mg/kg. Endocrinopathy and


neuropathy were important irAEs that were observed less frequently. The imARs were adjudicated in a blinded fashion based on sponsor-physician data review to exclude noninflammatory etiologies, such as infection or tumor progression, and to consider available evidence of inflammation, such as tumor biopsies or responsiveness to steroids, in an effort to determine whether specific AEs or abnormal hepatic laboratory values were likely to be immune mediated and associated with ipilimumab treatment.

# 2.2.3.2.3 Efficacy

In melanoma, four completed phase 3 studies (MDX010-20, CA184024, CA184029, and CA184169) have demonstrated a clinically meaningful and statistically significant survival benefit in pretreated advanced melanoma, in previously untreated advanced melanoma, and in adjuvant melanoma (Ipilimumab Investigator's Brochure, 2018).

The unique immune-based mechanism of action is reflected in the clinical patterns of anti-cancer activity in some patients (Ipilimumab Investigator's Brochure, 2018). Ipilimumab induces an immunologic response, and measurable clinical effects emerge after the immunological effects. Tumor infiltration with lymphocytes and the associated inflammation (documented by biopsy in some patients) is likely the cornerstone of the effect of ipilimumab and can manifest in various patterns of clinical activity leading to tumor control. In some cases, inflammation may not be noted by radiological examination, and objective response is observed with the first tumor assessment in a manner seen in patients receiving other types of anti-cancer treatments. In other cases, response may be preceded by an apparent increase in initial tumor volume and/or the appearance of new lesions, which may be mistaken for tumor progression on radiological evaluations. Therefore, in patients who are not experiencing rapid clinical deterioration, confirmation of progression is recommended (at the investigator's discretion) to better understand the prognosis, as well as to avoid unnecessarily initiating potentially toxic alternative therapies in patients who might be benefiting from treatment. Immune-related response criteria were developed based on these observations to systematically categorize novel patterns of clinical activity and are currently being prospectively evaluated in clinical studies. In metastatic diseases, stabilization is more common than response, and in some instances is associated with a slow, steady decline in tumor burden over many months, sometimes improving to PRs and/or CRs. Thus, the immune-based mechanism of action of ipilimumab results in durable disease control, sometimes with novel patterns of response, which contribute to improvements in OS.

Available preclinical data support the combinations of nivolumab and ipilimumab (Curran *et al.*, 2010). The combination of ipilimumab with nivolumab has been reported to result in improved responses in advanced melanoma, including decreased time to response, increased number of responses, improved depth and duration of responses, and increased PFS and OS compared to single agent ipilimumab (Wolchok *et al.*, 2013).

### 2.2.3.3 Marketing Experience

Ipilimumab monotherapy (Yervoy®) was approved in the US in March 2011 for the treatment of advanced melanoma (Ipilimumab Investigator's Brochure, 2018). Ipilimumab has demonstrated long-term OS benefit extending beyond 5 years in both previously treated and untreated patients


with metastatic melanoma. Ipilimumab continues to demonstrate an overall favorable benefitrisk profile. Based on review of nonclinical, clinical, and post-marketing data, there has been no change in the effectiveness or safety of ipilimumab for the approved indications. The totality of data continues to support a significant clinical benefit for patients receiving ipilimumab with various other types of concomitant cancer stimulatory therapies.

### 2.3 Rationale

The lack of permissive tumor microenvironment is one of the frequently cited reasons why poor response to immunotherapy has been seen in many patients with metastatic carcinomas (Spranger *et al.*, 2013; Sharma *et al.*, 2015). Tumors that respond favorably to immunotherapy have been characterized as having more effector CD8+ T cell infiltrating the tumor stroma and fewer regulatory T cells (T regs), MDSCs, and TAMs amongst other factors. Tumors that have not responded favorably to checkpoint inhibition have been shown to have fewer effector T cells and more immunosuppressive T regs, MDSCs, and TAMs infiltrating the tumor microenvironment.

With the increasing understanding of the complexity of cancer and its progression, it has become increasingly clear that successful cancer treatment involves a combinatorial approach. Although the benefits of cancer immunotherapy have been astonishingly durable, they are limited to a portion of patients with permissive tumor microenvironment. Understanding the limitations of certain tumors with immunosuppressive microenvironment that do not respond to immunotherapy, a sound scientific argument is to attempt to convert a tumor phenotype to an "inflamed phenotype" which is likely to respond to immunotherapy. Different strategies to alter the composition of the tumor microenvironment have been suggested, but none have shown clinical success in changing immunotherapy resistant tumors to a responsive one.

In patients with refractory urothelial carcinoma who received XL184 (cabozantinib) treatment, there was a decreased level of T regs and increased expression of PD-1 by the T cells (Apolo *et al.*, 2014). In a novel chimeric mouse model of metastatic castration-resistant prostate cancer (mCRPC), there was a robust synergistic response when a checkpoint blockade was combined with XL184 (cabozantinib) and BEZ235 (inhibitor of PI3K/mTOR kinases) to attenuate MDSC activity, though the individual approaches showed only minimal responses (Lu *et al.*, 2017).

A phase 1 study of combination of XL184 (cabozantinib) with the checkpoint inhibitors, nivolumab and ipilimumab, was conducted in patients with refractory metastatic genitourinary cancers (Apolo *et al.*, 2016; Apolo *et al.*, 2017). In part 1, patients received XL184 (cabozantinib) with nivolumab, while in part 2 XL184 (cabozantinib) was given with nivolumab and ipilimumab. In both parts of the study, the combination of was well tolerated with no dose limiting toxicities (DLTs). The recommended dose for the combination was XL184 (cabozantinib) 40 mg daily, nivolumab 3 mg/kg every 2 weeks from part 1 of the study, while XL184 (cabozantinib) 40 mg daily, nivolumab 3 mg/kg every 2 weeks, and ipilimumab 1 mg/kg every 3 weeks (ipilimumab for up to four doses) was recommended from the part 2 of the study. The ORR seen with the combination was 33% in part 1 and 32% in part 2, with all the responses ongoing at the time of report.


The findings of studies cited above suggest that the combination of immune checkpoint inhibitors with XL184 (cabozantinib) is well tolerated. However, some potential overlapping toxicities might include fatigue, rash, diarrhea, and elevated lipase. There is only one reported case of heart failure and one case of autoimmune hemolytic anemia in a phase 2 XL184 (cabozantinib) study (Chan *et al.*, 2017).

This study utilizes ORR as the primary endpoint. ORR is clinically relevant since traditional NET therapies have low response rates and there is an unmet medical need to improve response rate. This is particularly important for patient with widely metastatic disease and visceral crisis. We hypothesize that this combination can potentially alter the composition of the tumor microenvironment favorably to improve its responsiveness to immunotherapy.

### 2.4 Correlative Studies Background

A series of correlative studies are proposed to examine the impact of the multikinase inhibitor XL184 (cabozantinib) on biomarkers within the tumor microenvironment and systemically. The primary scientific objectives are to perform Next Generation exome sequencing on pretreatment biopsy and RNA sequencing on pretreatment and on-treatment biopsies for molecular characterization of the neuroendocrine carcinomas.

In addition to these integrated biomarkers, we will assess a number of exploratory biomarkers. like tumor infiltration by CD8+ T cells, MDSC, TAM, and PD-L1 expression in the context of correlative laboratory studies. Infiltrating lymphocytes will be compared in the tumor microenvironment before and after exposure to XL184 (cabozantinib), nivolumab, and ipilimumab. These are based on the rationale that (1) patients with greater PD-L1 expression or antigen presenting capacity (as measured by MHC expression) will have a better response to immunotherapy; (2) tumors with high infiltration with MDSC and TAM respond poorly to checkpoint inhibition.

These correlative studies will help us better understand the molecular composition of the neuroendocrine tumors, mechanism(s) underlying the roles of MET, AXL, TYRO3, VEGF in modulating tumor immunity, and possibly help identify biomarkers that may predict response to therapy in the context of this clinical trial. We hypothesize that patients receiving the combination of XL184 (cabozantinib), nivolumab, and ipilimumab will have increased CD8+ T cell infiltration of their tumors as compared to prior to exposure to these drugs. Further, we hypothesize that patients with increased CD8+ T cell infiltration will have a better clinical outcome.

2.4.1 Whole exome sequencing (WES) of tumor DNA and of matching germline DNA collected from peripheral blood

This is an integrated biomarker for the study. Next-Generation sequencing (NGS) of tumor DNA is crucial for molecular characterization of the poorly differentiated neuroendocrine carcinomas for better understanding of the disease biology and its treatment. Among the different approaches for NGS, WES of tumor DNA combined with that of germline DNA from a matching peripheral blood sample is the most informative and possibly cost-effective.


WES will provide a systematic analysis of the tumor genome of each patient, thus establishing genomic signatures for testing of their predictive and prognostic value. Tumor mutation burden (TMB) and microsatellite instability (MSI) will be assessed as part of the NGS. The WES output from the germline DNA will facilitate, in addition to providing novel candidate genes for outcome testing, identifying new genes associated with the side effects of the study drugs.

# 2.4.2 RNA sequencing

RNA sequencing will be used to compare gene expression patterns prior to and after exposure to the study drugs, XL184 (cabozantinib), nivolumab, and ipilimumab. This will help in better understanding of the disease biology and the effect of treatment on the behavior of disease and treatment emergent complications.

## 2.4.3 Tumor infiltrating CD8+ T cells

Various preclinical and early phase clinical studies have shown the impact of the multikinase inhibitor cabozantinib on the immune profile of the tumor microenvironment. The targets of cabozantinib like TYRO3, MER, and AXL have been implicated in promoting tumor immune suppression (Okunishi *et al.*, 2005; Coudriet *et al.*, 2010; Kwilas *et al.*, 2014). MEK inhibition can enhance T cell infiltration into tumors in murine models, limit their apoptosis and subsequently enhance the efficacy of immune checkpoint blockade.

In a mouse model, increased tumor infiltration by CD8+ T cells while reduced tumor infiltration by myeloid derived suppressor cells (MDSC) and tumor associated macrophages (TAM) creating an immune permissive environment was seen as a result of exposure to cabozantinib (Kwilas *et al.*, 2014).

We hypothesize that patients receiving the combination of cabozantinib, nivolumab and ipilimumab will have increased CD8+ T cell infiltration of their tumors as compared to prior to exposure to these drugs. Further, we hypothesize that patients with increased CD8+ T cell infiltration will have a better clinical outcome.

## 2.4.4 Tumor infiltrating MDSCs

Levels of immune suppressive MDSCs in the tumor microenvironment may impact the response to checkpoint inhibitors. We will compare the tumor infiltrating MDSCs before and after exposure to XL184 (cabozantinib), nivolumab, and ipilimumab. *In vitro* and *in vivo* models have shown increased expression of MHC-I, ICAM-1, Fas, calreticulin, as a result of exposure to XL184 (cabozantinib) that led to improved recognition and killing of cancer cells by T lymphocytes (Kwilas *et al.*, 2014). We hypothesize that treatment with the combination of XL184 (cabozantinib), nivolumab, and ipilimumab will decrease the MDSC infiltration in tumors as compared to prior to exposure to these drugs.


# 2.4.5 Tumor-associated macrophages

Tumor-associated macrophages (TAM) are known to exert an immune suppressive effect in the tumor microenvironment. MET signaling has been shown to suppress the inflammatory response of macrophages as well as the activation and function of dendritic cells (Kwilas *et al.*, 2014). In a mouse model reduced tumor infiltration by TAM helped create an immune permissive environment as a result of exposure to XL184 (cabozantinib). We will compare the TAM in the tumor microenvironment before and after exposure to XL184 (cabozantinib), nivolumab, and ipilimumab. We hypothesize that treatment with the study drugs will decrease the extent of TAM in tumors as compared to prior to exposure to these drugs.

### 2.4.6 PD-L1 expression on tumor and immune cells

Tumors that have high expression of PD-L1 have been noted to have better response to immune checkpoint inhibitors (Chen *et al.*, 2018; Yi *et al.*, 2018). We will study the expression of PD-L1 in the tumors before and after exposure to the drugs XL184 (cabozantinib), nivolumab, and ipilimumab.


#### 3. PATIENT SELECTION

### 3.1 Eligibility Criteria

- 3.1.1 Patients must have metastatic, histologically confirmed poorly-differentiated neuroendocrine neoplasms per 2018 WHO classification, with the exception of small cell lung cancer and Merkel cell carcinoma. All variations of poorly differentiated neuroendocrine carcinoma (small cell, large cell and mixed cells) are eligible.
- 3.1.2 Failure of only one line of prior systemic cancer treatment.
- 3.1.3 Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
- 3.1.4 Patients must have lesions that can be safely biopsied and be willing to have a pretreatment and an on-treatment biopsy (after 1 month of treatment with the combination regimen) and a blood collection at baseline.
- 3.1.5 Prior systemic cancer therapy must have been completed at least 4 weeks prior to Cycle 1 Day 1 of treatment with the combination regimen
- 3.1.6 Age ≥18 years. Because no dosing or adverse event data are currently available on the use of XL184 (cabozantinib), nivolumab, and ipilimumab in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
- 3.1.7 ECOG performance status  $\leq 2$  (Karnofsky  $\geq 60\%$ , see Appendix A).
- 3.1.8 Patients must have adequate organ and marrow function as defined below:

| _ | leukocytes | ≥3,000/mcL |
|---|---|---|
| _ | absolute neutrophil count | ≥1,500/mcL without granulocyte-colony stimulating |
| | | (GCSF) factor support |
| _ | hemoglobin | ≥9 g/dL |
| _ | serum TSH | within institutional normal limits |
| _ | platelets | ≥100,000/mcL |
| _ | total bilirubin | $\leq$ 1.5 × institutional upper limit of normal (ULN); |
| | | ≤3.0 × ULN for patients with Gilbert's syndrome |
| _ | AST(SGOT)/ALT(SGPT) | ≤3 × institutional ULN |
| _ | alkaline phosphatase | $\leq$ 3.0 × institutional ULN; $\leq$ 5.0 × ULN with |
| | | documented bone metastases |
| _ | creatinine | ≤ institutional ULN |
| | | OR |
| _ | creatinine clearance (CrCl) | ≥50 mL/min/1.73 m <sup>2</sup> (using the Cockcroft-Gault |
| | | formula, see Appendix B) |
| _ | serum albumin | $\geq 2.8 \text{ g/dL}$ |


lipase
 <2.0 × ULN and no radiologic or clinical evidence of pancreatitis</li>

urine protein/creatinine ratio (UPCR)

≤1 mg protein/mg creatinine

 serum phosphorus, calcium, magnesium, and potassium

within institutional normal limits

prothrombin time (PT)/International
 Normalized Ratio (INR) and partial
 thromboplestin time (PTT) test

thromboplastin time (PTT) test  $<1.3 \times ULN$ 

- 3.1.9 Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy utilizing agents that do not strongly induce or inhibit cytochrome P450 (CYP) 3A4 with undetectable viral load within 6 months prior to study registration are eligible for this trial.
- 3.1.10 For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
- 3.1.11 Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
- 3.1.12 Patients with **treated brain metastases** are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and are off steroid support for at least 4 weeks after treatment for metastases is complete and within 28 days prior to the first dose of study treatment. Radiotherapy should have been stopped at least 4 weeks prior to study registration. Brain surgery should not have occurred within 3 months of study registration to be eligible.
- 3.1.13 Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
- 3.1.14 The effects of XL184 (cabozantinib), nivolumab, and ipilimumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of study therapy. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity: 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study therapy. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of <1% per year. Men who receive study therapy and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of study therapy. Women who


are not of childbearing potential (*i.e.*, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.

WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level <40 mIU/mL.

WOCBP and men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 5 and 7 months, respectively, after the last dose of study therapy. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) must inform the treating physician immediately.

- 3.1.15 Patients must be able to swallow tablets
- 3.1.16 Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

### 3.2 Exclusion Criteria

- 3.2.1 Patients must not require systemic corticosteroids treatment (≥10 mg/day prednisone equivalents) or other immunosuppressive medications within 28 days prior to study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg/day prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids in patients with adrenal insufficiency are permitted, even if ≥10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted, as is steroid pre-medication for contrast allergy.
- 3.2.2 Patients must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell costimulation or immune checkpoint pathways.


3.2.3 Patients must not have had prior treatment with XL184 (cabozantinib), or any MET-targeting TKI, or any MET-targeting monoclonal antibody (MetMAb), such as onartuzumab.

- 3.2.4 Patients must not have received radiation therapy to any part of the body within 28 days
- 3.2.5 Patients must not have clinically relevant, ongoing complications from prior radiation therapy. No radiation therapy is allowed while the patient is on study. Palliative radiation therapy, if needed, should be completed at least 28 days prior to enrollment into the study as described above.
- 3.2.6 Patients must not require concomitant treatment with oral anticoagulants (*e.g.*, warfarin, direct thrombin, and Factor Xa inhibitors) or platelet inhibitors (*e.g.*, clopidogrel). The following anticoagulants are allowed:
  - Low-dose aspirin for cardioprotection (per local applicable guidelines),
  - Low-dose low molecular weight heparins (LMWH),
  - Therapeutic doses of LMWH are allowed in patients without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before the first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
- 3.2.7 Patients must not have had major surgery (e.g., GI surgery or removal or biopsy of brain metastasis) within 4 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment and from minor surgery (e.g., simple excision or tooth extraction) at least 10 days before the first dose. Patients with clinically relevant ongoing complications from prior surgery are not eligible.
- 3.2.8 Patients must not have received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (*e.g.*, cytokines or antibodies) within 4 weeks, or nitrosoureas/ mitomycin C within 4 weeks, before the first dose of study treatment. Patients may continue on bone-modifying agents (denosumab or bisphosphonates) with caution.
- 3.2.9 Patients who have not recovered to baseline from adverse events due to prior anti-cancer therapy (*i.e.*, have residual toxicities > Grade 1) according to Common Terminology Criteria for Adverse Events (CTCAE) v0.5 unless the AEs are clinically nonsignificant and/or stable on supportive therapy, with the exception of alopecia.
- 3.2.10 Patients who are receiving any other investigational agents. Patients must not have received any other type of investigational agent within 4 weeks before the first dose of study treatment to be eligible.


3.2.11 Patients must not have a corrected QT interval calculated by the Fridericia formula (QTcF) >500 msec by electrocardiogram (EKG) within 28 days before the first dose of study treatment.

Note: If a single EKG shows a QTcF with an absolute value >500 msec, two additional EKGs at intervals of approximately 3 min must be performed within 30 min after the initial EKG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

- 3.2.12 Patients should not have known, untreated brain metastases or leptomeningeal metastases because of poor prognosis and concerns that progressive neurologic dysfunction could confound the evaluation of neurologic and other adverse events.
- 3.2.13 History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
- 3.2.14 Patients must not have a history of severe hypersensitivity reactions to any monoclonal antibodies.
- 3.2.15 Patients must not require concomitant treatment with strong CYP3A4 inducers (*e.g.*, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, or St. John's Wort). Because lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, patients will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.

Appendix C contains a patient clinical trial wallet card that can be given to patients.

- 3.2.16 Patients must not have uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:
  - Cardiovascular disorders:
    - o Congestive heart failure New York Heart Association (NYHA) Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    - Uncontrolled hypertension defined as sustained blood pressure (BP) >140 mm Hg systolic or >90 mm Hg diastolic despite optimal antihypertensive treatment within seven days prior to the first dose of study treatment.
    - Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis [DVT], pulmonary embolism [PE]) within 6 months before first dose.
  - GI disorders including those associated with a high risk of perforation or fistula formation:
    - o The patient has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute

obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

- O Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Complete healing of an intra-abdominal abscess must be confirmed before first dose.
- Clinically significant hematuria, hematemesis, or hemoptysis or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.
- Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
- Lesions invading or encasing any major blood vessels.
- Other clinically significant disorders that would preclude safe study participation.
  - o Serious non-healing wound/ulcer/bone fracture.
  - o Uncompensated/symptomatic hypothyroidism.
  - o Moderate to severe hepatic impairment (Child-Pugh B or C).
- 3.2.17 Patients with psychiatric illness/social situations that would limit compliance with study requirements.
- 3.2.18 Pregnant women are excluded from this study because XL184 (cabozantinib) has the potential for teratogenic or abortifacient effects, and the effects of nivolumab and ipilimumab on the developing fetus are not well known. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother, breastfeeding must be discontinued if the mother is treated with XL184 (cabozantinib), nivolumab, or ipilimumab.
- 3.2.19 Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including high dose systemic corticosteroids, should be excluded. These include but are not limited to: immune-related neurologic disease, such as multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, or myasthenia gravis; systemic autoimmune disease such as Systemic Lupus Erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, or autoimmune hepatitis. Patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, type I diabetes mellitus (DM), or endocrine deficiencies (e.g., thyroiditis) managed with replacement hormones, including physiologic corticosteroids, are eligible.

Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication, and patients with positive serology, (e.g., antinuclear antibodies (ANA) or anti-thyroid antibodies) should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.


#### 3.3 Inclusion of Women and Minorities

NIH policy requires that women and members of minority groups and their subpopulations be included in all NIH-supported biomedical and behavioral research projects involving NIH-defined clinical research unless a clear and compelling rationale and justification establishes to the satisfaction of the funding Institute & Center (IC) Director that inclusion is inappropriate with respect to the health of the subjects or the purpose of the research. Exclusion under other circumstances must be designated by the Director, NIH, upon the recommendation of an IC Director based on a compelling rationale and justification. Cost is not an acceptable reason for exclusion except when the study would duplicate data from other sources. Women of childbearing potential should not be routinely excluded from participation in clinical research. Please see http://grants.nih.gov/grants/funding/phs398/phs398.pdf.

Please refer to the table in Section 9.2 for the planned distribution of patients by sex, race, and ethnicity.


#### 4. REGISTRATION PROCEDURES

# 4.1 Investigator and Research Associate Registration with CTEP

Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all individuals contributing to NCI-sponsored trials to register and to renew their registration annually. To register, all individuals must obtain a Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) account at <a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>. In addition, persons with a registration type of Investigator (IVR), Non-Physician Investigator (NPIVR), or Associate Plus (AP) (*i.e.*, clinical site staff requiring write access to Oncology Patient Enrollment Network (OPEN), Rave, or acting as a primary site contact) must complete their annual registration using CTEP's web-based Registration and Credential Repository (RCR) at <a href="https://ctepcore.nci.nih.gov/rcr">https://ctepcore.nci.nih.gov/rcr</a>.

RCR utilizes five person registration types.

- IVR: MD, DO, or international equivalent,
- NPIVR: advanced practice providers (e.g., NP or PA) or graduate level researchers (e.g., PhD),
- AP: clinical site staff (e.g., RN or CRA) with data entry access to CTSU applications (e.g., Roster Update Management System [RUMS], OPEN, Rave,),
- Associate (A): other clinical site staff involved in the conduct of NCI-sponsored trials, and
- Associate Basic (AB): individuals (e.g., pharmaceutical company employees) with limited access to NCI-supported systems.

RCR requires the following registration documents:

| Documentation Required | IVR | NPIVR | AP | A | AB |
|---|---|---|---|---|---|
| FDA Form 1572 | ✓ | ✓ | | | |
| Financial Disclosure Form | <b>✓</b> | ✓ | <b>✓</b> | | |
| NCI Biosketch (education, training, employment, license, | <b>√</b> | ✓ | <b>√</b> | | |
| and certification) | | | | | |
| GCP training | <b>√</b> | ✓ | <b>√</b> | | |
| Agent Shipment Form (if applicable) | <b>√</b> | | | | |
| CV (optional) | <b>✓</b> | ✓ | <b>√</b> | | |

An active CTEP-IAM user account and appropriate RCR registration is required to access all CTEP and Cancer Trials Support Unit (CTSU) websites and applications. In addition, IVRs and NPIVRs must list all clinical practice sites and Institutional Review Boards (IRBs) covering their practice sites on the FDA Form 1572 in RCR to allow the following:

1. Addition to a site roster,


- 2. Assign the treating, credit, consenting, or drug shipment (IVR only) tasks in OPEN,
- 3. Act as the site-protocol Principal Investigator (PI) on the IRB approval.

In addition, all investigators act as the Site-Protocol PI, consenting/treating/drug shipment, must be rostered at the enrolling site with a participating organization (*i.e.*, Alliance).

Additional information is located on the CTEP website at <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR Help Desk by email at RCRHelpDesk@nih.gov.

# 4.2 Site Registration

This study is supported by the NCI Cancer Trials Support Unit (CTSU).

# IRB Approval

Sites participating with the NCI Central Institutional Review Board (NCI CIRB) must submit the Study Specific Worksheet for Local Context (SSW) to the CIRB using IRB Manager to indicate their intent to open the study locally. The NCI CIRB's approval of the SSW is automatically communicated to the CTSU Regulatory Office, but sites are required to contact the CTSU Regulatory Office at <a href="https://creativecommunicates/creat

Sites using their local IRB or REB must submit their approval to the CTSU Regulatory Office using the Regulatory Submission Portal located in the Regulatory section of the CTSU website. Acceptable documentation of local IRB/REB approval includes:

- Local IRB documentation,
- IRB-signed CTSU IRB Certification Form, and/or
- Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form.

In addition, the Site-Protocol PI (*i.e.*, the investigator on the IRB/REB approval) must meet the following five criteria to complete processing of the IRB/REB approval record:

- Holds an Active CTEP status,
- Rostered at the site on the IRB/REB approval (applies to US and Canadian sites only) and on at least one participating roster,
- If using NCI CIRB, rostered on the NCI CIRB Signatory record,
- Includes the IRB number of the IRB providing approval in the Form FDA 1572 in the RCR profile, and
- Holds the appropriate CTEP registration type for the protocol.

# **Additional Requirements**

Additional requirements to obtain an approved site registration status include:


• An active Federalwide Assurance (FWA) number,

- An active roster affiliation with the Lead Protocol Organization (LPO) or a Participating Organization, and
- Compliance with all protocol-specific requirements (PSRs).

# 4.2.1 Downloading Regulatory Documents

Download the site registration forms from the protocol-specific page located on the CTSU members' website. Permission to view and download this protocol and its supporting documents is restricted to institutions and their associated investigators and staff on a participating roster. To view/download site registration forms:

- Log in to the CTSU members' website (https://www.ctsu.org),
- Click on *Protocols* in the upper left of the screen
  - o Enter the protocol number in the search field at the top of the protocol tree, or
  - Click on the By Lead Organization folder to expand, then select *LAO-MD017*, and protocol number *10315*,
- Click on *Documents*, *Protocol Related Documents*, and use the *Document Type* filter and select *Site Registration* to download and complete the forms provided. (Note: For sites under the CIRB, IRB data will load automatically to the CTSU.)

# 4.2.2 <u>Submitting Regulatory Documents</u>

Submit required forms and documents to the CTSU Regulatory Office using the Regulatory Submission Portal on the CTSU members' website.

To access the Regulatory Submission Portal, log on to the CTSU members' website, go to the *Regulatory* section, and select *Regulatory Submission*.

# **Delegation of Tasks Log (DTL)**

Each site must complete a protocol-specific DTL using the DTL application which is accessible via the Delegation Log link on the CTSU members' website or directly at <a href="https://dtl.ctsu.org">https://dtl.ctsu.org</a>. The Clinical Investigator (CI) is required to review and electronically sign the DTL prior to the site receiving an approved site registration status and enrolling patients to the study. To maintain an approved site registration status the CI must re-sign the DTL at least annually and when a new version of the DTL is released; and activate new task assignments requiring CI sign-off. Any individual at the enrolling site on a participating roster may initiate the site DTL. Once the DTL is submitted for CI approval, only the designated DTL Administrators or the CI may update the DTL. Instructions on completing the DTL are available in the Help Topics button in the DTL


application and describes DTL task assignments, CI signature, and CTEP registration requirements, as well as include a Master Task List.

The DTL for this study has training requirements as follows:

All staff assigned the Rave CRA task on the DTL for this study must complete the *Theradex Specimen Tracking System (STS) Training* course.

1. The training is a one-time only requirement per individual. If an individual has previously completed the training for another ETCTN study with the same course requirement, the training does not need to be completed again. However, new versions of the Specimen Tracking System may require new training.

A task-related training requirement is satisfied by completing the course in the Compliance, Learning, and SOP Solutions (CLASS) application at <a href="https://classlms.org">https://classlms.org</a>; until that takes place, the task assignment will remain in a Pending status.

When a Rave CRA is assigned the task on an ETCTN DTL, the system will check to see
if they have completed the appropriate course, and if not, they will be automatically
enrolled in the course. They will receive an enrollment email from
<u>CLASSHelpDesk@westat.com</u> that will include instructions on how to access the course.

When an assignee completes the necessary course, their completion will be automatically communicated from CLASS to the DTL application and the task status will go to Active or Awaiting CI Approval, depending on the situation (please allow up to four hours for this to happen). The DTL cannot be submitted for CI sign-off until the minimum number of persons are assigned to the task(s) and have met all task requirements including any training requirements.

# 4.2.3 Checking Site Registration Status

You can verify your site's registration status on the members' side of the CTSU website.

- Log on to the CTSU members' website
- Click on *Regulatory* at the top of your screen
- Click on Site Registration
- Enter your 5-character CTEP Institution Code and click on Go

Note: The status shown only reflects institutional compliance with site registration requirements as outlined above. It does not reflect compliance with protocol requirements for individuals participating on the protocol or the enrolling investigator's status with the NCI or their affiliated networks.

#### 4.3 Patient Registration


## 4.3.1 OPEN / IWRS

The Oncology Patient Enrollment Network (OPEN) is a web-based registration system available on a 24/7 basis. OPEN is integrated with CTSU regulatory and roster data and with the Lead Protocol Organization (LPOs) registration/randomization systems or Theradex Interactive Web Response System (IWRS) for retrieval of patient registration/randomization assignment. OPEN will populate the patient enrollment data in NCI's clinical data management system, Medidata Rave.

# Requirements for OPEN access:

- A valid CTEP-IAM account.
- To perform enrollments or request slot reservations: Be on an LPO roster, ETCTN Corresponding roster, or Participating Organization roster with the role of Registrar. Registrars must hold a minimum of an AP registration type.
- Have an approved site registration for a protocol prior to patient enrollment.

To assign an Investigator (IVR) or Non-Physician Investigator (NPIVR) as the treating, crediting, consenting, drug shipment (IVR only), or receiving investigator for a patient transfer in OPEN, the IVR or NPIVR must list the IRB number used on the site's IRB approval on their Form FDA 1572 in RCR.

Prior to accessing OPEN, site staff should verify the following:

- Patient has met all eligibility criteria within the protocol stated timeframes, and
- All patients have signed an appropriate consent form and HIPAA authorization form (if applicable).

Note: The OPEN system will provide the site with a printable confirmation of registration and treatment information. Please print this confirmation for your records.

Access OPEN at <a href="https://open.ctsu.org">https://open.ctsu.org</a> or from the OPEN link on the CTSU members' website. Further instructional information is in the OPEN section of the CTSU website at <a href="https://www.ctsu.org">https://open.ctsu.org</a>. For any additional questions, contact the CTSU Help Desk at 1-888-823-5923 or <a href="mailto:ctsu.org">ctsucontact@westat.com</a>.

Patient enrollment for this study will be facilitated using the Slot Reservation System in conjunction with the registration system in OPEN. Prior to discussing protocol entry with the patient, all site staff must use the CTSU OPEN Slot Reservation System to ensure that a slot on the protocol is available to the patient. Once a slot reservation confirmation is obtained, site staff may then proceed to enroll the patient to this study.

# 4.3.2 OPEN/IWRS Questions?


Further instructional information on OPEN is provided on the OPEN link of the CTSU website at <a href="https://www.ctsu.org">https://www.ctsu.org</a> or at <a href="https://open.ctsu.org">https://open.ctsu.org</a>. For any additional questions contact the CTSU Help Desk at 1-888-823-5923 or <a href="ctsucontact@westat.com">ctsucontact@westat.com</a>.

Theradex has developed a Slot Reservations and Cohort Management User Guide, which is available on the Theradex website: <a href="http://www.theradex.com/clinicalTechnologies/?National-Cancer-Institute-NCI-11">http://www.theradex.com/clinicalTechnologies/?National-Cancer-Institute-NCI-11</a>. This link to the Theradex website is also on the CTSU website OPEN tab. For questions about the use of IWRS for slot reservations, contact the Theradex Helpdesk at 609-619-7862 or Theradex main number 609-799-7580; <a href="mailto:CTMSSupport@theradex.com">CTMSSupport@theradex.com</a>.

# 4.4 General Guidelines

Following registration, patients should begin protocol treatment within a minimum of 7 days and no more than 14 days. Issues that would cause treatment delays should be discussed with the Principal Investigator. If a patient does not receive protocol therapy following registration, the patient's registration on the study may be canceled. The Study Coordinator should be notified of cancellations as soon as possible.


# 5. BIOMARKER, CORRELATIVE, AND SPECIAL STUDIES

# 5.1 Summary Table for Specimen Collection.

All specimen collections on this study are mandatory.

| <b>Time Point</b> | Specimen | Send Specimens To: |
|---|---|---|
| Pre-treatment (B | Pre-treatment (Baseline) | |
| | • 4 tissue cores in formalin <sup>1</sup> | EET Biobank |
| | 10 mL blood in cfDNA Streck | |
| Cycle 2 (within Days 28 – 35) | | |
| | • 4 tissue cores in formalin <sup>1</sup> | EET Biobank |
| <sup>1</sup> A a copy of the radiology and operative reports from the tissue removal procedure and the | | |

<sup>&</sup>lt;sup>1</sup>A a copy of the radiology and operative reports from the tissue removal procedure and the diagnostic anatomic pathology report must be sent with the tissue to the EET Biobank. When completed, upload the corresponding pathology reports to Rave.

# 5.2 Summary Table(s) for Interventional Radiologist for Research Biopsies

| Biopsy # | Biopsy #: 1 | | | |
|---|---|---|---|---|
| Trial Tin | Trial Time Point: Pre-treatment (Baseline) | | | |
| IR Biops | IR Biopsy Definition: Research – No Clinical Impact (All cores from a single biopsy | | | |
| procedure | e impact research | goals, but do not | directly impact pa | tient care or benefit the patient.) |
| Core | Use in the | Biomarker | Tumor | Post-Biopsy Processing |
| Priority | Trial | Name(s) | Content<br>Required | |
| 1 | Integrated | Whole exome sequencing | >50% | Formalin-fixed |
| 2 | Integrated | RNA<br>sequencing | >50% | Formalin-fixed |
| 3 | Exploratory | Tumor infiltrating lymphocytes, tumor infiltrating MDSC | >50% | Formalin-fixed |
| 4 | Exploratory | Tumor<br>associated<br>macrophages,<br>PD-L1<br>expression | >50% | Formalin-fixed |


| Rioney # | . 2 | | | |
|---|---|---|---|---|
| | Biopsy #: 2 | | | |
| | Trial Time Point: Cycle 2 (within Days 28 – 35) | | | |
| _ | <b>IR Biopsy Definition:</b> Research – No Clinical Impact (All cores from a single biopsy | | | |
| procedure | e impact research | n goals, but do not | directly impact | patient care or benefit the patient.) |
| Core | Use in the | Biomarker | Tumor | <b>Post-Biopsy Processing</b> |
| Priority | Trial | Name(s) | Content | |
| | | | Required | |
| 1 | Integrated | RNA | >50% | Formalin-fixed |
| | | sequencing | | |
| 2 | Exploratory | Tumor | >50% | Formalin-fixed |
| | | infiltrating | | |
| | | lymphocytes | | |
| 3 | Exploratory | Tumor | >50% | Formalin-fixed |
| | 1 5 | infiltrating | | |
| | | MDSCs, | | |
| | | Tumor- | | |
| | | associated | | |
| | | macrophages | | |
| 4 | Exploratory | PD-L1 | >50% | Formalin-fixed |
| | | expression | | |

**Note:** Pre-biopsy assessments will be reported and tracked through a trial-specific case report form (CRF) within the CTEP Medidata Rave system (see Appendix D).

# 5.3 Specimen Procurement Kits and Scheduling

# 5.3.1 Specimen Procurement Kits

Kits for the collection and shipment of specimens to the EET Biobankcan be ordered online via the Kit Management system: (<a href="https://ricapps.nationwidechildrens.org/KitManagement">https://ricapps.nationwidechildrens.org/KitManagement</a>).

Users at the clinical sites will need to set up an account in the Kit Management system and select a specific clinical trial protocol to request a kit. Please note that protocol may include more than one type of kit. Each user may order two kit types per protocol per day (daily max = 6 kits). Kits are shipped ground, so please allow 5-7 days for receipt. A complete list of kit contents for each kit type is located on the Kit Management system website.

<u>Note</u>: Kits or supplies are only provided for specimens shipped to the Biorepository. Institutional supplies must be used for all other specimen collection and processing.

# 5.3.2 Scheduling of Specimen Collections

Please adhere to the following guidelines when scheduling procedures to collect tissue:

• Tumor tissue specimens collected during biopsy procedures and fixed in formalin must be shipped on the same day of collection.


• Tissue in formalin can be collected Monday through Wednesday and shipped overnight for arrival on Tuesday through Thursday at the EET Biobank at Nationwide Children's Hospital.

• Fresh blood specimens may be collected and shipped Monday through Friday.

# 5.4 Specimen Tracking System Instructions

This Study will use the ETCTN Specimen Tracking System (STS).

- All biospecimens collected for this trial must be submitted using the ETCTN STS unless otherwise noted.
- The system is accessed through Rave user roles: "Rave CRA" and "Rave CRA (Labadmin)" for data entry at the treating institutions. The "Biorepository" role is assigned to users receiving the specimens for processing and storage at reference labs and the NCI Early-Phase and Experimental Clinical Trials Biospecimen Bank (EET Biobank, formerly known as the EET Biobank).

Important: Failure to complete required fields in STS may result in a delay in sample processing. Any case reimbursements associated with sample submissions will not be credited if samples requiring STS submission are not logged into STS.

Detailed instructions on use of the STS can be found below.

# 5.4.1 Specimen Tracking System Overview and Enrollment Instructions

For the ETCTN STS, the following information will be requested:

- Protocol Number
- Investigator Identification
  - o Institution and affiliate name
  - o Investigator's name
- Eligibility Verification: Patients must meet all the eligibility requirements listed in Section 0.
- Additional Requirements:
  - o Patients must provide a signed and dated, written informed consent form.

Upon enrolling a patient, IWRS will communicate with OPEN, assigning two separate and unique identification numbers to the patient, a Universal patient ID (UPID) and a Treatment patient ID. The UPID is associated with the patient and used each and every time the patient engages with the portion of this protocol that uses the ETCTN Specimen Tracking System. The UPID contains no information or link to the treatment protocol. IWRS will maintain an association between the UPID for ETCTN biobanking and molecular characterization and any treatment protocols the patient participates in, thereby allowing analysis of the molecular characterization results with the clinical data.


Immediately following enrollment, the institutional anatomical pathology report for the diagnosis under which the patient is being enrolled must be uploaded into Rave. The report must include the surgical pathology ID (SPID), collection date, block number, and the IWRS-assigned UPID and patient study ID for this trial. For newly acquired biopsies, the radiology and operative report(s) must also be uploaded into Rave. <u>Important</u>: Remove any personally identifying information, including, but not limited to, the patient's name, initials, medical record number, and patient contact information from the institutional pathology report prior to submission.

Additionally, please note that the STS software creates pop-up windows when reports are generated, so you will need to enable pop-ups within your web browser while using the software.

For questions regarding the Specimen Tracking System, please contact the Theradex Help Desk at CTMSSupport@theradex.com.

A shipping manifest **must** be included with all sample submissions.

# 5.4.2 Specimen Labeling

# 5.4.2.1 Blood Specimen Labels

Include the following on blood specimens (including whole blood and frozen, processed blood products – like serum and plasma):

- Patient Study ID
- Universal Patient ID (UPID)
- Specimen ID (automatically generated by Rave)
- Time point
- Specimen type (*e.g.*, blood, serum)
- Collection date [if the study also requires recording the collection time on the label, include the time] (to be added by hand)

# 5.4.2.2 Tissue Specimen Labels

Include the following on all tissue specimens or containers (e.g., formalin jar):

- Patient Study ID
- Universal Patient ID (UPID)
- Specimen ID (automatically generated by Rave)
- Time point
- Specimen type (*e.g.*, formalin-fixed paraffin-embedded [FFPE] Block, Formalin Fixed Tissue, Fresh Tissue in Media, *etc.*)
- Tissue type (P for primary, M for metastatic or N for normal)
- Surgical pathology ID (SPID) number
- Block number from the corresponding pathology report (archival only)
- Collection date and time (to be added by hand)


# 5.4.2.3 Example of Specimen Label

The following image is an example of a tissue specimen label printed on a standard Avery label that is 1" high and 2.625" wide.



The QR code in the above example is for the Specimen ID shown on the second line. **NOTE:** The QR code label is currently under development at Theradex as of 31-Aug-2018; therefore, labels generated by the STS for this study may not include a QR code.

The second line item from the end includes four data points joined together:

- 1. Tissue only: Primary (P), Metastatic (M), Normal (N) tissue indicated at the beginning of the specimen ID; this field is blank if not relevant (e.g., for blood)
- 2. Block ID or blank if not relevant
- 3. SPID (Surgical Pathology ID) or blank if none
- 4. The last alpha-numeric code is protocol specific and is only included if the protocol requires an additional special code classification

The last line on the example label is for the handwritten date and optional time.

#### 5.4.3 Overview of Process at Treating Site

#### 5.4.3.1 OPEN Registration

All registrations will be performed using the Oncology Patient Enrollment Network (OPEN) system. OPEN communicates automatically with the Interactive Web Response System (IWRS) which handles identifier assignments, any study randomization, and any prescribed slot assignments. If specimen analysis is required to determine eligibility, the protocol will be setup with multi-step registration.

Registration without eligibility specimen analysis:

- 1. Site enters registration data into OPEN during one or more steps.
- 2. IWRS receives data from OPEN, generates the Patient Study ID and the Universal Patient ID, both of which are sent back to OPEN.
- 3. IWRS sends all applicable registration data directly to Rave at the end of the final registration step.


Any data entry errors made during enrollment should be corrected in Rave.

# 5.4.3.2 Rave Specimen Tracking Process Steps

**Step 1**: Complete the **Histology and Disease** form (but do not upload reports until a specimen label can be applied to them) and the Baseline forms regarding **Prior Therapies**. Enter the initial clinical specimen data:

• **Specimen Tracking Enrollment** CRF: Enter Time Point, Specimen Category, Specimen Type, Block number, Tissue type, Surgical Path ID, and number of labels needed (include extra labels to apply to reports to be uploaded). CRF generates unique Specimen ID.

**Step 2**: Print labels using report in EDC and collect specimen.

- Label specimen containers and write collection date and time on each label.
- After collection, store labeled specimens as described in Section 5.4.2.
- Apply an extra specimen label to <u>each</u> report before scanning. Return to the **Histology** and **Disease** form to upload any initial Pathology, Radiology, Molecular Reports (up to 4), Surgical (or Operative) reports and Pathology Verification form (when applicable). Return to **Specimen Tracking Enrollment** CRF to upload any molecular report (one per specimen) and/or specimen specific pathology or related report (one per specimen). Uploaded reports should have protected health information (PHI) data, like name, mailing address, medical record number or social security number (SSN), redacted. Do not redact SPID, block number or relevant dates, and include the UPID and patient study ID on each document.

# **Step 3**: Complete specimen data entry.

• **Specimen Transmittal** Form: Enter collection date and time and other required specimen details.

**Step 4**: When ready to ship, enter shipment information.

- **Shipping Status** CRF: Enter tracking number, your contact information, recipient, number of containers and ship date once for the first specimen in a shipment.
- Copy Shipping CRF: Select additional specimens to add to an existing shipment referenced by the tracking number.

**Step 5**: Print shipping list report and prepare to ship.

- Print two copies of the shipping list, one to provide in the box, the other for your own records.
- Print pathology or other required reports to include in the box. Be sure the printed copy includes the specimen label.

# Step 6: Send email notification.

• For only one of the specimens in the shipment, click "Send Email Alert" checkbox on the **Shipping Status** CRF to email recipient.


**Step 7:** Ship the specimen(s).

# 5.5 Specimen Collection

# 5.5.1 Formalin-Fixed Tumor Biopsies

- 1. Label formalin-filled containers according to instructions in Section 5.4.2.
- 2. Obtain [number] 16-gauge or 18-gauge core needle biopsy specimens, and place one core in each cassette.
- 3. Snap the cassette lids closed and place cassettes into a formalin-filled pre-labeled container as soon as possible after collection to prevent air drying. Up to two cassettes may be placed in one formalin jar.
- 4. Secure the container lids and package containers into the shipping kit according to instructions in Section 5.6. Keep tissue in formalin jars at room temperature until shipment to the EET Biobank.

#### 5.5.2 Blood Collection

#### 5.5.2.1 Collection of Blood in cfDNA Streck Tube

- 1. Label one 10 mL cfDNA Streck tube according to the instructions in Section 5.4.2.
- 2. Collect 10 mL of blood into the pre-labeled tube and gently invert to mix. Note: blood must be thoroughly mixed to ensure preservation of specimen. [Include the following language if patients may have an indwelling catheter: heparin should be avoided in pre-collection flush procedures. If therapeutic heparin dosing contamination is a possibility, then venipuncture is recommended as a first choice collection method. If a cfDNA Streck tube immediately follows a heparin tube in the draw order, then collecting an EDTA tube as a waste tube prior to collection in the Streck Cell-Free DNA BCT is recommended.]
- 3. **After collection, blood in cfDNA Streck tubes should never be refrigerated,** as this will compromise the specimen. Blood collected in cfDNA Streck tubes is stable at room temperature.

# 5.6 Shipping Specimens from Clinical Site to the EET Biobank

# 5.6.1 General Shipping Information

Core biopsies that are fixed in formalin and fresh blood should be shipped as one shipment at ambient temperature, whenever possible. The same box sent with kit contents should be used to ship specimens to the EET Biobank. In winter months, please include extra insulation, such as bubble wrap, inside the shipping container.


For formalin-fixed biopsies, if the corresponding anatomical pathology report is not available at the time of shipment, then the surgical and/or radiology report must be uploaded to the ETCTN specimen tracking system and included in the package, or the specimen will not be processed.

# 5.6.2 Specimen Shipping Instructions

Tissue in formalin must be shipped on the day of collection. Collect and ship on Monday through Wednesday.

Fresh blood may be shipped on Monday through Friday. Please select "Saturday Delivery" when shipping fresh blood on a Friday.

# 5.6.2.1 Shipping Blood in an Ambient Shipper

- 1. Before packaging specimens, verify that each specimen is labeled according to the instructions above and that the lids of all primary receptacles containing liquid are tightly sealed.
- 2. Prepare the SAF-T-TEMP Gel Pak for shipment. **Note:** If contents of the Pak are crunchy, place Pak in a warm water bath until gel is smooth. **Do not refrigerate, freeze, or microwave.**
- 3. Place the SAF-T-TEMP Pak in bottom of insulated chest. **Note:** The insulated chest must be shipped inside the provided cardboard box(es).
- 4. Place the blood collection tubes in zip-lock bags.
- 5. Next, place blood into a biohazard envelope with absorbent material. Expel as much air as possible and seal the envelope securely.
- 6. Place the biohazard envelope into a Tyvek envelope. Expel as much air as possible and seal securely.
- 7. Place packaged blood collection tube(s) and a copy of the shipping manifest from the Sample Tracking System on top of SAF-T-TEMP Pak.
- 8. Place the lid on the insulated chest.
- 9. Close the outer flaps of the shipping box and tape shut.
- 10. Attach a shipping label to the top of the shipping container.
- 11. Attach an Exempt Human Specimen sticker to the side of the box.
- 12. Ship specimens via overnight courier to the address below. FedEx Priority Overnight is strongly recommended to prevent delays in package receipt.

# 5.6.2.2 Shipping Ambient Tissue and Blood in a Single-Chamber Kit

- 1. Before packaging specimens, verify that each specimen is labeled according to the instructions above and that the lids of all primary receptacles containing liquid are tightly sealed. Formalin jars should be wrapped in parafilm.
- 2. Place the specimens in zip-lock bags. Use a separate bag for each specimen type.
- 3. Place specimens into a biohazard envelope with absorbent material. Expel as much air as possible and seal the envelope securely.
- 4. Place the biohazard envelope into a Tyvek envelope. Expel as much air as possible and seal securely.


- 5. Place the specimen(s) and a copy of the shipping manifest and corresponding reports such as surgical or radiology reports into the insulated shipping container. In winter months, please include extra insulation, such as bubble wrap, inside the shipping container, to prevent specimens from freezing.
- 6. Place the lid on top of the container. Close the outer flaps and tape shut.
- 7. Attach a shipping label to the top of the shipping container.
- 8. Attach an Exempt Human Specimen sticker to the side of the container.
- 9. Ship specimens via overnight courier to the address below. FedEx Priority Overnight is strongly recommended to prevent delays in package receipt.

# 5.6.3 Shipping Address

Ship to the address below. Ship formalin-fixed and fresh blood specimens the same day of specimen collection. Do not ship specimens the day before a holiday.

EET Biobank2200 International Street

Columbus, OH 43228 PH: (614) 722-2865 FAX: (614) 722-2897

Email: BPCBank@nationwidechildrens.org

FedEx Priority Overnight service is very strongly preferred.

**NOTE:** The EET Biobank FedEx Account will not be provided to submitting institutions.

# 5.6.4 Contact Information for Assistance

For all queries, please use the contact information below:

**EET Biobank** 

Toll-free Phone: (614) 722-2865

E-mail: BPCBank@nationwidechildrens.org

# 5.7 Shipping of Specimens from Clinical Site to Other Laboratories

N/A

#### Biomarker Plan


List of Biomarker Assays in Order of Priority

| Priority | Biomarker<br>Name | Assay<br>(CLIA: Y/N) | Use in the Trial and<br>Purpose | Specimens<br>Tested | Collection Time<br>Points | Mandatory<br>or<br>Optional | Assay Laboratory and<br>Lab PI |
|---|---|---|---|---|---|---|---|
| Tissue-based | l Biomarkers | | | | | | |
| 1 | Whole Exome<br>Sequencing | WES CLIA: N | Integrated Molecular characterization of the tumors | Tissue | Pre-treatment<br>(Baseline) | M | MoCha, Frederick<br>National Laboratory for<br>Cancer Research<br>(FNLCR)<br>Chris Karlovich<br>chris.karlovich@nih.gov |
| 2 | RNA Seq | NGS<br>CLIA: N | Integrated Molecular characterization of the tumors | Tissue | Pre-treatment<br>(Baseline) and<br>Cycle 2 (within<br>Days 28 – 35) | M | MoCha, Frederick National Laboratory for Cancer Research (FNLCR) Chris Karlovich chris.karlovich@nih.gov |
| 3 | Tumor<br>Infiltrating<br>CD8+ T Cells | IHC<br>CLIA: N | Exploratory Compare the effect of treatment on the tumor microenvironment | Tissue | Pre-treatment<br>(Baseline) and<br>Cycle 2 (within<br>Days 28 – 35) | M | Wayne State University<br>Kang Chen, Ph.D.<br>kang@wayne.edu |
| 5 | Tumor<br>Infiltrating<br>MDSCs | IHC<br>CLIA: N | Exploratory Compare the effect of treatment on the tumor microenvironment | Tissue | Pre-treatment<br>(Baseline) and<br>Cycle 2 (within<br>Days 28 – 35) | M | Wayne State University<br>Kang Chen, Ph.D.<br>kang@wayne.edu |
| 6 | Tumor<br>Associated<br>Macrophages | IHC<br>CLIA: N | Exploratory Compare the effect of treatment on the tumor microenvironment | Tissue | Pre-treatment<br>(Baseline) and<br>Cycle 2 (within<br>Days 28 – 35) | M | Wayne State University<br>Kang Chen, Ph.D.<br>kang@wayne.edu |


| Priority | Biomarker<br>Name | Assay<br>(CLIA: Y/N) | Use in the Trial and<br>Purpose | Specimens<br>Tested | Collection Time<br>Points | Mandatory<br>or | Assay Laboratory and<br>Lab PI |
|---|---|---|---|---|---|---|---|
| | | | | | | Optional | |
| Tissue-based | Biomarkers | | | | | | |
| 7 | PD-L1 | IHC | Exploratory | Tissue | Pre-treatment | M | Wayne State University |
| | Expression on | | | | (Baseline) and | | Kang Chen, Ph.D. |
| | Tumor and | CLIA: N | Compare the effect of | | Cycle 2 (within | | kang@wayne.edu |
| | Immune Cells | | treatment on the | | Days 28 – 35) | | |
| | | Commercial | tumor | | • | | |
| | | Kit | microenvironment | | | | |
| Blood-based I | Biomarkers | | | | | | |
| 1 | Whole Exome | WES | Integrated | Whole Blood | Pre-treatment | M | MoCha, Frederick |
| | Sequencing | | | | (Baseline) | | National Laboratory for |
| | | CLIA: N | Molecular | 10 mL in Streck | | | Cancer Research |
| | | | characterization of the | tube | | | (FNLCR) |
| | | | tumors | | | | Chris Karlovich |
| | | | | | | | chris.karlovich@nih.gov |

# **5.8** Integrated Correlative Studies

# 5.8.1 Whole Exome Sequencing (WES)

# 5.8.1.1 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded. All FFPE blocks will be sectioned to generate an initial H&E-stained slide, and for nucleic acid extractions, additional RNase-free slides.

Whole blood collected in Streck tubes will be centrifuged to separate buffy coat and plasma and will be stored in a -80°C freezer.

DNA and RNA will be co-extracted from tumor tissue. The nucleic acids will be analyzed to determine concentration and quality. Aliquots of DNA and RNA will be shipped to the central sequencing laboratory for analysis.

# 5.8.1.2 Site Performing Correlative Study

WES will be conducted at the MoCha, Frederick National Laboratory for Cancer Research (FNLCR) under the supervision of Chris Karlovich, Ph.D. (chris.karlovich@nih.gov).

5.8.1.3 Shipment of Specimens from the EET Biobank to Site Performing Correlative Study

Specimens will be shipped from the EET Biobank to:

MoCha Lab, Frederick National Laboratory for Cancer Research (FNLCR) 1050 Boyles St. Bldg. 459, Rm. 125

Bldg. 459, Rm. 125 Frederick, MD 21702

Attn: Alyssa Chapman or Ruth Thornton

# 5.8.1.4 Contact information for notification of specimen shipment

Thomas Forbes, mochasamplereceiving@nih.gov

RNA Sequencing (RNAseq)

# 5.8.1.5 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded. All FFPE blocks will be sectioned to generate an initial H&E-stained slide, and for nucleic acid extractions, additional RNase-free slides.

DNA and RNA will be co-extracted from tumor tissue. The nucleic acids will be analyzed to determine concentration and quality. Aliquots of DNA and RNA will be shipped to the central sequencing laboratory for analysis.

# 5.8.1.6 Site Performing Correlative Study

RNAseq will be conducted at the MoCha, Frederick National Laboratory for Cancer Research (FNLCR) under the supervision of Chris Karlovich, Ph.D. (chris.karlovich@nih.gov).

# 5.8.1.7 Shipment of Specimens from the EET Biobank to Site Performing Correlative Study

Specimens will be shipped from the EET Biobank to:

MoCha Lab, Frederick National Laboratory for Cancer Research (FNLCR) 1050 Boyles St.
Bldg. 459, Rm. 125
Frederick, MD 21702

Attn: Alyssa Chapman or Ruth Thornton

# 5.8.1.8 Contact information for notification of specimen shipment

Thomas Forbes, mochasamplereceiving@nih.gov

## **5.9** Exploratory/Ancillary Correlative Studies

# 5.9.1 Tumor Infiltrating CD8+ T Cells

# 5.9.1.1 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded and sectioned. FFPE tumor tissue will be used to produce 20 unstained sections, cut at 5 micrometers thickness and mounted on glass slides. About 5 slides will be used for each exploratory assay.

# 5.9.1.2 Site Performing Correlative Study

This assay will be conducted at Wayne State University under the leadership of Kang Chen, Ph.D. Samples from EET Biobank should be shipped to address below:

Kang Chen 421 East Canfield Street, Room 2221 Detroit, MI 48202 Phone number: 313-578-4339

Email: kang@wayne.edu

# 5.9.2 Tumor Infiltrating MDSCs

# 5.9.2.1 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded and sectioned. FFPE tumor tissue will be used to produce 20 unstained sections, cut at 5 micrometers thickness and mounted on glass slides. About 5 slides will be used for each exploratory assay.

# 5.9.2.2 Site Performing Correlative Study

This assay will be conducted at Wayne State University under the leadership of Kang Chen, Ph.D. Samples from EET Biobank should be shipped to address below:

Kang Chen

421 East Canfield Street, Room 2221

Detroit, MI 48202

Phone number: 313-578-4339 Email: kang@wayne.edu

# 5.9.3 Tumor Associated Macrophages

#### 5.9.3.1 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded and sectioned. FFPE tumor tissue will be used to produce 20 unstained sections, cut at 5 micrometers thickness and mounted on glass slides. About 5 slides will be used for each exploratory assay.

# 5.9.3.2 Site Performing Correlative Study

This assay will be conducted at Wayne State University under the leadership of Kang Chen, Ph.D. Samples from EET Biobank should be shipped to address below:

Kang Chen

421 East Canfield Street, Room 2221

Detroit, MI 48202

Phone number: 313-578-4339 Email: <u>kang@wayne.edu</u>

# 5.9.4 PD-L1 Expression on Tumor and Immune Cells

#### 5.9.4.1 Specimens Receipt and Processing at the EET Biobank

Tumor tissue received in formalin will be paraffin-embedded and sectioned. FFPE tumor tissue will be used to produce 20 unstained sections, cut at 5 micrometers thickness and mounted on glass slides. About 5 slides will be used per each exploratory assay.

# 5.9.4.2 Site Performing Correlative Study

This assay will be conducted at Wayne State University under the leadership of Kang Chen, Ph.D. using a commercial kit. Samples from EET Biobank should be shipped to address below:

Kang Chen 421 East Canfield Street, Room 2221 Detroit, MI 48202

Phone number: 313-578-4339 Email: <u>kang@wayne.edu</u>

#### 6. TREATMENT PLAN

# 6.1 Agent Administration

Treatment will be administered on an outpatient basis. Reported adverse events and potential risks are described in Section 10. Appropriate dose modifications are described in Section 7. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

| | Regimen Description | | | | | |
|---|---|---|---|---|---|---|
| Cycles | Agent | Premedications; Precautions | Dose | Route | Schedule | Cycle<br>Length |
| 1-4 | XL184 (cabozantinib) | XL184 (cabozantinib) should be taken on an empty stomach. Patients should not eat for at least 2 hours before, and 1 hour after each dose. | 40 mg | PO | Days 1-21 | 21 days |
| 1-4 | Nivolumab | N/A | 3 mg/kg | IV | Day 1 of Cycles<br>1-4<br>(4 total doses) | (3 weeks) |
| | Ipilimumab | N/A | 1 mg/kg | IV | Day 1 of Cycles<br>1-4<br>(4 total doses) | |
| 5+ | XL184<br>(cabozantinib) | XL184 (cabozantinib) should be taken on an empty stomach. Patients should not eat for at least 2 hours before, and 1 hour after each dose. | 40 mg | РО | Days 1-28 | 28 days<br>(4 weeks) |
| DO O | Nivolumab | N/A | 480 mg | IV | Day 1of Cycles<br>5+ | |

PO = Oral; IV = Intravenous

Treatment will be continued until criteria for removal from the study are met (See Section 6.5 Duration of Therapy)

Screening and baseline biopsy will be done within 28 days prior to starting treatment.

Patients will receive XL184 (cabozantinib) 40 mg by mouth (PO) once daily. Nivolumab will be given at a dose of 3 mg/kg on Day 1 (±3 days) of each 3-week cycle for the first 4 cycles (12 weeks). Ipilimumab is to be administered at a dose of 1 mg/kg immediately following nivolumab administration on Day 1 of each 3-week cycle for the first 4 cycles. No more than four doses of ipilimumab should be administered.

Starting Cycle 5, patients will continue to take cabozantinib 40 mg PO daily and receive IV infusion of nivolumab 480 mg every 4 weeks. Treatment will be continued until criteria for removal from the study is met (See Section 6.5 Duration of Therapy). The study is projected to complete accrual in about 2 years. All patients will be followed until death unless consent has been withdrawn.

The frequency of nivolumab and ipilimumab infusion is supported by the label insert and prior studies, respectively (Nivolumab Package Insert, 2014; Ansell *et al.*, 2009). The dose level of XL184 (cabozantinib), in combination with nivolumab, and ipilimumab was selected as this was shown to be very well tolerated in this combination (Apolo *et al.*, 2017).

# 6.1.1 XL184 (cabozantinib)

Patients will receive XL184 (cabozantinib) PO at a dose of 40 mg once daily. XL184 (cabozantinib) must be taken on an empty stomach. Patients should be instructed not to eat for at least 2 hours before and at least 1 hour after taking XL184 (cabozantinib). Patients should be instructed to take their dose at approximately the same time every day. If a patient misses a dose, the dose may be taken later only if it is within 12 hours of when the missed dose should have been taken. The missed dose should not be made up if it is within 12 hours of the next scheduled dose. If a patient vomits after taking a dose, the dose should not be made up. The patient should be instructed to take the next dose at the regularly scheduled time.

XL184 (cabozantinib) tablets should be swallowed whole with at least 8 ounces of water. The tablets should not be crushed. Grapefruit, grapefruit juice, Seville oranges, and their products should be avoided by patients taking XL184 (cabozantinib). Patients will be asked to maintain a medication diary for each dose of medication (Appendix E). The medication diary should be returned to clinic staff at the end of each month.

Dose reductions and delays to manage toxicity are allowed under the guidelines in Section 7.1 below. XL184 (cabozantinib) administration will continue until disease progression or unacceptable toxicity.

#### 6.1.2 Nivolumab

Nivolumab will be given at a dose of 3 mg/kg on Day 1 ( $\pm 3$  days) of each 3-week cycle for the first 4 cycles (12 weeks). Starting with Cycle 5, nivolumab will be given every 4 weeks ( $\pm 3$  days) at a dose of 480 mg on Day 1 of each 4-week cycle. No dose modifications are allowed for Nivolumab. Nivolumab administration will continue until disease progression or unacceptable toxicity.

Nivolumab is to be administered as an approximate 30-minute IV infusion, using a volumetric pump with a 0.2-1.2 micron in-line filter. When the dose is based on patient weight (*i.e.*, mg/kg), nivolumab injection can be infused undiluted, or diluted with 0.9% normal saline or 5% dextrose in water to protein concentrations as low as 0.35 mg/mL. When the dose is fixed (*e.g.*, 480 mg flat dose), nivolumab injection can be infused undiluted or diluted so as not to exceed a total infusion volume of 160 mL. For patients weighing less than 40 kg, the total volume of infusion

must not exceed 4 mL per kg of patient weight. It is not to be administered as an IV push or bolus injection. At the end of the infusion, flush the line with a sufficient quantity of normal saline.

Nivolumab dosing calculations should be based on the actual body weight. If the patient's weight differs by >10% from the weight used to calculate the original dose, the dose may be recalculated. All doses should be rounded to the nearest milligram.

When infusions of ipilimumab and nivolumab are given on the same day, the preferred treatment is to give nivolumab followed by ipilimumab. Separate infusion bags and filters must be used for each drug. The infusion line must be flushed with normal saline between infusions.

Toxicity management should follow the guidelines and algorithms provided in Section 7 and Appendix E.

# 6.1.3 Ipilimumab

Ipilimumab is to be administered as an approximate 90-minute IV infusion at a dose of 1 mg/kg immediately following nivolumab administration on Day 1 of each 3-week cycle for the first 4 cycles (12 weeks), using a volumetric pump with a 0.2-1.2 micron in-line filter. The drug can be diluted with 0.9% normal saline for delivery or 5% dextrose in water, but the total drug concentration of the solution must stay within the range of 1 mg/mL to 4 mg/mL. It is not to be administered as an IV push or bolus injection. At the end of the infusion, flush the line with a sufficient quantity of normal saline. No more than four doses of ipilimumab should be administered.

Ipilimumab dosing calculations should be based on the actual body weight. If the patient's weight differs by >10% from the weight used to calculate the original dose, the dose may be recalculated. All doses should be rounded to the nearest milligram.

Toxicity management for ipilimumab should follow the same guidelines and algorithms that are provided in Section 7 and Appendix E.

# 6.2 General Concomitant Medication and Supportive Care Guidelines

Because there is a potential for interaction of XL184 (cabozantinib) with other concomitantly administered drugs, the CRF must capture the concurrent use of all other drugs, over-the-counter medications, or alternative therapies. The PI should be alerted if the patient is taking any agent known to affect or with the potential for drug interactions. For example, the potential targets for drug interaction can involve, but are not limited to CYPs 450, glucuronidation, P-glycoprotein, protein binding, or reduced absorption from proton-pump inhibitors. Check the Investigator's Brochures for each study agent for potential sources of drug interactions. The study team should check a frequently-updated medical reference for a list of drugs to avoid or minimize use of. Appendix B (Patient Clinical Trial Wallet Card) should be provided to patients if available.

## 6.2.1 Concomitant Medications and Therapies

# 6.2.1.1 Anticancer Therapy

If a patient requires additional systemic anticancer treatment, study treatment must be discontinued. Patients who require palliative radiation therapy while being treated in the study will need to come off the study. The need for local intervention will be considered a clinical disease progression. The addition of radiation therapy to a combination of immunotherapeutic agents may also make the interpretation of the results of this study difficult through the abscopal effect. Patients who may benefit from palliative radiation therapy must complete such intervention prior to enrollment into the study.

#### 6.2.1.2 Other Medications

Patients must be instructed to inform the treating physicians of the current or planned use of all other medications during the study (including prescription medications, over-the-counter medications, vitamins, and herbal and nutritional supplements). It is the responsibility of the treating physician to ensure that details regarding all medications are documented.

Bisphosphonates or denosumab started prior to screening activities or initiated during the course of the study to control bone pain may be used with caution. Start date and end dates for such treatments must be documented.

Pain medications administered as dictated by standard practice are acceptable while the patient is enrolled in the study.

No concurrent investigational agents are permitted.

# 6.2.1.3 Potential Drug Interactions

#### 6.2.1.3.1 Cytochrome P450

Co-administration of XL184 (cabozantinib) with strong inducers of the CYP3A4 family (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's Wort) may significantly decrease XL184 (cabozantinib) concentrations. The chronic use of strong CYP3A4 inducers should be avoided. Other drugs that induce CYP3A4 (e.g., chronic use of modafinil) should be used with caution because these drugs have the potential to decrease exposure to XL184 (cabozantinib). Selection of alternate concomitant medications with no or minimal CYP3A4 enzyme induction potential is recommended. In addition, caution must be used when discontinuing treatment with a strong CYP3A4 inducer in a patient who has been concurrently receiving a stable dose of XL184 (cabozantinib), as this could significantly increase the exposure to XL184 (cabozantinib).

Strong CYP3A4 inhibitors (*e.g.*, ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, and ritonavir) and other drugs that inhibit CYP3A4 should be avoided because these drugs have the potential to increase exposure to XL184 (cabozantinib).

Grapefruit, grapefruit juice, and Seville oranges may also increase plasma concentrations of XL184 (cabozantinib). Selection of alternate concomitant medications with no or minimal CYP3A4 enzyme inhibition potential is recommended.

Because *in vitro* studies only assessed the metabolizing capacity of the CYP3A4, CYP2C9, and CYP2D6 pathways, the potential for drugs that inhibit/induce other CYPs (*e.g.*, CYP2C8, CYP2C19, CYP2B6, CYP1A2) to alter XL184 (cabozantinib) exposure is not known. Therefore, these drugs should be used with caution when given with XL184 (cabozantinib).

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.

# 6.2.1.3.2 Protein Binding

XL184 (cabozantinib) is highly protein bound (approximately 99.9%) to human plasma proteins. Therefore, highly-protein-bound drugs should be used with caution with XL184 (cabozantinib) because the potential displacement interaction could increase free concentrations of XL184 (cabozantinib) and/or co-administered highly protein-bound drugs and lead to corresponding increases in pharmacologic effect(s). Factors that influence plasma protein binding may affect individual tolerance to XL184 (cabozantinib). Concomitant medications that are highly protein bound (e.g., diazepam, furosemide, dicloxacillin, and propranolol) should be used with caution. Because warfarin is a highly protein bound drug with a narrow therapeutic index, administration of warfarin at therapeutic doses should be avoided in patients receiving XL184 (cabozantinib) due to the potential for a protein binding displacement interaction.

#### 6.2.1.3.3 Drugs Associated with QTc Prolongation

Treatment with XL184 (cabozantinib) has been associated with a mild prolongation of the QTc interval. Caution should be used when treating patients on XL184 (cabozantinib) with other drugs associated with QTc prolongation (see <a href="http://www.qtdrugs.org">http://www.qtdrugs.org</a>). Additional QTc monitoring is suggested for patients who are treated concomitantly with QTc-prolonging drugs.

# 6.2.1.3.4 Other Interactions

Co-administration of gastric pH modifying drugs such as PPI, H<sub>2</sub>-blockers, or antacids has had no clinically relevant effect on XL184 (cabozantinib) plasma PK in healthy volunteers; thus, concomitant use of these drugs with XL184 (cabozantinib) **is allowed**.

*In vitro* data suggest that XL184 (cabozantinib) is unlikely to be a substrate for P glycoprotein (P-gp), but it does appear to have the potential to inhibit the P-gp transport activity.

Additional details related to these overall conclusions are provided in the most recent version of the XL184 (cabozantinib) Investigator's Brochure.

# 6.3 Duration of Therapy

In the absence of treatment delays due to adverse event(s), treatment may continue for until one of the following criteria applies:

- Disease progression
- Intercurrent illness that prevents further administration of treatment
- Unacceptable adverse event(s) (See also Section 7 and specific algorithms in Appendix E)
- Patient decides to withdraw from the study
- General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator
- Clinical progression
- Patient non-compliance
- Pregnancy
  - All women of child bearing potential should be instructed to contact the investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
  - The investigator must immediately notify CTEP in the event of a confirmed pregnancy in a patient participating in the study.
- Termination of the study by sponsor
- The drug manufacturer can no longer provide the study agent

The reason(s) for protocol therapy discontinuation, the reason(s) for study removal, and the corresponding dates must be documented in the Case Report Form (CRF).

# 6.4 Duration of Follow-Up

Patients will need to come in for an initial clinical follow up at 4 weeks after the last dose of the study drugs. Thereafter, patients will be followed as part of the off-study evaluation every 3 months until death or withdrawal of consent. Patients removed from study for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event. Off study follow-up can occur via a phone call.

# 7. DOSING DELAYS/DOSE MODIFICATIONS

Toxicity evaluation will be done monthly for as long as the patient is on active treatment. Complete blood counts with differential, comprehensive metabolic panel, and TSH will be done the beginning of each treatment cycle.

XL184 (cabozantinib), and nivolumab and ipilimumab have class-specific safety profiles based on their mechanisms of action, but may also cause AEs that overlap. The management of these toxicities generally includes holding drug for moderate (Grade 2) toxicities and using systemic immunosuppression for severe (Grade 3/4) or prolonged moderate (> 1 week) toxicities per the treating clinician's discretion as guided by the package insert of the respective drugs. Additional immunosuppression (e.g., anti-TNF $\alpha$  therapy, infliximab) may be used if IV steroids are ineffective at the discretion of the treating clinician using the package insert as a guide.

For management of AEs which can be clearly attributed to either XL184 (cabozantinib) or immunotherapy, independent dose modification for either component of study treatment is allowed. Examples of VEGFR TKI-associated AEs caused by XL184 (cabozantinib) are hypertension and hand-foot syndrome. Examples of immune-related AEs caused by nivolumab and ipilimumab are pneumonitis and endocrinopathies. For AEs without clear attribution to either component of study treatment, management of toxicity should include dose modifications of XL184 (cabozantinib) and immunotherapy, at the discretion of the investigator. Examples of overlapping AEs are diarrhea and transaminase increases. Patients who experience a Grade 3 or greater toxicity that is attributed to study medication and cannot be ameliorated by the use of adequate medical intervention should have their treatment interrupted until the toxicity improves to Grade 2 or lower. Patients may subsequently be re-started on study drug, including at a reduced dose in the case of XL184 (cabozantinib).

## 7.1 XL184 (Cabozantinib)

The following should be taken into consideration in decisions regarding dose modifications (reductions or interruption):

- As a general approach all AEs should be managed with supportive care at the earliest signs of toxicity considered related to the study treatment. Should this be ineffective, dose interruptions and/or reductions should be considered to prevent worsening of toxicity.
- The assigned starting dose for XL184 (cabozantinib) is 40 mg/day. Two dose reduction levels of XL184 (cabozantinib) are permitted (see Section 7.1.2).
- Study treatment dose adjustment is only needed if the AE is deemed possibly, probably, or definitely related to XL184 (cabozantinib) treatment.
- Dose modification criteria for XL184 (cabozantinib) are shown below in Section 7.1.2. Dose interruptions and/or reductions should be implemented for unacceptable toxicity. Doses may be modified at any time while a patient is on treatment.
- Dose reductions or interruptions may also occur in the setting of lower grade toxicity than defined below, if the investigator feels it is in the interest of a patient's safety and will optimize drug tolerability.

• XL184 (cabozantinib) should be held for 2 days (48 hours) prior to any biopsy procedure, and may be resumed 2 days (48 hours) following the procedure, unless there is evidence of biopsy wound-related complications or incomplete wound healing. Due to the risk of perforation and fistula with XL184 (cabozantinib), transesophageal and other transluminal biopsies should not be performed, and biopsies should not be performed in areas of prior fistula formation, surgery, or radiation.

- In patients requiring interruption of XL184 (cabozantinib) treatment due to any reason for >4 consecutive weeks, XL184 (cabozantinib) should be discontinued. In this situation, a patient may continue to receive ipilimumab and/or nivolumab per the discretion of the investigator.
- Patients on CaboNivoIpi who require permanent discontinuation of XL184 (cabozantinib) due to any reason may continue with nivolumab and ipilimumab at the investigator's discretion. Patients on XL184 (cabozantinib) plus nivolumab who require permanent discontinuation of XL184 (cabozantinib) due to any reason may continue with nivolumab at the investigator's discretion.

Many AEs can occur early (within the first few weeks) in the course of treatment, as XL184 (cabozantinib) is expected to reach steady state exposure at approximately 2 weeks following the first dose. General guidelines for the management of non-hematologic and hematologic toxicities are provided below.

#### 7.1.1 Potential Adverse Events

Calcium, magnesium, potassium, and phosphorus should be kept above the LLN. For more specific guidelines on GI AEs (GI perforation, GI fistula, intra-abdominal and pelvic abscess, diarrhea, nausea/vomiting, stomatitis/mucositis), non-GI fistula, hepatobiliary disorders, pancreatic conditions, thromboembolic events, hypertension, skin disorders (*e.g.*, palmar-plantar erythrodysesthesia syndrome [PPES]), wound healing and surgery, proteinuria, nervous system disorders, infections and infestations, corrected QT prolongation, electrolyte disorders, and endocrine disorders, refer to Section 7.1.3 below.

Guidance for the management of fatigue; anorexia; weight loss; eye disorders; musculoskeletal and connective tissue disorders; nervous system disorders; respiratory/thoracic/mediastinal disorders; and congenital, familial, and genetic disorders can be found in the XL184 (cabozantinib) Investigator's Brochure.

Patients will be monitored for AEs from the time of signing informed consent through their last follow-up visit. Patients will be instructed to notify their physician immediately at the onset of any AE. Seriousness, severity grade, and relationship to study treatment of AEs will be determined by the investigator. AE severity will be graded by the investigator in accordance with CTCAE v5.0. Management of severe or intolerable adverse reactions may require temporary dose reduction and/or interruption.

The most frequent AEs experienced by  $\geq$ 20% of patients treated with XL184 (cabozantinib) in descending order of frequency were diarrhea, fatigue, decreased appetite, nausea, weight decreased, PPES, vomiting, constipation, hypertension, dysgeusia, dysphonia, asthenia, and

dyspnea. For a full description of the safety profile of XL184 (cabozantinib), refer to the most recent Investigator's Brochure.

Other medically important but less frequent AEs including arterial thrombotic AEs (*e.g.*, TIA, and MI) and venous thrombotic AEs (*e.g.*, DVT and PE), severe hemorrhagic events, proteinuria, wound healing complications, gastrointestinal (GI) perforation, abscesses including intra-abdominal and pelvic abscess, GI and non-GI fistula formation, osteonecrosis, and reversible posterior leukoencephalopathy syndrome (RPLS).

Adverse events associated with laboratory abnormalities experienced by ≥5% of patients treated with XL184 (cabozantinib) in descending order of frequency were anemia, AST increased, ALT increased, hypothyroidism, hypokalemia, hypomagnesemia, thrombocytopenia, hypocalcemia, hypophosphatemia, lactate dehydrogenase (LDH) increased, lipase increased, neutropenia, hyponatremia, ALP increased, leukopenia, and hyperglycemia.

Adverse events may occur within the first few weeks in the course of treatment with XL184 (cabozantinib), as the drug is expected to reach steady-state exposure at approximately 2 weeks following first dose. Events that generally have an early onset include hypocalcemia, hypokalemia, thrombocytopenia, hypertension, PPES, abdominal pain, mucosal inflammation, constipation, diarrhea, and vomiting. AEs should be managed with supportive care at the earliest signs of toxicity. Dose reductions and treatment interruptions should be considered. Dose reductions are recommended for events that, if persistent, could become serious or intolerable.

XL184 (cabozantinib) should be discontinued for the following AEs: visceral perforation or fistula formation, severe hemorrhage, serious arterial thromboembolic events, nephrotic syndrome, hypertensive emergency, persistent uncontrolled hypertension despite optimal medical management, and RPLS.

# 7.1.2 General Dose Modifications for XL184 (Cabozantinib)

# Dose Reductions of XL184 (cabozantinib)

| Dose Level | XL184 (cabozantinib) dose |
|------------|---------------------------|
| 1 | 40 mg PO daily |
| -1 | 20 mg PO daily |
| -2 | 20 mg PO every other day |

PO=orally

If a patient experiences several AEs, and there are conflicting recommendations, the treating physician should use the recommended dose adjustment that reduces the dose to the lowest level.

# 7.1.2.1 XL184 (Cabozantinib) Dose Re-institution and Re-escalation

If the patient recovers from an AE to  $\leq$  grade 1 or to baseline, and the toxicity was deemed at least possibly related to study treatment, then study treatment may be resumed at a reduced dose (see above for the schedule of dose reductions).

Patients receiving a daily dose of 20 mg (Dose Level -1) may resume at the same dose if deemed safe at the investigator's discretion. Patients unable to tolerate Dose Level -1 should be reduced to receiving 20 mg every other day (Dose Level -2).

Re-escalation to the previous XL184 (cabozantinib) dose may be allowed after the first six months of study treatment, at the investigator's discretion, for AEs which have resolved to grade 1 (or baseline) and deemed tolerable and easily managed by optimized supportive treatment. Dose re-escalation is not allowed after drug-related dose reductions triggered by grade 4 hematological AEs or by grade 4 AEs affecting major organs (*e.g.*, central nervous, cardiac, hepatic, or renal systems). The XL184 (cabozantinib) dose should not exceed 40 mg/day.

# 7.1.2.2 Dose Modifications for Treatment-Related Non-Hematologic Adverse Events

| CTCAE v5.0 Grade | Recommended Dose Management |
|---|---|
| Grade 1 AEs | Add supportive care as indicated. Continue XL184 (cabozantinib) therapy at the current dose level if AE is manageable and tolerable. |
| Grade 2 AEs which are subjectively tolerable and easily managed | Add supportive care as indicated. Continue XL184 (cabozantinib) therapy at the current dose level with supportive care. |
| Grade 2 AEs which are intolerable to the patient, deemed unacceptable in the treating physician's judgment, recur after previously improving to ≤ grade 1, or are not easily managed or corrected. | Add supportive care as indicated and reduce the XL184 (cabozantinib) dose by one level. If the AE does not improve to $\leq$ grade 1 or baseline within 10 days, or worsens at any time, hold XL184 (cabozantinib). Upon resolution to baseline or $\leq$ grade 1, the previously reduced dose should be restarted. If the AE resolves to $\leq$ grade 1 or baseline without a dose interruption, continue at the reduced dose. |
| Grade 3 AEs that occur without optimal prophylaxis or which is easily managed by medical intervention or resolves quickly | Add supportive care as indicated and hold XL184 (cabozantinib). For AEs that are easily managed (e.g., electrolyte correction) and resolve to baseline or ≤ grade 1 within 24 hours, XL184 (cabozantinib) may be resumed at either the same dose or one dose level lower, at the investigator's discretion. If supportive care is required, XL184 (cabozantinib) should be held while supportive care is initiated and optimized. If this is a recurring AE, reduce the XL184 (cabozantinib) dose by one level. |

| CTCAE v5.0 Grade | Recommended Dose Management |
|---|---|
| Grade 3 AEs that occur | Hold XL184 (cabozantinib) until recovery to ≤ grade 1 or |
| despite optimal prophylaxis<br>or are not easily managed<br>by medical intervention | baseline, then resume at one dose level lower. |
| <b>Grade 4</b> AEs | For AEs that are easily managed ( <i>e.g.</i> , correction of electrolytes) with resolution to baseline or $\leq$ grade 1 within 24 hours, hold XL184 (cabozantinib) until resolution then resume one dose level lower. For other AEs, permanently discontinue XL184 (cabozantinib) unless it is determined that the patient is unequivocally deriving clinical benefit. In this case, upon recovery to $\leq$ grade 1 or baseline, the patient may be re-treated at a reduced dose, as determined by the treating physician and protocol chair (or co-chair) after consultation with the study sponsor (CTEP). |

<u>Note:</u> Dose reductions or delays may occur in the setting of lower grade toxicity than defined above if the treating physician believes that it is in the interest of the patient's safety.

<u>Note:</u> The dose modification and management guidelines for specific medical conditions are provided below. For re-treatment and re-escalation criteria, see Section 7.1.4.

# 7.1.2.3 Dose Modifications for XL184 (Cabozantinib) for Treatment-Related Hematologic Adverse Events

| Neutropenia | Recommended Guidelines for Management |
|---|---|
| Tintection Carade a tasting | Hold XL184 (cabozantinib) until resolution to ≤ grade 1, then resume with a one dose level reduction. |

| Thrombocytopenia | Recommended Guidelines for Management |
|---|---|
| Grade 3 with clinically significant bleeding or Grade 4 | Hold XL184 (cabozantinib) until platelet count is ≥100,000/mm <sup>3</sup> , then resume with a one dose level reduction. |

| Febrile Neutropenia | Recommended Guidelines for Management |
|---|---|
| Grade 3 | Hold XL184 (cabozantinib) until recovery of ANC to ≤ grade 1 and temperature to ≤38 °C and resume with a one dose level reduction. Provide supportive care as indicated. |

| Febrile Neutropenia | Recommended Guidelines for Management |
|---|---|
| Grade 4 | Permanently discontinue XL184 (cabozantinib) therapy unless |
| | the investigator determines that the patient is unequivocally |
| | deriving clinical benefit. In this case, upon recovery to $\leq$ grade 1, |
| | the patient may be re-treated at a reduced dose, as determined by |
| | the treating physician and protocol chair (or co-chair) in |
| | consultation with the study sponsor (CTEP). |

| Anemia | Recommended Guidelines for Management |
|---|---|
| Grade 4 | Permanent XL184 (cabozantinib) discontinuation for grade 4 anemia is not required. Dose reductions or delays for anemia should be applied as clinically indicated. Supportive care such as red blood cell transfusions should be managed according to |
| | institutional guidelines. |

| Other Hematological AEs | Recommended Guidelines for Management |
|---|---|
| Grade 4 | Permanently discontinue XL184 (cabozantinib) therapy unless |
| | the investigator determines that the patient is clearly deriving |
| | clinical benefit. In this case, upon recovery to $\leq$ grade 1 or |
| | baseline, the patient may be re-treated at a reduced dose, as |
| | determined by the treating physician and protocol chair (or co- |
| | chair) in consultation with the study sponsor (CTEP). |

# 7.1.3 Guidelines for Management of Potential Adverse Events

# 7.1.3.1 Gastrointestinal Disorders

# 7.1.3.1.1 Gastrointestinal perforation, GI fistula, and intra-abdominal and pelvic abscess

GI perforation/fistula have been reported with FDA-approved drugs that inhibit VEGF pathways as well as with XL184 (cabozantinib). Carefully monitor for episodes of abdominal pain, especially in patients with known risk factors for developing GI perforation/fistula or non-GI fistula, to allow for early diagnosis. Such risk factors include (but may not be limited to) the following:

- Intra-abdominal tumor/metastases invading GI mucosa;
- Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis or symptomatic cholangitis, or appendicitis;
- History of abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess;
- Prior GI surgery (particularly when associated with delayed or incomplete healing). Complete healing following abdominal surgery or resolution of intra-abdominal abscess must be confirmed prior to initiating treatment with XL184 (cabozantinib).

Complete healing following abdominal surgery or resolution of intra-abdominal abscess must be confirmed prior to initiating treatment with XL184 (cabozantinib). After starting cabozantinib, subjects should be monitored for early signs of GI perforation such as abdominal pain, nausea, emesis, constipation, and fever especially if known risk factors for developing GI perforation or fistula are present. Additional risk factors include concurrent chronic use of steroid treatment or non-steroidal anti-inflammatory drugs. Constipation indicative of bowel obstruction should be monitored and effectively managed.

Permanently discontinue XL184 (cabozantinib) therapy and initiate appropriate management in patients who have been diagnosed with GI perforation or fistula.

Rectal and perirectal abscesses have been reported, sometimes in patients with concurrent diarrhea. These should be treated with appropriate local care and antibiotic therapy. XL184 (cabozantinib) should be held until adequate healing has taken place.

# 7.1.3.1.2 Diarrhea

Patients should be instructed to notify their physician immediately at the first signs of poorly formed or loose stool or an increased frequency of bowel movements. Administration of antidiarrheal/antimotility agents is recommended at the first sign of treatment-related diarrhea as initial management. Loperamide is recommended as standard first line therapy. Alternatively, diphenoxylate/atropine can be used. Additional agents to consider in patients with diarrhea that is refractory to the above include deodorized tincture of opium and colestipol. Some patients may require concomitant therapy with loperamide, diphenoxylate/atropine, and deodorized tincture of opium to control diarrhea. Infectious work-up may be carried out as needed per physician discretion. Dose modification guidelines for non-hematologic AEs should be followed. In addition, general supportive measures should be implemented such as continuous oral isotonic hydration, correction of fluid and electrolyte abnormalities, small frequent meals, and stopping lactose-containing products, high-fat meals, and alcohol.

Recurrent or prolonged diarrhea can be associated with anal or perianal skin erosions which increase the risk for anal abscesses, fistulas, or proctitis. Good personal hygiene should be emphasized. Regular examinations of the perianal region should be performed whenever diarrhea has occurred during treatment with XL184 (cabozantinib). Infections of the perianal region should be treated per local guidelines.

#### 7.1.3.1.3 Nausea and vomiting

Anti-emetic agents along with supportive care are recommended as clinically appropriate at the first sign of nausea and vomiting. The dose modification guidance for non-hematologic AEs in Section 7.1.1.1 should be followed. 5-HT3 receptor antagonists are recommended over chronic use of NK-1 receptor antagonists and dexamethasone (NK-1 receptor antagonists and glucocorticoids can interact with CYP3A4 and thus change XL184 [cabozantinib] exposure). Caution is also recommended with the use of nabilone, which is a weak inhibitor of CYP3A4. Please note that caution should be used when using ondansetron (a 5-HT3 antagonist) as it can prolong QTc intervals. Dehydration and electrolyte abnormalities may be associated with
vomiting and monitoring for and correction of fluid and electrolyte imbalances should be implemented.

#### 7.1.3.1.4 Stomatitis and Mucositis

Preventive measures may include a comprehensive oral examination to identify and treat any potential risk for complications before XL184 (cabozantinib) therapy is initiated. Appropriate correction of local factors should be instituted as indicated, such as modification of ill-fitting dentures and appropriate care of gingivitis. During XL184 (cabozantinib) therapy, good oral hygiene and standard local treatments such as non-traumatic and non-irritating cleansing, and oral rinses (*e.g.*, with a weak solution of salt and baking soda) should be maintained. Lips should be kept moisturized with lip balm. The use of lipstick, lip-gloss, and Vaseline should be avoided. Local treatment should be instituted at the earliest onset of symptoms. Obtain bacterial/viral culture if oral infection is suspected and treat infection as clinically indicated.

## 7.1.3.2 Non-Gastrointestinal Fistula

Complications from radiation therapy especially of the thoracic cavity including mediastinum have been identified as a possible predisposing risk factor for non-GI fistula formation in patients undergoing treatment with VEGF pathway inhibitors. In addition, patients who have undergone extensive surgery may be at increased risk of developing a fistula of the involved organs. Permanently discontinue XL184 (cabozantinib) therapy and initiate appropriate management in patients who have been diagnosed with a non-GI fistula.

# 7.1.3.3 Hepatobiliary disorders

## 7.1.3.3.1 Elevation of aminotransferases (ALT and AST):

Evaluation of patients with elevated transaminases or bilirubin should be individualized and guided by the presence of specific risk factors such as liver conditions (*e.g.*, liver cirrhosis, metastases to the liver, thrombosis of portal or hepatic vein, hepatocellular carcinoma, or hepatitis), concomitant hepatotoxic medication, alcohol consumption, and cancer related causes.

Elevations of transaminases have been observed during treatment with XL184 (cabozantinib). In general, it is recommended that patients with elevation of ALT, AST, and/or bilirubin have more frequent liver function tests (LFTs). If possible, hepatotoxic concomitant medications and alcohol should be discontinued in patients who develop elevated transaminases. Since patients may enter the study with elevations of AST/ALT at baseline, the following guideline should be used for dose modifications:

| <b>Transaminase Elevation</b> | Intervention |
|---|---|
| Grade 1 | No change in XL184 (cabozantinib) dose, and no additional tests unless clinically indicated. |

| <b>Transaminase Elevation</b> | Intervention |
|---|---|
| Grade 2 | Continue XL184 (cabozantinib) with at least twice weekly monitoring of LFTs for 2 weeks. Then weekly for 4 weeks. If LFTs continue to rise within grade 2, hold XL184 (cabozantinib), and continue with at least weekly LFTs until improvement to ≤ grade 1. XL184 (cabozantinib) may then be resumed with a one dose level reduction. |
| Grade 3 | Hold XL184 (cabozantinib) and monitor with at least twice weekly LFTs until ≤ grade 2, then with at least weekly LFTs until ≤ grade 1. XL184 (cabozantinib) may then be resumed with a one dose level reduction. |
| Grade 4 | Permanently discontinue XL184 (cabozantinib) therapy. LFTs should be monitored as clinically indicated, at least 2-3 times per week, until improvement to ≤ grade 1. If the patient was unequivocally deriving clinical benefit, XL184 (cabozantinib) may be restarted at a reduced dose, as determined by the treating physician and protocol chair (or co-chair) in consultation with the study sponsor (CTEP). |

XL184 (cabozantinib) treatment should also be interrupted when transaminase increases are accompanied by progressive elevations of total bilirubin, and/or elevations of coagulation tests (e.g., International Normalized Ratio [INR]). Monitoring of transaminases should be intensified (2-3 times per week) and XL184 (cabozantinib) should be held until the etiology of the abnormalities is determined and these abnormalities are corrected or stabilize at clinically acceptable levels (INR  $<1.5 \times ULN$ , total bilirubin  $<1.5 \times ULN$ , aminotransferases  $\le$  baseline grade).

XL184 (cabozantinib) should be permanently discontinued if transaminase elevations are accompanied by evidence of impaired hepatic function (bilirubin elevation > 1.5 x ULN unless Gilbert's syndrome), in the absence of evidence of biliary obstruction (*i.e.*, significant elevation of alkaline phosphatase), or some other explanation of the injury (*e.g.*, viral hepatitis, alcohol hepatitis), as the combined finding represents a signal of a potential for the drug to cause severe liver injury (*i.e.*, Hy's Law cases).

All patients who develop isolated bilirubin elevations of grade 3 should have XL184 (cabozantinib) held until recovery to ≤ grade 1 or baseline (or lower). If this occurs within 4 weeks of the dosing delay, XL184 (cabozantinib) therapy may continue with a one dose level reduction. In patients without biliary obstruction and grade 4 bilirubin elevation, or with recurrence of grade 3 bilirubin elevation after a dose reduction, XL184 (cabozantinib) therapy must be discontinued.

## 7.1.3.4 Pancreatic conditions

Amylase and lipase elevations have been observed in clinical studies with XL184 (cabozantinib). The clinical significance of asymptomatic elevations of enzymes is not known but in general have not been associated with clinically apparent sequelae. It is recommended that patients with lipase elevation and/or symptoms of pancreatitis have more frequent laboratory monitoring of lipase and/or amylase (2-3 times per week). Patients with symptomatic pancreatitis should be treated with standard supportive measures.

| Asymptomatic Lipase or<br>Amylase Elevations | Intervention |
|---|---|
| Grade 1 or Grade 2 | Continue at current dose level. More frequent monitoring is recommended. |
| Grade 3 | Hold XL184 (cabozantinib) and monitor lipase and amylase twice weekly. Upon improvement to ≤ grade 1 or baseline, XL184 (cabozantinib) therapy may resume at the same dose or one dose level lower, at the investigator's discretion. If retreatment following grade 3 lipase or amylase elevation is at the same dose and grade 3 or 4 elevations recur, then XL184 (cabozantinib) must be held again until lipase and amylase levels have resolved to ≤ grade 1 or baseline and re-treatment must be with a one dose level reduction. |
| Grade 4 | Hold XL184 (cabozantinib) and monitor lipase and amylase twice weekly. Upon resolution to ≤ grade 1 or baseline, and if resolution occurred within four days, XL184 (cabozantinib) therapy may resume at the same dose or one dose level lower, at the investigator's discretion. If resolution takes more than four days, the dose must be reduced, provided that resolution occurs within 4 weeks. If XL184 (cabozantinib) is resumed at the same dose following a grade 4 lipase or amylase elevation and grade 3 or 4 elevations recur, then XL184 (cabozantinib) must be held again until lipase and amylase have resolved to ≤ grade 1 or baseline and must be resumed with a one dose level reduction. |

| Pancreatitis | Intervention |
|---|---|
| Grade 2 | Continue at current dose level. More frequent monitoring of lipase and amylase and radiographic evaluation is recommended. |
| Grade 3 | Hold and monitor lipase and amylase twice weekly. Upon resolution to ≤ grade 1 or baseline, XL184 (cabozantinib) may be resumed with a one dose level reduction, if resolution occurs within 4 weeks. |

| Pancreatitis | Intervention |
|---|---|
| | Permanently discontinue XL184 (cabozantinib) therapy. |
| | However, if the patient was unequivocally deriving benefit from |
| Grade 4 | XL184 (cabozantinib) therapy, treatment may be restarted at a |
| | reduced dose, as determined by treating physician and protocol |
| | chair (or co-chair) in consultation with the study sponsor (CTEP). |

## 7.1.3.5 Hemorrhage

Hemorrhagic events, including serious and sometimes fatal events, have been reported with XL184 (cabozantinib). Patients should be monitored for bleeding events with serial complete blood counts and physical examination while on study. The risk of hemorrhage in XL184 (cabozantinib)-treated patients with brain metastases has not been thoroughly analyzed. Patients enrolled with treated and stable brain metastases should be monitored with a high index of suspicion if symptoms attributable to CNS hemorrhage occur.

XL184 (cabozantinib) therapy should be permanently discontinued in patients with serious and life-threatening bleeding events or recent clinically significant hemoptysis. Treatment with XL184 (cabozantinib) should be held if less severe forms of clinically significant hemorrhage occur. After the cause of hemorrhage has been identified and the risk of bleeding has subsided, XL184 (cabozantinib) may be resumed at a dose agreed to by the protocol chair (or co-chair) and the treating physician. Therapy of bleeding events should include supportive care and standard medical interventions.

#### 7.1.3.6 Thromboembolic events

Thromboembolic events are frequent in cancer patients due to procoagulant changes induced by the malignancy or anticancer therapy. DVT and PE have been observed in clinical studies with XL184 (cabozantinib), including fatal events. Patients who develop DVT and/or PE should have study treatment interrupted until therapeutic anticoagulation is established. Treatment with XL184 (cabozantinib) may be resumed at one dose level lower in patients with uncomplicated PE or DVT if it is determined that the patient is deriving clinical benefit from XL184 (cabozantinib) treatment and that anticoagulation does not place them at a significant risk that outweighs the benefit of resuming treatment per discretion of the investigator and according to individual protocols. Patients with life-threatening DVT or PE should have XL184 (cabozantinib) therapy discontinued unless toxicity can be managed, and the patient is deriving clear clinical benefit as determined by the treating physician in consultation with the study sponsor (CTEP). Venous filters (e.g. vena cava filters) are not recommended due to the high incidence of complications associated with their use. Once a patient is fully anticoagulated, treatment can be restarted at the investigator's discretion with a one dose level reduction. XL184 (cabozantinib) therapy should be permanently discontinued after a second thrombotic event. Although routine prophylactic anticoagulation is not necessary for all patients, prophylactic anticoagulation is allowed for individual patients at the investigator's discretion. Low molecular weight heparins are the preferred management for thrombotic events; oral anticoagulants (e.g., warfarin or other coumarin-related agents, direct thrombin, direct factor Xa inhibitors,

antiplatelet agents, or chronic use of aspirin above low dose levels for cardioprotection) are not allowed.

Arterial thrombotic events (e.g., TIA, MI) have been observed in studies with XL184 (cabozantinib). Further treatment with XL184 (cabozantinib) should be permanently discontinued in patients who develop an acute MI, cerebral infarction, or any other clinically significant arterial thromboembolic complication.

## 7.1.3.7 Hypertension

Hypertension is a relatively common complication of other VEGF-pathway inhibitors and has been observed in XL184 (cabozantinib) clinical studies. Decisions to decrease or hold the dose of XL184 (cabozantinib) must be based on BP readings taken by a medical professional and must be confirmed with a second measurement at least 5 minutes following the first measurement. Patients with known hypertension should be optimally managed prior to study entry. Clinical judgment should be used in deciding whether new or worsened hypertension emerging during treatment requires immediate therapy, or whether therapeutic intervention can be delayed in order to confirm the finding of new or worsened hypertension at a second visit before taking new therapeutic action. It is recommended that this second visit occur within one week (such a visit can be with a local physician or a study physician). BP should be monitored in a constant position visit to visit, either sitting or supine.

XL184 (cabozantinib) should be held in patients with severe hypertension ( $\geq$ 180 mm Hg systolic or  $\geq$ 120 mm Hg diastolic; or sustained  $\geq$ 160 mm Hg systolic or  $\geq$ 110 diastolic) who cannot be controlled with medical interventions and should be permanently discontinued in patients with hypertensive emergency. The table below provides treatment guidelines for hypertension deemed related to XL184 (cabozantinib). BP should be monitored in a constant position visit to visit, either sitting or supine in a relaxed setting. XL184 (cabozantinib) dose modification decisions must be based on BP readings taken by a medical professional and must be confirmed with a second measurement at least 5 minutes following the first measurement.

| Criteria for Dose<br>Modifications | Treatment/XL184 (cabozantinib) Dose Modification |
|---|---|
| Patients NOT receiving opt | timized anti-hypertensive therapy |
| Systolic ≥140 and | Optimize antihypertensive therapy (i.e., increase dose of existing |
| <160 mm Hg | medications and/or add new antihypertensive medications) and |
| | continue XL184 (cabozantinib) with no change. If optimal |
| OR | antihypertensive therapy (usually to include three agents) does |
| | not result in BP <140 mm Hg systolic and <90 mm Hg diastolic, |
| Diastolic ≥90 and | or if the patient is symptomatic, the dose of XL184 |
| <110 mm Hg | (cabozantinib) should be reduced by one level. |
| | , |

| Criteria for Dose<br>Modifications | Treatment/XL184 (cabozantinib) Dose Modification |
|---|---|
| Systolic ≥160 and<br><180 mm Hg | Reduce XL184 (cabozantinib) by one dose level. Optimize antihypertensive therapy ( <i>i.e.</i> , increase the dose of existing medications and/or add new antihypertensive medications). |
| OR | Monitor the patient closely for hypotension. If optimal antihypertensive therapy (usually to include three agents) does |
| Diastolic ≥110 and<br><120 mm Hg | not result in BP <140 mm Hg systolic and <90 mm Hg diastolic, the dose of XL184 (cabozantinib) should be reduced further. |
| Systolic ≥180 mm Hg<br>OR | Hold XL184 (cabozantinib) and add new or additional antihypertensive medications and/or increase the dose of existing medications. Monitor the patient closely for hypotension. When BP <140 mm Hg systolic and <90 mm Hg diastolic, resume XL184 (cabozantinib) treatment with a one dose level reduction. |
| Diastolic ≥120 mm Hg | If optimal antihypertensive therapy (usually to include three agents) does not result in BP <140 systolic or < 90 diastolic, the dose should be reduced further. |
| Hypertensive emergency* | Permanently discontinue XL184 (cabozantinib) therapy. |

<sup>\*</sup> Hypertensive emergency is defined as uncontrolled elevated BP with clinical evidence of progressive or impending end-organ damage (*e.g.*, myocardial infarction/ischemia, intracranial hemorrhage, cerebral ischemia, pulmonary edema, encephalopathy, or kidney damage).

<u>Note:</u> If systolic and diastolic BP meet different criteria in the table, manage according to the higher dose-modification criterion.

<u>Note:</u> In patients deemed to have a component of white coat hypertension, a home BP log can be used at the investigator's discretion.

#### 7.1.3.8 Palmar-plantar erythrodysesthesia syndrome (PPES)

PPES (also known as hand-foot syndrome), skin rash (including blister, erythematous rash, macular rash, skin exfoliation, dermatitis acneiform, and papular rash), pruritus, dry skin, erythema, pigmentary changes, and alopecia have been reported with XL184 (cabozantinib). All patients on study should be advised on prophylactic measures including the use of emollients, removal of calluses, avoidance of exposure of hands and feet to hot water leading to vasodilatation, protection of pressure-sensitive areas of hands and feet, and use of cotton gloves and socks to prevent injury and keep the palms and soles dry. Early manifestations include tingling, numbness, mild hyperkeratosis, and symmetrical red and swollen areas on the palms and soles. The lateral sides of the fingers or periungual zones may also be affected. Adequate interventions are required to prevent worsening of skin symptoms such as blisters, desquamations, ulcerations, or necrosis of affected areas. Analgesics may be required for pain control.

Aggressive management of symptoms is recommended, including early dermatology referral. Treatment recommendations in response to PPES are summarized below.

| PPES | Action to be Taken |
|---|---|
| Grade 1 | XL184 (cabozantinib) may be continued at the current dose if PPES is clinically insignificant and tolerable. Otherwise, the XL184 (cabozantinib) dose should be reduced by one level. Start or continue treatment with urea 20-40% cream twice daily and high potency steroid cream (e.g. clobetasol 0.05% cream twice daily). A topical lidocaine 5% ointment or NSAIDs/GABA agonists/narcotics may also be used for pain control. Patients should be reassessed at least weekly for changes in severity. Patients should be instructed to notify their treating physician immediately if severity worsens. |
| Grade 2 | XL184 (cabozantinib) may be continued at the same dose level if PPES is tolerated. The XL184 (cabozantinib) dose should be reduced or held if PPES is intolerable. Start or continue treatment with urea 20-40% cream twice daily and high potency steroid cream (e.g. clobetasol 0.05% cream twice daily). A topical lidocaine 5% ointment or NSAIDs/GABA agonists/narcotics may also be used for pain control. Patients should be reassessed at least weekly for changes in severity. If XL184 (cabozantinib) was held (but not reduced), it may be resumed at the same dose or one dose level lower upon resolution to ≤ grade 1. If a second interruption is required, the XL184 (cabozantinib) dose must be reduced by one level when treatment resumes. Patients should be instructed to notify their treating physician immediately if the severity worsens. If the severity worsens at any time, or affects self-care, proceed to the management guidelines for grade 3 PPES. |
| Grade 3 | Hold XL184 (cabozantinib) until severity decreases ≤ to grade 1. Start or continue treatment with urea 20-40% cream twice daily and high potency steroid cream (e.g. clobetasol 0.05% cream twice daily). A topical lidocaine 5% ointment or NSAIDs/GABA agonists/narcotics may also be used for pain control. Resume XL184 (cabozantinib) at one dose level lower upon resolution to ≤ grade 1. Permanently discontinue XL184 (cabozantinib) therapy if PPES worsens or does not improve within 4 weeks. |

#### 7.1.3.9 Osteonecrosis

Osteonecrosis has been reported in patients treated with XL184 (cabozantinib). Additional risk factors include use of bisphosphonates and denosumab, chemotherapy and anti-angiogenic drugs, use of corticosteroids, local radiotherapy, and dental or orofacial surgery procedures.

Osteonecrosis of the jaw (ONJ) can manifest as jaw pain, osteomyelitis, osteitis, bone erosion, tooth or periodontal infection, toothache, gingival ulceration, or gingival erosion. Persistent pain or slow healing of the mouth or jaw after dental surgery may also be manifestations of osteonecrosis. Advise patients regarding oral hygiene practice and to quickly report symptoms to investigator. Caution should be used in patients receiving bisphosphonates.

Invasive dental procedures should be avoided. In cases where dental procedures are unavoidable, the risks and benefits of a dental procedure and the extent of the procedure as well as the risk of developing osteonecrosis of the jaw need to be considered when deciding on the duration of a temporary treatment interruption of XL184 (cabozantinib). If clinically possible, treatment with XL184 (cabozantinib) should be interrupted for at least 4 weeks prior to the procedure and resumed after complete wound healing has occurred. Bone healing may often require a protracted time.

Patients with any documented case of osteonecrosis should stop XL184 (cabozantinib) therapy, and appropriate clinical management should be initiated. Re-initiation of study treatment must be discussed with and approved by the study sponsor (CTEP) on a case by case basis

## 7.1.3.10 Wound healing and surgery

XL184 (cabozantinib) has the potential to cause wound healing complications and wound dehiscence which may even occur long after a wound has been considered healed. Therefore, surgical, and traumatic wounds must not only be completely healed prior to starting XL184 (cabozantinib) treatment but must also be monitored for wound dehiscence, wound infection, and other signs of impaired wound healing while the patient is being treated. If dehiscence occurs, XL184 (cabozantinib) treatment should not be restarted until complete healing has taken place.

Treatment with XL184 (cabozantinib) must be interrupted for any wound healing complication which needs medical intervention. Treatment with XL184 (cabozantinib) can be resumed once wound healing has occurred unless otherwise prohibited in specific protocols. XL184 (cabozantinib) should be discontinued in patients with serious or chronic wound healing complications.

The appropriate dose hold interval prior to elective surgery to reduce the risk for wound healing complications has not been determined. In general, XL184 (cabozantinib) should be stopped at least 3 weeks (5 half-lives) prior to elective major surgery. The decision to resume treatment with XL184 (cabozantinib) after surgery should be based on clinical judgment of adequate wound healing.

## 7.1.3.11 Proteinuria

Proteinuria has been reported with XL184 (cabozantinib). Proteinuria should be monitored by measuring UPCR. The following table provides treatment guidelines for proteinuria deemed related to XL184 (cabozantinib). XL184 (cabozantinib) should be permanently discontinued in patients who develop nephrotic syndrome (proteinuria >3.5 grams per day in combination with hypoalbuminemia, edema, and hyperlipidemia).

| Severity of Proteinuria (UPCR) | Management of Proteinuria |
|---|---|
| <b>≤1 mg/mg</b> (≤113.1 mg/mmol) | No change in XL184 (cabozantinib) dose or UPCR monitoring |
| >1 and ≤2 mg/mg<br>(>113.1 and ≤226.2<br>mg/mmol) | No change in XL184 (cabozantinib) dose. A nephrology consultation is recommended. Monitor UPCR once a week. If UPCR ≤1 mg/mg on two consecutive readings, UPCR monitoring can revert to protocol-specific times. The second reading is confirmatory and can be done within 1 week of first reading. If UPCR remains >1 mg/mg and ≤2 mg/mg for one month, or is determined to be stable (<20% change) for one month, UPCR monitoring can revert to protocol-specific times and as clinically indicated. |
| >2 and <3.5 mg/mg<br>(>226.2 and <395.9<br>mg/mmol) | Hold XL184 (cabozantinib). A nephrology consultation is recommended. 24-hour urine protein assessment must be sent off within 7 days. If urine protein is >2 mg/mg, continue to hold XL184 (cabozantinib), check UPCR again within 7 days, and repeat once a week until UPCR decreases to ≤2 mg/mg. Resume XL184 (cabozantinib) at 1 dose level lower once UPCR is ≤2 mg/mg. Repeat UPCR test within 7 days of resuming XL184 (cabozantinib). Monitoring of UPCR should continue weekly until the UPCR decreases to ≤1 mg/mg. If UPCR remains >1 mg/mg and ≤2 mg/mg for 1 month or is determined to be stable (<20% change) for 1 month, UPCR monitoring can revert to protocol-specific times and as clinically indicated. |

| Severity of Proteinuria (UPCR) | Management of Proteinuria |
|---|---|
| ≥3.5 mg/mg<br>(≥395.9 mg/mmol) | Hold XL184 (cabozantinib). A nephrology consultation is mandatory. 24-hour urine for protein assessment must be sent off within 7 days. If 24-hour urine protein is ≥3.5 mg/mg, continue to hold XL184 (cabozantinib), check UPCR again within 7 days and repeat once a week. If UPCR decreases to ≤2 mg/mg, restart XL184 (cabozantinib) treatment at one dose level lower than previous dose. Repeat UPCR within 7 days of resuming XL184 (cabozantinib). Monitoring of UPCR should continue weekly until the UPCR decreases to <1 mg/mg. If UPCR remains >1 mg/mg and <2 mg/mg for 1 month or is determined to be stable (<20% change) for 1 month, UPCR monitoring can revert to protocol-specific times and as clinically indicated. |
| Nephrotic syndrome | Permanently discontinue XL184 (cabozantinib) therapy |

## 7.1.3.12 Nervous System Disorders

XL184 (cabozantinib) appears to represent minimal risk of adverse neurological effects based on nonclinical toxicology studies. However, dysphonia, dysgeusia, headache, dizziness, confused state, convulsion, depression, memory impairment, hypoesthesia, peripheral neuropathy, insomnia, ataxia, and encephalopathy have been observed in clinical studies with XL184 (cabozantinib). The development of any new or progressive, unexplained neurological symptoms should be assessed for underlying causes.

RPLS has been reported and should be considered in any patient presenting with seizures, headache, visual disturbances, confusion or altered mental function. XL184 (cabozantinib) therapy should be permanently discontinued in patients with RPLS.

#### 7.1.3.13 Infections and Infestations

Infections are commonly observed in cancer patients. Risk factors include decreased immune status (*e.g.*, after myelosuppressive anticancer therapies or splenectomy), destructive growth of the underlying malignancy including bone marrow infiltration with suppression of normal hematopoiesis, and the presence of IV devices. Infections and abscesses should be treated with appropriate local care and systemic therapy. XL184 (cabozantinib) should be held until adequate healing has taken place.

## 7.1.3.14 QTc Prolongation

Review of the larger safety database (~5000 patients exposed to XL184 (cabozantinib) in clinical trials and in post-marketing experience) showed no safety concerns associated with QT prolongation. There were no events of torsades de pointes reported.

Concomitant treatment with strong cytochrome P450 (CYP) 3A4 inhibitors, which may increase XL184 (cabozantinib) plasma concentrations, should be avoided. If at any time on study there is an increase in QTcF to an absolute value >500 msec, two additional EKGs must be performed with intervals not less than 3 min apart within 30 min after the initial EKG. If the average QTcF from the three EKGs is >500 msec, the following actions must be taken:

- Hold XL184 (cabozantinib)
- Hospitalize symptomatic patients (e.g., with palpitations, dizziness, syncope, orthostatic hypotension, or a significant ventricular arrhythmia on EKG) for a thorough cardiology evaluation and management
  - Consider cardiology consultation for asymptomatic patients for evaluation and management
- Check electrolytes, especially magnesium, potassium, and calcium; correct abnormalities as clinically indicated
- Check concomitant medications for any medication that may have contributed to QT prolongation, and if possible, discontinue these medications (http://www.qtdrugs.org)
- Repeat EKG triplicates hourly until the average QTcF is ≤500 msec, or otherwise determined by consultation with a cardiologist or appropriate expert.

Patients with QTc prolongation and symptoms must be monitored closely until the QTc elevation and symptoms have resolved. XL184 (cabozantinib) treatment may be resumed at a reduced dose level if all of the following conditions are met:

- Symptoms are determined to be unrelated to the QT interval prolongation,
- The QTcF value >500 msec is not confirmed,
- XL184 (cabozantinib) has been held through a minimum of 1 week following the return of the QTcF to ≤500 msec,
- QT prolongation can be unequivocally associated with an event other than XL184 (cabozantinib) administration and is treatable/has been resolved.

Once XL184 (cabozantinib) therapy has resumed, EKGs must be repeated weekly for 2 weeks, then every 2 weeks for 1 month, then according to the protocol-defined time points. XL184 (cabozantinib) therapy must be permanently discontinued if either of the following applies:

- Cardiac evaluation confirms that symptoms are the consequence of QT interval prolongation
- Recurrence of QTc prolongation after re-initiation of study treatment at a reduced dose

#### 7.1.3.15 Electrolyte Disorders

Serum electrolyte disorders including hyponatremia, hypokalemia, hypomagnesemia, and hypophosphatemia have been reported during treatment with XL184 (cabozantinib), and serum electrolyte levels should be monitored frequently while receiving XL184 (cabozantinib). Clinically relevant electrolyte disorders should be managed according to the dose modification

guidelines or as clinically indicated. Standard clinical practice guidelines should be used for management of electrolyte disorders and may include oral or intravenous replacement.

#### 7.1.3.16 Endocrine Disorders

Treatment-emergent elevation of thyroid-stimulating hormone (TSH) has been observed with XL184 (cabozantinib) treatment. Currently available data are insufficient to determine the mechanism of thyroid function test alterations and its clinical relevance. Management of thyroid dysfunction (*e.g.*, symptomatic hypothyroidism) should follow accepted clinical practice guidelines.

Other endocrine disorders leading to hypocalcemia and hyperglycemia, and associated laboratory changes, have been observed in less than 10% of patients. Monitoring with standard laboratory tests for endocrine disorders and clinical examination prior to initiating and during XL184 (cabozantinib) therapy is required. XL184 (cabozantinib) therapy should be discontinued in patients with severe or life-threatening endocrine dysfunction.

## 7.2 Nivolumab and Ipilimumab

Patients receiving ipilimumab in combination with nivolumab that have drug-related toxicities that meet the criteria for dose delay, should have both drugs (ipilimumab and nivolumab) delayed until retreatment criteria are met (see tables below).

- 1. In addition to the AEs identified in the tables below, ipilimumab and nivolumab doses should be delayed for any AE, laboratory abnormality or intercurrent illness which, in the judgment of the investigator, warrants a delay.
  - (a) Patients who develop alopecia and/or altered taste may continue treatment without reduction or interruption. In addition, no dose reductions or interruptions will be required for anemia (nonhemolytic) as it can be satisfactorily managed by transfusion.
- 2. Patients requiring a delay of >4 weeks due to ipilimumab- and/or nivolumab-related AEs or who experience immune-related toxicity requiring ≥10 mg/day prednisone must permanently discontinue nivolumab and ipilimumab therapy, but may continue XL184 (cabozantinib) therapy.
  - (a) Patients who receive systemic corticosteroids for management of any drug-related immunologic toxicity must be off corticosteroids or must have tapered down to a dose equivalent to <10 mg/day prednisone.
- 3. Patients requiring a delay of >4 weeks due to non-immune related AE from nivolumaband/or ipilimumab should permanently discontinue nivolumab and ipilimumab therapy, but may continue XL184 (cabozantinib) therapy.
- 4. Doses missed due to adverse events or toxicity will not be made up.
- 5. Allowance for dose synchronization:
  - (a) Nivolumab is allowed to be delayed until the next planned ipilimumab dose <u>if the</u> next ipilimumab dose is scheduled within the next 12 days.
    - (i) Nivolumab and ipilimumab doses can be re-synced, at the investigator's discretion, where possible, within the guidance indicated above.

- (ii) This will permit periodic ipilimumab dosing to be synchronized with nivolumab dosing.
- (iii) Patients who require treatment-related delay of nivolumab should be reevaluated weekly, or more frequently if clinically indicated, and may resume nivolumab dosing when re-treatment criteria are met.

# Assessments should continue even if dosing is delayed.

- (b) Allowance for ipilimumab dose delays:
  - (i) In general, patients who meet criteria to resume ipilimumab will also have met criteria to resume nivolumab with ipilimumab, so it should be feasible to synchronize dosing of both drugs when resuming ipilimumab. In order to facilitate this, the dosing days of nivolumab and ipilimumab may be adjusted within a ±5-day window, as long as consecutive nivolumab doses are given at least 12 days apart.
  - (ii) If an ipilimumab dose is delayed for >4 weeks from the prior dose, then subsequent doses should be rescheduled to maintain at least a 6-week interval between consecutive ipilimumab doses.
  - (iii) Dosing delays up to 6 weeks to manage drug-related adverse events, such as prolonged steroid tapers, are allowed.

# Assessments should continue even if dosing is delayed.

(iv) In the event that a patient experiences a grade 2 AE while on combination CaboNivoIpi therapy, the patient may resume treatment/may be continued on nivolumab and XL184 (cabozantinib) therapy, at the discretion of the treating investigator (ipilimumab will not be given without nivolumab).

If a patient experiences several AEs, and there are conflicting recommendations, the investigator should use the recommended treatment modification for the most serious event when that has a higher level of modification, *i.e.* discontinuing *versus* holding drug.

Below are AE management tables for nivolumab and combination nivolumab with ipilimumab for the following treatment-related adverse events. Please use as written and contact the drug monitor for any proposed changes.

Please refer to the most recent Nivolumab and Ipilimumab Investigator's Brochures or Appendix F for toxicity management algorithms which include specific treatment guidelines. These algorithms should be followed unless there are specific clinical circumstances for which the treating physician decides an alternative treatment approach is clinically appropriate. Consultation with the study PI or drug monitor is recommended. In several places there are differences from the algorithms regarding protocol directed drug modifications. In these cases, please follow the protocol-specific guidelines in this section. Generally, we strongly encourage early evaluation while withholding drug, and appropriate treatment as indicated in the management tables and event specific guidelines.

# 7.2.1 Guidelines for Management of Potential Adverse Events

| Skin Rash and | Management/Next Dose for | Management/Next Dose for |
|---|---|---|
| <b>Oral Lesions</b> | Nivolumab | Nivolumab plus Ipilimumab |
| ≤ Grade 1 | No change.* | No change.* |
| Grade 2-3 | Hold* nivolumab until ≤ grade 1, | Hold* both drugs until ≤ grade 1, |
| | then resume. | then resume. |
| Grade 4 | Permanently discontinue | Permanently discontinue |
| Grade 4 | nivolumab therapy. | nivolumab and ipilimumab therapy. |

<sup>\*</sup>Patients with purpuric or bullous lesions must be evaluated for vasculitis, Steven-Johnson syndrome, TEN, or autoimmune bullous disease including oral lesions of bullous pemphigus/pemphagoid. Pruritus may occur with or without skin rash and should be treated symptomatically if there is no associated liver or GI toxicity. Skin rash typically occurs early and may be followed by additional events, particularly during steroids tapering.

Recommended management: AE management guidelines.

| Drug-related uveitis, eye pain, blurred vision | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change.* | No change.* |
| Grade 2 | Hold* until < grade 1 or baseline, then resume at same dose. If a grade 2 event does not respond to topical therapy and does not improve to grade 1 within the retreatment period OR requires systemic therapy, permanently discontinue nivolumab therapy. | Hold both drugs until ≤grade 1 or baseline, then resume at same doses. If grade 2 event does not respond to topical therapy and does not improve to grade 1 within the re-treatment period OR requires systemic therapy, permanently discontinue nivolumab and ipilimumab therapy. |
| Grade 3 | Permanently discontinue nivolumab therapy. | Permanently discontinue ipilimumab and hold nivolumab until ≤ grade 1 and then resume nivolumab monotherapy. If grade 3 event does not respond to topical therapy and does not improve to grade 1 within the re-treatment period OR requires systemic therapy, permanently discontinue nivolumab as well. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |
| Recommended management: AE management guidelines. | | |

| Liver Function<br>AST, ALT,<br>Bilirubin | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | Hold nivolumab, at investigator's discretion, until values return to ULN or baseline, then resume. | Hold both drugs, at investigator's discretion, until values return to ULN or baseline, then resume. |
| Grade 2<br>(3-5 × ULN) | Hold nivolumab until values return to baseline or ≤ grade 1, then resume. | Hold both drugs until values return to baseline or ≤ grade 1, then resume. |
| Grade 3<br>(5-20 × ULN) | Hold nivolumab and monitor with at least weekly LFTs until grade ≤2. Then resume nivolumab and continue with at least weekly LFTs until improvement to grade ≤ 1. If no improvement is seen, or the condition worsens by 4 weeks, nivolumab should be held, and steroid treatment initiated. If AST/ALT >8 × ULN or bilirubin >5 × ULN, permanently discontinue nivolumab therapy. | Hold both drugs and monitor with at least weekly LFTs until grade ≤2. Then resume both drugs and continue with at least weekly LFTs until improvement to grade ≤1. If no improvement is seen, or the condition worsens by 4 weeks, both drugs should be held, and steroid treatment initiated. If AST/ALT >8 × ULN or bilirubin >5 × ULN, ipilimumab should be permanently discontinued. Manage subsequent events according to nivolumab guidelines. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue ipilimumab and hold nivolumab. Monitor with at least weekly LFTs until grade ≤2, then resume nivolumab. Continue with at least weekly LFTs until improvement to grade ≤1. Manage subsequent dose delays under Management/Next Dose for Nivolumab alone. If no improvement is seen, or the condition worsens by 4 weeks, hold nivolumab and initiate steroid treatment. |

Continued treatment of active immune mediated hepatitis may exacerbate ongoing inflammation. Holding drug to evaluate LFT changes and early treatment are recommended. LFT changes may occur during steroid tapers from other events and may occur together with other GI events including cholecystitis/pancreatitis.

**Note:** Grades for liver function follow multiples of ULN, rather than multiples of baseline.

Recommended management: see Hepatic AE management algorithm.

| Diarrhea<br>(immune related<br>enterocolitis) | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change. | No change. |
| Grade 2 | Hold nivolumab until ≤ grade 1. Treat symptomatically, and resume nivolumab if improved to ≤ grade 1, at investigator's discretion. If after 4 weeks no improvement is seen, the condition worsens, or colitis is documented by colonoscopy, permanently discontinue nivolumab therapy and initiate steroid treatment. | Hold both drugs until ≤grade 1. Treat symptomatically, and resume both drugs if improved to ≤ grade 1, at investigator's discretion. If after 4 weeks, no improvement is seen, the condition worsens, or colitis is documented by colonoscopy, permanently discontinue ipilimumab and manage according to nivolumab guidelines. |
| Grade 3 | Hold nivolumab until ≤ grade 1 and obtain colonoscopy. Treat symptomatically, and resume nivolumab if colonoscopy shows no colitis and patient improves to ≤ grade 1, at investigator's discretion. If after 4 weeks no improvement is seen, the condition worsens, or colitis is documented by colonoscopy, permanently discontinue nivolumab therapy and initiate steroid treatment. | Permanently discontinue ipilimumab. Hold nivolumab until ≤ grade 1 and obtain colonoscopy. Treat symptomatically, and resume nivolumab if colonoscopy shows no colitis and patient improves to ≤ grade 1, at investigator's discretion. If after 4 weeks no improvement is seen, the condition worsens, or colitis is documented by colonoscopy, permanently discontinue nivolumab therapy and initiate steroid treatment. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |

Patients with grade 2 symptoms but normal colonoscopy and biopsies may be retreated after resolution. Patients who require systemic steroids should be taken off study treatment. Evaluate pituitary function prior to starting steroids if possible without compromising acute care. Patients should be evaluated for additional causes including *C. diff*, acute and self-limited infectious and foodborne illness, ischemic bowel, diverticulitis, and IBD at the discretion of the treating physician.

Recommended management: see GI AE management Algorithm.

| Amylase/Lipase<br>Increased and<br>Pancreatitis | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1<br>(Amylase/Lipase<br>Increased Only) | Continue nivolumab therapy, if asymptomatic, at the investigator's discretion. | Continue both drugs, if asymptomatic, at the investigator's discretion. |
| Grade 2 | Continue nivolumab therapy, if asymptomatic, at the investigator's discretion. If symptomatic, resume nivolumab therapy once resolved. | Continue both drugs, if asymptomatic, at the investigator's discretion. If symptomatic, resume nivolumab and ipilimumab therapy once resolved. |
| Grade 3<br>Amylase/Lipase<br>Increased | Continue nivolumab, at the investigator's discretion. Monitor lipase and amylase once or twice weekly. Radiographic evaluation is optional if asymptomatic with no evidence of pancreatitis-associated gallbladder disease, no evidence of worsening, or no new onset of DM. | Continue both drugs, at the investigator's discretion. Monitor lipase and amylase once or twice weekly. Radiographic evaluation is optional if asymptomatic with no evidence of pancreatitis-associated gallbladder disease, no evidence of worsening, or no new onset of DM. |
| Grade 3<br>Pancreatitis | Continue nivolumab therapy, if asymptomatic, at investigator's discretion. Patients should have imaging done when clinically indicated ( <i>i.e.</i> , grade 3 pancreatitis) before resuming treatment. Patients who develop symptomatic pancreatitis or DM should permanently discontinue nivolumab therapy. | Continue both drugs, if asymptomatic, at investigator's discretion. Patients should have imaging done when clinically indicated ( <i>i.e.</i> , grade 3 pancreatitis) before resuming treatment. Patients who develop symptomatic pancreatitis or DM should permanently discontinue nivolumab and ipilimumab therapy. |
| Grade 4 | Hold nivolumab until grade 2. Resume if asymptomatic. Patients should have imaging done before resuming treatment, and when clinically indicated. Patients who develop symptomatic pancreatitis or DM should permanently discontinue nivolumab therapy. | Hold both drugs until grade 2. Resume if asymptomatic. Patients should have imaging done before resuming treatment, and when clinically indicated. Patients who develop symptomatic pancreatitis or DM should permanently discontinue nivolumab and ipilimumab therapy. |

Patients may develop symptomatic and radiologic evidence of pancreatitis as well as DM and diabetic ketoacidosis. Lipase elevation may occur during the period of steroid withdrawal and with other immune mediated events or associated with colitis, hepatitis, and patients who have asymptomatic lipase elevation typically have self-limited course and may be re-treated.

For treatment management of symptomatic pancreatitis please follow the Hepatic Adverse Event Management Algorithm

| Pneumonitis,<br>Bronchospasm,<br>Pulmonary<br>Toxicity, or<br>Interstitial Lung<br>Disease | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | Hold nivolumab pending evaluation and resolution to baseline, including baseline O <sub>2</sub> saturation. Resume after pulmonary and/or infectious disease consultation excludes lymphocytic pneumonitis. | Hold both drugs pending evaluation and resolution to baseline including baseline O <sub>2</sub> saturation. Resume after pulmonary and/or infectious disease consultation excludes lymphocytic pneumonitis. |
| Grade 2 | Hold nivolumab pending evaluation. Resume after pulmonary and/or infectious disease consultation excludes associated lymphocytic pneumonitis as the cause of the pneumonitis. Patients should permanently discontinue nivolumab therapy if steroids are required. | Hold both drugs pending evaluation. Resume after pulmonary and/or infectious disease consultation excludes ipilimumab and associated lymphocytic pneumonitis as the cause of the pneumonitis. Patients should permanently discontinue nivolumab and ipilimumab therapy if steroids are required. |
| Grade 3 | Hold nivolumab pending evaluation. Resume after pulmonary and/or infectious disease consultation excludes associated lymphocytic pneumonitis as the cause of the pneumonitis. Patients should permanently discontinue nivolumab therapy if steroids are required. | Hold both drugs pending evaluation. Resume after pulmonary and/or infectious disease consultation excludes ipilimumab and associated lymphocytic pneumonitis as the cause of the pneumonitis. Patients should permanently discontinue nivolumab and ipilimumab therapy if steroids are required. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |

Distinguishing inflammatory pneumonitis is often a diagnosis of exclusion for patients who do not respond to antibiotics and have no causal organism identified including influenza. Most patients with respiratory failure or hypoxia will be treated with steroids. Bronchoscopy may be required and analysis of lavage fluid for lymphocytic predominance may be helpful. Patients with new lung nodules should be evaluated for sarcoid like granuloma. Seasonal influenza killed vaccine is recommended for all patients. **The above does not include infusion reactions.** 

Recommended management: See Pulmonary Adverse Event Management Algorithm.

| Other GI<br>Nausea-Vomiting | Management/Next Dose for Nivolumab Monotherapy | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change. | No change. |
| Grade 2 | Hold nivolumab pending evaluation for gastritis duodenitis and other immune AEs or other causes. Resume after resolution to ≤ grade 1. | Hold both drugs pending evaluation for gastritis duodenitis and other immune AEs or other causes. Resume after resolution to ≤ grade 1. |
| Grade 3 | Hold nivolumab until resolution to ≤ grade 1. If symptoms do not resolve within 7 days with symptomatic treatment, permanently discontinue nivolumab therapy. | Hold both drugs until resolution to ≤ grade 1. If symptoms do not resolve within 7 days with symptomatic treatment, permanently discontinue nivolumab and ipilimumab therapy. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |

Patients with grade 2 or 3 nausea or vomiting should be evaluated for upper GI inflammation and other immune related events.

| <u>Fatigue</u> | Management/Next Dose for<br>Nivolumab Monotherapy | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 2 | No change in dose. | No change in dose. |
| Grade 3 | Hold until $\leq$ grade 2. | Permanently discontinue ipilimumab. Hold both drugs until ≤ grade 2, then resume both drugs. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue both drugs. |

Fatigue is the most common adverse event associated with immune checkpoint therapy. Fatigue  $\geq$  grade 2 should be evaluated for associated or underlying organ involvement including pituitary, thyroid, and hepatic, or muscle (CPK) inflammation.

| Neurological events | Management/Next Dose for Nivolumab Monotherapy | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | Hold pending evaluation and observation. Resume when resolved to baseline. | Hold both drugs pending evaluation and observation. Resume when resolved to baseline. |
| Grade 2 | Hold nivolumab pending evaluation and observation. Resume when improved to ≤ grade 1 or baseline. Patients should permanently discontinue nivolumab therapy if treatment with steroids is required. | Hold both drugs pending evaluation and observation. Resume when improved to ≤ grade 1 or baseline. Patients should permanently discontinue nivolumab and ipilimumab therapy if treatment with steroids is required. |
| Grade 3 | Permanently discontinue nivolumab therapy. | Permanently discontinue ipilimumab. Hold nivolumab until improved to ≤ grade 1 or baseline, then resume. Manage subsequent events according to nivolumab guidelines. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |
| Recommended management: See Neurologic Adverse Event Management Algorithm | | |

| Cardiac* | Management/Next Dose for Nivolumab or Nivolumab plus<br>Ipilimumab |
|---|---|
| ≤ Grade 1 | Hold dose pending evaluation.** Evaluate for signs and symptoms of CHF, ischemia, arrhythmia, or myositis. Obtain history EKG, CK (for concomitant myositis), and CK-MB. Repeat troponin, CK and EKG after 2-3 days. If troponin and labs normalize, patient may resume therapy. If labs worsen or symptoms develop then treat as below. |
| ≥ Grade 2 with suspected myocarditis | Hold dose pending evaluation.** Admit to hospital and consult with a cardiologist. Rule out MI and other causes of cardiac disease. Continue to monitor and obtain echocardiogram. Also consider cardiac MRI and a cardiac biopsy. Initiate high dose methylprednisolone. If no improvement is seen within 24 hours, add either infliximab, ATG, or tacrolimus. Resume therapy if there is a return to baseline AND myocarditis is excluded or considered unlikely. |
| ≥ Grade 2 with confirmed myocarditis | Permanently discontinue nivolumab and ipilimumab therapy and admit to CCU. Treat as above. Consider high dose methylprednisolone and electrophysiology consultation. Begin telemetry or event monitoring. Add ATG or tacrolimus if no improvement is seen. |

| Cardiac* | Management/Next Dose for Nivolumab or Nivolumab plus<br>Ipilimumab |
|---|---|
| Grade 4 | Permanently discontinue nivolumab or nivolumab and ipilimumab therapy. |

<sup>\*</sup> Including CHF, LV systolic dysfunction, Myocarditis, CPK elevation, and troponin.

<u>Note:</u> The optimal treatment regimen for immune mediated myocarditis has not been established. Since this toxicity has caused patient deaths, an aggressive approach is recommended.

| Endocrine<br>(Hypophysitis,<br>Adrenal<br>Insufficiency, Type<br>1 Diabetes) | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab and Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change. | No change. |
| Grade 2-3 | Hold until ≤ grade 1 and patients are on a stable replacement hormone regimen. If treated with steroids, patients must be stable off steroids for 2 weeks. | Hold both drugs until ≤ grade 1 and patients are on a stable replacement hormone regimen. If treated with steroids, patients must be stable off steroids for 2 weeks. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |

<u>Note:</u> Symptomatic pituitary enlargement, exclusive of hormone deficiency, but including severe headache or enlarged pituitary on MRI should be considered a grade 3 event. Isolated thyroid or testosterone deficiency may be treated as grade 2 if there are no other associated deficiencies and adrenal function is monitored. Evaluate pituitary function before beginning steroid therapy or hormone replacement therapy of any kind.

<u>Note:</u> Patients with thyroiditis may be re-treated on replacement therapy. Patients must be evaluated to rule out pituitary disease prior to initiating thyroid hormone replacement.

Recommended management: See Endocrinopathy Management Algorithm.

| Nephritis<br>(Creatinine<br>Increased*) | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change. | No change. |
| Grade 2-3 | Hold until $\leq$ grade 1, then resume. | Hold both drugs until $\leq$ grade 1, then resume. |

<sup>\*\*</sup> Patients with evidence of myositis without myocarditis may be treated according to "other event."

| Nephritis<br>(Creatinine<br>Increased*) | S | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue both drugs. |

<sup>\*</sup> Rule out noninflammatory (non-immune-mediated) causes. If cause is non-inflammatory, treat accordingly and continue immunotherapy.

Patients with fever should be evaluated as clinically appropriate. Isolated fever may occur during infusion reactions or up to several days after infusion. Evaluate over 1-2 weeks for other autoimmune events that may present as fever.

Recommended management: See Renal AE Management Algorithm.

| Infusion/<br>Hypersensitivity<br>reactions* | Management/Next Dose for Nivolumab and Nivolumab plus<br>Ipilimumab |
|---|---|
| ≤ Grade 1 | Remain at bedside and monitor patient until symptoms recover. Infusion rate may be slowed or interrupted and restarted at 50% of the original infusion rate when symptoms resolve; if no further complications ensue after 30 minutes, the rate may be increased to 100% of the original rate. Monitor patient closely. The following pre-medications are recommended at least 30 minutes before future infusions: diphenhydramine 50 mg (or equivalent) and/or acetaminophen/paracetamol 325-1000 mg. Slowing the infusion rate as above is also recommended. |
| Grade 2 | Stop infusion, begin an IV infusion of normal saline, and treat the patient with diphenhydramine 50 mg IV (or equivalent) and/or acetaminophen/paracetamol 325-1000 mg; remain at bedside and monitor patient until symptoms resolve. Corticosteroid ( <i>e.g.</i> hydrocortisone 50-100 mg) and/or bronchodilator therapy may also be administered as appropriate if reaction is severe or patient does not respond to diphenhydramine or acetaminophen. When symptoms resolve, restart infusion at 50% of the original rate; if no further complications ensue after 30 minutes, the rate may be increased to 100% of the original infusion rate. Monitor patient closely. If symptoms recur, then no further drug should be administered at that visit. Administer diphenhydramine 50 mg IV, remain at bedside, and monitor the patient until symptoms resolve. The amount of study drug infused must be recorded on the CRF. The following prophylactic premedications are recommended at least 30 minutes before future study drug administrations: diphenhydramine 50 mg (or equivalent) and/or acetaminophen/paracetamol 325-1000 mg. If those are not sufficient to |

| Infusion/<br>Hypersensitivity<br>reactions* | Management/Next Dose for Nivolumab and Nivolumab plus<br>Ipilimumab |
|---|---|
| | prevent infusion reactions, corticosteroids (up to 25 mg of methylprednisolone or equivalent) may be used. |
| Grade 3 or 4 | <ul> <li>Immediately discontinue infusion. Begin an IV infusion of normal saline and treat the patient as follows:</li> <li>Bronchodilators (recommended) such as epinephrine 0.2-1 mg of a 1:1000 solution for subcutaneous administration or 0.1-0.25 mg of a 1:10,000 solution injected slowly for IV administration;</li> <li>diphenhydramine 50 mg IV;</li> <li>methylprednisolone 100 mg IV (or equivalent), as needed.</li> </ul> Patient should be monitored until the investigator is comfortable that the symptoms will not recur. Permanently discontinue nivolumab therapy in patients on nivolumab and permanently discontinue both ipilimumab and nivolumab in patients on the combination. Investigators should follow their institutional guidelines for the treatment of anaphylaxis. Remain at bedside and monitor patient until recovery. In case of late-occurring hypersensitivity symptoms, symptomatic treatment may be given (e.g., oral antihistamine or corticosteroids). |

<sup>\*</sup> Manifestation may include fever, chills, rigors, headache, rash, pruritus, arthralgia, hypotension, hypertension, and/or bronchospasm.

All Grade 3 or 4 infusion reactions should be reported within 24 hours to the Study Chair or co-Chair AND reported as an SAE if criteria are met. Infusion reactions should be graded according to NCI CTCAE v5.0 guidelines.

Note: Treatment guidelines may be modified based local institutional standards, as appropriate.

| Fever | Management/Next Dose for<br>Nivolumab Monotherapy | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | Evaluate and continue nivolumab therapy. | Evaluate and continue both drugs. |
| Grade 2-3 | Hold until $\leq$ grade 1, then resume nivolumab. | Hold both drugs until $\leq$ grade 1, then resume both drugs. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue both drugs. |

Patients with fever should be evaluated as clinically appropriate. Patients may experience isolated fever during infusion reactions or up to several days after infusion. Evaluation over the course of 1-2 weeks should be done for other autoimmune events that may present as fever.

Also consult the guidelines for infusion reactions, above.

| All Other Events | Management/Next Dose for<br>Nivolumab | Management/Next Dose for<br>Nivolumab plus Ipilimumab |
|---|---|---|
| ≤ Grade 1 | No change in dose. | No change in dose. |
| Grade 2 | Hold nivolumab until ≤ grade 1 or baseline (exceptions as noted below) then resume nivolumab. | Hold both drugs until ≤ grade 1 or baseline (exceptions as noted below), then resume both drugs. |
| Grade 3 | Hold nivolumab until ≤ grade 1 or baseline, then resume nivolumab. | Permanently discontinue ipilimumab. Hold nivolumab until ≤ grade 1 or baseline, then resume nivolumab alone. |
| Grade 4 | Permanently discontinue nivolumab therapy. | Permanently discontinue nivolumab and ipilimumab therapy. |
| Recommended management: As clinically indicated. | | |

If a patient has any AE, laboratory abnormality, or intercurrent illness which, in the judgment of the investigator, presents a substantial clinical risk to the patient with continued study drug dosing should go off protocol treatment.

If a patient has any grade 3 or 4 drug-related laboratory abnormality (except those mentioned above) or electrolyte abnormality, that can be managed indecently from the underlying organ pathology with electrolyte replacement, hormone replacement, insulin, or that does not require treatment **does not** require discontinuation.

If treatment is delayed >4 weeks for an AE, nivolumab or nivolumab and ipilimumab therapy should be permanently discontinued.

Patients with grade 3 thyroiditis and skin rash may continue therapy as for grade 2 events with resolution and stable replacement treatment.

Patients with thyroiditis or hypopituitarism who are stable as above may be restarted with replacement hormones including thyroid hormone and physiologic doses of corticosteroids. Please note that grading for hypophysitis with symptoms of headache, visual or neurologic changes or radiologic evidence of pituitary enlargement and other CNS events such as aseptic meningitis or encephalitis should be considered grade 3 events.

Any patients who require additional immune suppressive treatment beyond steroids should go off study treatment

Patients requiring more than two dose delays for the same event should permanently discontinue nivolumab or nivolumab and ipilimumab therapy.

Prior to starting corticosteroids or hormone replacement for any reason, appropriate endocrine testing including cortisol, ACTH, TSH and T4 must be obtained to document baseline.

Please note that in some cases the treatment algorithms recommend steroids if symptoms do not resolve in 7 days. However, this recommendation is not meant to delay steroid treatment at any time it is clinically indicated.

Doses may be delayed for evaluation and patients may resume depending on results. Any patient started on corticosteroids initially who is determined to not require steroid treatment for an autoimmune adverse event may resume therapy after a 2-week observation period without further symptoms at the discretion of the treating investigator.

#### 8. PHARMACEUTICAL INFORMATION

A list of the adverse events and potential risks associated with the investigational agents administered in this study can be found in Section 10.1.

## 8.1 CTEP IND Agents

8.1.1 XL184 (cabozantinib), NSC 761968

**Chemical Name:** *N*-{4-[(6,7-dimethoxyquinolin-4-yl)oxy]phenyl}-*N*'-(4-fluorophenyl) cyclopropane-1,1-dicarboxamide, (2S)-hydroxybutanedioate

Other Names: Cabozantinib s-malate, EXEL-7184, EXEL-02977184, Cabometyx®

**Classification:** Receptor Tyrosine Kinases Inhibitor (RTK)

CAS Registry Number: 1140909-48-3

Molecular Formula: C28H24FN3O5·C4H6O5 M.W.: 635.6 Daltons (L-malate salt)

**Mode of Action:** XL184 (cabozantinib) inhibits multiple RTKs implicated in tumor growth, metastasis, and angiogenesis, and targets primarily MET and VEGFR2. Other targets are VEGFR3, RET, AXL, KIT, TIE-2, FLT-3, ROS1, and RON.

**How Supplied:** Exelixis supplies and the PMB, CTEP, DCTD, NCI distributes XL184 (cabozantinib) tablets. The composition of the tablets is listed in the table below. The yellow film-coated tablets are available in the following free-base equivalent strengths and bottle configurations:

1. 20 mg: round (5.6 mm); 30 tablets per HDPE bottle

XL184 (cabozantinib) Tablet Components and Composition

| Ingredient | Function | % w/w |
|---|---|---|
| XL184 (cabozantinib) malate (25% drug load as cabozantinib) | Active Ingredient | 31.7 |
| Microcrystalline Cellulose (Avicel PH-102) | Filler | 38.9 |
| Lactose Anhydrous (60M) | Filler | 19.4 |
| Hydroxypropyl Cellulose (EXF) | Binder | 3.0 |
| Croscarmellose Sodium (Ac-Di-Sol) | Disenegrant | 6.0 |
| Colloidal Silicon Dioxide, | Glidant | 0.3 |
| Magnesium Stearate | Lubricant | 0.75 |
| Opadry Yellow Film Coating which includes: | | |
| • HPMC 2910 / Hypromellose 6 cp | | |
| Titanium dioxide | Film Coating | 4.00 |
| • Triacetin | C | |
| <ul> <li>Iron Oxide Yellow</li> </ul> | | |

**Storage:** Store intact bottles at controlled room temperature 20°C to 25°C (68°F to 77°F); temperature excursions are permitted between 15°C and 30°C (59°F to 86°F) [see USP Controlled Room Temperature].

If a storage temperature excursion outside of 15°C and 30°C (59°F to 86°F) is identified, promptly return XL184 (cabozantinib) to 20°C to 25°C (68°F to 77°F) and quarantine the supplies. Provide a detailed report of the excursion (including documentation of temperature monitoring and duration of the excursion) to <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> for determination of suitability.

**Stability:** Refer to the drug label for expiration date. Dispense XL184 (Cabozantinib) in original bottles.

#### However, if dispensing the exact quantity of cabozantinib tablets is an institutional guideline:

- Removing the extra tablets from the original bottle is allowed, and it must be used within 30 days of the preparation date. Document the extra tablets as waste in Oral DARF.
- Adding additional cabozantinib tablets into the original bottle in which the original bottle is exceeding its 30 Count bottle, is **Not Allowed**.

Repackaging XL184 (cabozantinib) for a short period of time is acceptable and limited to:

- Up to 24 hours when dispensed in an open container such as a pill cup.
- Up to 7 days when dispensed in a closed container (e.g., a pharmacy dispensing bottle).

#### Route of Administration: Oral.

**Method of Administration**: Take XL184 (cabozantinib) on an empty stomach; *i.e.*, do not eat 2 hours before and 1 hour after each dosing. Take the dose with a full glass of water at approximately the same time each day. Do not crush or chew. Do not take a missed dose within 12 hours of the next dose.

## **Potential Drug Interactions:**

#### CYP450 isozymes:

In vitro, XL184 (cabozantinib) is a substrate of CYP3A4 and a weak substrate of CYP2C9. In healthy volunteers, XL184 (cabozantinib) AUC increased 38% with co-administration of ketoconazole, a strong inhibitor of CYP3A4, and decreased by 77% with a strong CYP3A4 inducer rifampin. Therefore, avoid chronic use of strong CYP3A4 inducers such as rifampin, dexamethasone, phenytoin, carbamazepine, rifabutin, rifapentine, phenobarbital, and St. John's Wort while taking XL184 (cabozantinib). Avoid chronic use of strong CYP3A4 inhibitors such as ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, and ritonavir. Use alternative medications.

**Note:** Use caution when discontinuing medication that is a strong inducer of CYP3A4 in patients who have been on stable doses of XL184 (cabozantinib), as this could significantly increase the exposure to XL184 (cabozantinib).

XL184 (cabozantinib) is a noncompetitive inhibitor of CYP2C8 ( $K_{iapp} = 4.6 \, \mu M$ ), a mixed-type inhibitor of both CYP2C9 ( $K_{iapp} = 10.4 \, \mu M$ ) and CYP2C19 ( $K_{iapp} = 28.8 \, \mu M$ ), and a weak competitive inhibitor of CYP3A4 (estimated  $K_{iapp} = 282 \, \mu M$ ) in human liver microsomal (HLM) stability assays. IC<sub>50</sub> values >20  $\, \mu M$  were observed for CYP1A2, CYP2D6, and CYP3A4 isozymes. XL184 (cabozantinib) is an inducer of CYP1A1 mRNA in human hepatocyte incubations.

Avoid grapefruit, grapefruit juice, and Seville oranges while participating in this trial.

## P-glycoprotein/MRP2:

In vitro data indicate that XL184 (cabozantinib) is an inhibitor of P-glycoprotein transport activity (IC<sub>50</sub> =  $7.0 \mu M$ ). Co-administration of XL184 (cabozantinib) with a P-gp substrate may result in an increase in P-gp substrate plasma concentration. Therefore, use caution when administering XL-184 (cabozantinib) with drugs known to be P-gp substrates (e.g., fexofenadine, aliskiren, ambrisentan, digoxin, colchicine, maraviroc, posaconazole, tolvaptan, etc.).

XL184 (cabozantinib) is also a substrate of drug transporter MRP2, which may result in an increase plasma concentration of XL184 (cabozantinib) when administered with an inhibitor of MRP2. Use caution and monitor adverse events when administering XL184 (cabozantinib) with MRP2 inhibitors such as cyclosporine, delavirine, efavirenz, or emtricitabine.

## Protein binding:

XL184 (cabozantinib) is highly protein bound (≥99.9%). Use caution when co-administering XL184 (cabozantinib) with medications that are highly protein-bound (*e.g.*, diazepam, furosemide, dicloxacillin, or propranolol). Avoid administration of warfarin with XL184 (cabozantinib) as warfarin is highly protein-bound and has a very narrow therapeutic index.

## Antacids, H2-blockers, PPIs:

Co-administration of gastric pH modifying drugs such as PPI, H2-blockers, or antacids has no clinically-relevant effect on XL184 (cabozantinib) plasma PK in healthy volunteers; thus, concomitant use of these drugs with XL184 (cabozantinib) is allowed.

#### OTc prolongation:

Use caution when administering XL184 (cabozantinib) in patients with QT prolongation risk, a history of QT interval prolongation, or who are receiving antiarrhythmic drugs. Concomitant use of strong CYP3A4 inhibitors should be avoided as it may increase XL184 (cabozantinib) plasma concentrations. Refer to the protocol for QTcF criteria.

## **Potential Food Effect**

A high fat meal increased both XL184 (cabozantinib)  $C_{max}$  and AUC values by 41% and 57%, respectively, relative to fasted conditions. Therefore, XL184 (cabozantinib) should be taken on an empty stomach (fasting is required 2 hours before and 1 hour after each dose).

**Patient Care Implications**: Women of childbearing potential must use highly effective contraception while receiving XL184 (cabozantinib) and for 4 months after the last dose. Breastfeeding is not allowed while on study. Sexually active males must use highly effective contraception while on study and for 4 months after the last dose.

**Availability**: XL184 (cabozantinib) is an investigational agent supplied to investigators by the Division of Cancer Treatment and Diagnosis (DCTD), NCI.

If the study agent is provided by the NCI under a Collaborative Agreement with the agent manufacturer, the text below must be included in the protocol. Information on the study agent's Collaborative Agreement status will be provided in the approved LOI response letter.

XL184 (cabozantinib) is provided to the NCI under a Collaborative Agreement between the Pharmaceutical Collaborator and the DCTD, NCI (see Section 13.5).

## 8.1.2 Nivolumab (NSC 748726)

**Amino Acid Sequence:** 4 polypeptide chains, which include 2 identical heavy chains with 440 amino acids and 2 identical light chains.

Other Names: BMS-936558, MDX1106

Classification: Anti-PD-1 mAb

**M.W.:** 146,221 Daltons

**Mode of Action:** Nivolumab targets the PD-1, CD279 cell surface membrane receptor. PD-1 is a negative regulatory receptor expressed by activated T and B lymphocytes. Binding of PD-1 to its ligands, PD-L1 and PD-L2, results in the down-regulation of lymphocyte activation. Nivolumab inhibits the binding of PD-1 to PD-L1 and PD-L2. Inhibition of the interaction between PD-1 and its ligands promotes immune responses and antigen-specific T-cell responses to both foreign antigens as well as self-antigens.

**Description:** Nivolumab Injection is a clear to opalescent, colorless to pale yellow liquid; light (few) particulates may be present. The drug product is a sterile, nonpyrogenic, single-use, isotonic aqueous solution formulated in sodium citrate dihydrate, sodium chloride, mannitol, diethylenetriaminepentacetic acid (pentetic acid), polysorbate 80 (Tween® 80), and water for injection. Dilute solutions of hydrochloric acid and/or sodium hydroxide may be used for pH adjustment (pH 5.5-6.5).

**How Supplied:** Nivolumab is supplied by Bristol-Myers Squibb (BMS) and distributed by the Pharmaceutical Management Branch (PMB), CTEP/DCTD/NCI as 100 mg vials (10 mg/mL) with a 0.7 mL overfill. It is supplied in 10 mL type I flint glass vials, with fluoropolymer film-laminated rubber stoppers and aluminum seals.

**Preparation:** Nivolumab injection can be infused undiluted (10 mg/mL) or diluted with 0.9% Sodium Chloride Injection, USP or 5% Dextrose. When the dose is based on patient weight (*i.e.*, mg/kg), nivolumab injection can be infused undiluted or diluted to protein concentrations as low as 0.35 mg/mL. When the dose is fixed (*e.g.*, 240 mg, 360 mg, or 480 mg flat dose), nivolumab injection can be infused undiluted or diluted so as not to exceed a total infusion volume of 160 mL. For patients weighing less than 40 kg, the total volume of infusion must not exceed 4 mL per kg of patient weight. During drug product preparation and handling, vigorous mixing or shaking is to be avoided.

Nivolumab infusions are compatible with polyvinyl chloride (PVC) or polyolefin containers and infusion sets, and glass bottles.

**Storage:** Vials of Nivolumab injection must be stored at 2-8 °C (36-46 °F) and protected from light and freezing. The unopened vials can be stored at room temperature (up to 25 °C, 77 °F) and room light for up to 48 hours.

If a storage temperature excursion is identified, promptly return Nivolumab to 2-8 °C (36-46 °F) and quarantine the supplies. Provide a detailed report of the excursion (including documentation of temperature monitoring and duration of the excursion) to <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> for determination of suitability.

**Stability:** Shelf-life surveillance of the intact vials is ongoing. The administration of undiluted and diluted solutions of nivolumab must be completed within 24 hours of preparation. If not used immediately, the infusion solution may be stored up to <u>7 days</u> in a refrigerator at 2°-8°C (36°46°F) and a maximum of 8 hours of the total <u>7 days</u> can be at room temperature (up to 25°C, 77°F) and room light. The maximum 8-hour period under room temperature and room light conditions includes the product administration period.

**CAUTION:** The single-use dosage form contains no antibacterial preservative or bacteriostatic agent. Therefore, it is advised that the product be discarded 8 hours after initial entry.

**Route of Administration:** Intravenous infusion over 30 minutes. Do not administer as an IV push or bolus injection.

**Method of Administration:** Administer through a 0.2 micron to 1.2-micron pore size, low-protein binding (polyethersulfone membrane) in-line filter.

**Potential Drug Interactions:** The indirect drug-drug interaction potential of nivolumab was assessed using systemic cytokine modulation data for cytokines known to modulate CYP enzymes. There were no meaningful changes in cytokines known to have indirect effects on CYP enzymes across all dose levels of nivolumab. This lack of cytokine modulation suggests that nivolumab has no or low potential for modulating CYP enzymes, thereby indicating a low risk of therapeutic protein-drug interaction.

**Patient Care Implications:** WOCBP receiving nivolumab must continue contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are

sexually active with WOCBP must continue contraception for a period of 7 months after the last dose of nivolumab.

**Availability:** Nivolumab is an investigational agent supplied to investigators by the Division of Cancer Treatment and Diagnosis (DCTD), NCI.

If the study agent is provided by the NCI under a Collaborative Agreement with the agent manufacturer, the text below must be included in the protocol. Information on the study agent's Collaborative Agreement status will be provided in the approved LOI response letter.

Nivolumab is provided to the NCI under a Collaborative Agreement between the Pharmaceutical Collaborator and the DCTD, NCI (see Section 13.5).

8.1.3 Ipilimumab (NSC 732442)

**Other Names:** BMS-734016, BMS-734016-01, Anti-CTLA-4 monoclonal antibody, MDX-010, Yervov<sup>TM</sup>

Classification: Human monoclonal antibody

**M.W.:** 147,991 Daltons

**Mode of Action:** CTLA-4 is a negative regulator of T-cell activity. Ipilimumab is a mAb that binds to CTLA-4 and blocks the interaction of CTLA-4 with its ligands, CD80/CD86. Blockade of CTLA-4 has been shown to augment T cell activation and proliferation, including the activation and proliferation of tumor-infiltrating T-effector cells. Inhibition of CTLA-4 signaling can also reduce Treg function, which may contribute to a general increase in T-cell responsiveness, including the anti-tumor response.

**Description:** Ipilimumab (BMS-734016, MDX-010) is a fully human  $IgG1\kappa$  consisting of 4 polypeptide chains; 2 identical heavy chains primarily consisting of 447 amino acids each with 2 identical kappa light chains consisting of 215 amino acids each linked through inter-chain disulfide bonds. Ipilimumab is produced from cell culture using a Chinese Hamster Ovary (CHO) cell line.

**How Supplied:** Bristol-Myers-Squibb (BMS) supplies Ipilimumab to the Pharmaceutical Management Branch, CTEP/DCTD/NCI. Ipilimumab injection, 200 mg/40 mL (5 mg/mL), is packaged in a 50-cc Type I flint molded glass vials, stoppered with 20-mm gray butyl rubber stoppers, and sealed with 20-mm aluminum flip-off seals. Each vial includes a 2.6-mL overfill for vial, needle, and syringe holdup.

**Preparation:** Do not shake. Allow the vials to stand at room temperature for approximately 5 minutes prior to preparation of infusion. Ipilimumab is given undiluted or further diluted in 0.9% NaCl Injection, USP or 5% Dextrose Injection, USP in concentrations between 1 mg/mL and 4 mg/mL. Ipilimumab is stable in a polyvinyl chloride (PVC), non-PVC/non DEHP (di-(2-ethylhexyl) phthalate) IV bag or glass container up to 24 hours refrigerated at (20 to 80 C) or at room temperature/ room light.

Recommended safety measures for preparation and handling include protective clothing, gloves, and safety cabinets.

**Storage:** Store intact vials refrigerated at (2<sup>0</sup> to 8<sup>0</sup> C), protected from light. Do not freeze.

**Stability:** Refer to the package label for expiration. Solution as described above is stable up to 24 hours refrigerated at  $(2^0 \text{ to } 8^0 \text{ C})$  or at room temperature/ room light.

*CAUTION:* Ipilimumab does not contain antibacterial preservatives. Use prepared IV solution immediately. Discard partially used vials.

**Route of Administration:** Intravenous infusion at the protocol-specific rate. Do not administer ipilimumab as an IV push or bolus injection.

**Method of Administration:** Can use a volumetric pump to infuse ipilimumab at the protocol-specific dose(s) and rate(s) via a PVC IV infusion set with an in-line, sterile, non-pyrogenic, low-protein-binding filter (0.2 micron to 1.2 micron).

**Patient Care Implications:** Monitor patients for immune-related adverse events, *e.g.*, rash/vitiligo, diarrhea/colitis, uveitis/episcleritis, hepatitis, and hypothyroidism. If you suspect toxicity, refer to the protocol guidelines for ruling out other causes.

Women of childbearing potential should be advised to continue contraception for 3 months following the last dose of Ipilimumab.

Post-marketing surveillance identified a fatal toxic epidermal necrolysis (TEN) event in a patient who received ipilimumab after experiencing a severe or life-threatening skin adverse reaction on a prior cancer immune stimulating therapy. Caution should be used when considering the use of ipilimumab in a patient who has previously experienced a severe or life-threatening skin adverse reaction on a prior cancer immune stimulating therapy.

**Availability:** Ipilimumab (BMS-734016, MDX-010) is an investigational agent supplied to investigators by the Division of Cancer Treatment and Diagnosis (DCTD), NCI.

If the study agent is provided by the NCI under a Collaborative Agreement with the agent manufacturer, the text below must be included in the protocol. Information on the study agent's Collaborative Agreement status will be provided in the approved LOI response letter.

Ipilimumab (BMS-734016, MDX-010) is provided to the NCI under a Collaborative Agreement between the Pharmaceutical Collaborator and the DCTD, NCI (see Section 13.5).

## 8.1.4 Agent Ordering and Agent Accountability

8.1.4.1 NCI-supplied agents may be requested by eligible participating Investigators (or their authorized designee) at each participating institution. The CTEP-assigned protocol

number must be used for ordering all CTEP-supplied investigational agents. The eligible participating investigators at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA Form 1572 (Statement of Investigator), NCI Biosketch, Agent Shipment Form, and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP-supplied investigational agents for the study should be ordered under the name of one lead participating investigator at that institution.

Sites may request a starter supply (2 bottles of cabozantinib 20 mg, 4 vials of ipilimumab, and 5 vials of nivolumab) once a patient is in screening.

Submit agent requests through the PMB AURORA application. Access to AURORA requires the establishment of credentials necessary to access secure NCI Clinical Oncology Research Enterprise (CORE) systems, maintenance of an "active" account status, a "current" password, and active person registration status. For questions about drug orders, transfers, returns, or accountability, call or email PMB any time or use the dialog function in AURORA to communicate with PMB staff. Refer to the PMB's website for specific policies and guidelines related to agent management.

8.1.4.2 <u>Agent Inventory Records</u> – The investigator, or a responsible party designated by the investigator, must maintain a complete accountability of the receipt, dispensing and final disposition of all agents received from the PMB using the appropriate NCI Investigational Agent (Drug) Accountability Record (DARF) available on the CTEP forms page. Store and maintain separate NCI Investigational Agent Accountability Records for each agent, strength, formulation and ordering investigator on this protocol.

Product Quality Complaint (PQC): A product quality complaint is defined as any suspicion of a product defect related to a potential quality issue during manufacturing, packaging, release testing, stability monitoring, dose preparation, storage or distribution of the product, or delivery system. Not all PQCs involve a study subject. Lot or batch numbers are of high significance and need to be provided where and when possible. PQC must be reported to the PMB as soon as the PQC is identified. Report PQC to PMB at <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> or by using the dialog function in AURORA to communicate with PMB staff.

## 8.1.5 Material Safety Data Sheets

The current versions of the material safety data sheets (MSDS or SDS) for PMB-distributed agents will be accessible to site investigators and research staff through the PMB AURORA application. Questions about MSDS access may be directed to the PMB at <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> or by using the dialog function in AURORA to communicate with PMB staff.

## 8.1.6 Investigator Brochure Availability

The current versions of the IBs for the agents will be accessible to site investigators and research staff through the PMB AURORA application. Access to AURORA requires the establishment of credentials necessary to access secure NCI Clinical Oncology Research Enterprise (CORE) systems, maintenance of an "active" account status, a "current" password and active person registration status. Questions about IB access may be directed to the PMB IB Coordinator via email.

## 8.1.7 <u>Useful Links and Contacts</u>

- CTEP Forms, Templates, Documents: http://ctep.cancer.gov/forms/
- NCI CTEP Investigator Registration: <u>RCRHelpDesk@nih.gov</u>
- PMB policies and guidelines: http://ctep.cancer.gov/branches/pmb/agent\_management.htm
- PMB Online Agent Order Processing (OAOP) application: <a href="https://ctepcore.nci.nih.gov/OAOP">https://ctepcore.nci.nih.gov/OAOP</a> PMB Agent Inventory Management System (AURORA) application: <a href="https://ctepcore.nci.nih.gov/aurora/login">https://ctepcore.nci.nih.gov/aurora/login</a>
- CTEP Identity and Access Management (IAM) account: <a href="https://ctepcore.nci.nih.gov/iam/">https://ctepcore.nci.nih.gov/iam/</a>
- CTEP IAM account help: <a href="mailto:ctepreghelp@ctep.nci.nih.gov">ctepreghelp@ctep.nci.nih.gov</a>
- IB Coordinator: <a href="mailto:IBCoordinator@mail.nih.gov">IBCoordinator@mail.nih.gov</a>
- PMB email: PMBAfterHours@mail.nih.gov
- PMB phone and hours of service: (240) 276-6575 Monday through Friday between 8:30 am and 4:30 pm (ET)

## 8.1.8 Agent Shortages

Specific guidance on how to address agent shortages for patients already enrolled on a clinical study as well as how to manage potential enrollment of new patients is provided at https://ctep.cancer.gov/branches/pmb/drug\_shortages.htm.

Treatment plan modifications being made to avoid immediate hazard to patients is permissible under the Department of Health and Human Services (HHS) regulations at 45 CFR 46.103(b)(4)(iii). In accordance with HHS regulations, local investigators must promptly inform the IRB of record of this unanticipated problem and the management plan for the trial.

#### 9. STATISTICAL CONSIDERATIONS

## 9.1 Study Design/Endpoints

This phase 2 study has a two-stage Simon minimax design with a primary endpoint of overall response rate (ORR) (complete responses [CRs] plus partial responses [PRs]). The hypothesis of the study is that combination of XL184 (cabozantinib), nivolumab, and ipilimumab improves ORR in the treatment of poorly differentiated neuroendocrine carcinomas, after the failure of at least one line of prior systemic cancer treatment, to more than 45%. The null hypothesis is a 45% true response rate versus alternative hypothesis of 70% true response. This design will have a type 1 error of 0.10 and 90% power ( $\beta$ =0.10). The response rate will be determined by the number of patients, each, who reach a PR or CR within 6 months of their initiation of treatment.

For the primary objective, the binary endpoint will be the achievement of either a CR or a PR (yes/no). Response will be determined via the RECIST v1.1 criteria (See Section 12.0). The relevant statistical endpoint will be the CR+PR rate, evaluated for all registered patients, and for all response-evaluable (r-e) patients. The r-e population is defined as patients who receive at least one dose of the study drugs, have measurable disease at baseline, and have at least 1 post-baseline disease assessment. CR+PR rate will be summarized with a point estimate and a 2-sided Wilson type CI estimate. These two estimates will be made for all registered and for all r-e patients. For the primary and the interim analyses, the confirmed responses need to be seen within 6 months of treatment initiation. Further patient enrollment may be suspended while already enrolled patients continue their treatment until the needed response rate is observed as described below in Section 9.2. Patients already on treatment will continue their treatment as long as any criterion for discontinuation is not met.

The study design will include the following interim safety analysis. If 4 or fewer of the first 15 patients experience a delay in any of the study therapies, lasting at least four weeks, due to toxicity, or is discontinued due to toxicity, and the first stage response target (*i.e.* at least 7 out of 15 achieved an objective response) is reached, the trial could proceed to the second stage. However, if at least 5 of the first 15 patients experience such a treatment delay or discontinuation (and the first stage response target is reached), accrual would remain suspended and these findings would need to be discussed with CTEP. Note that if the first stage response target is not reached, the study would be closed due to futility, regardless of the level of toxicity.

This is not a stratified study design, although the primary organ of origin, if known and morphologic description of the poorly differentiated NECs (small cell, large cell or mixed histology) will be recorded, when available, for descriptive purposes.

## 9.2 Sample Size/Accrual Rate

The overall sample size is 25 patients. In order to allow for occasional ineligibility or response inevaluability, this trial will have a maximum accrual goal of 30 patients. Stage 1 will recruit up to 18 patients to obtain 15 eligible and treated patients, and Stage 2 (if needed) will recruit up to 12 patients to obtain 10 eligible and treated patients. If there are 7 or more objective responses in Stage 1, the study will advance to Stage 2, otherwise the study will be terminated early for

futility. Accrual will be suspended to allow assessment of response among the last few Stage 1 patients (until an objective response is observed or a total of 6 months have elapsed since the accrual of the last patient in stage 1, whichever comes first). After completing Stage 2, if among the resulting 25 evaluable patients, there are 15 or more objective responses (an objective response rate of  $\geq$  60%), the combination will be recommended for further evaluation. Otherwise, the 3-drug combination will be deemed to have insufficient efficacy in this study population.

Under the null hypothesis, the study design has an average sample number (ASN) of 19.10 patients, and a probability of early termination (PET) of 0.452. Its sample sizes, Stage-specific response milestones, and operating characteristics were computed using the "Two-Stage Phase II Clinical Trials" program in PASS 2019 software.

The estimated accrual rate for this trial is 1 patient per month.

#### PLANNED ENROLLMENT REPORT

| DOMESTIC PLANNED ENROLLMENT REPORT (TREATMENT) | | | | | |
|---|---|---|---|---|---|
| | Ethnic Categories | | | | |
| Racial Categories | Not Hispanic or Latino | | Hispanic or Latino | | Total |
| | Female | Male | Female | Male | |
| American Indian/ Alaska<br>Native | 0 | 0 | 0 | 0 | 0 |
| Asian | 1 | 1 | 0 | 0 | 2 |
| Native Hawaiian or<br>Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |
| Black or African<br>American | 2 | 1 | 0 | 0 | 3 |
| White | 10 | 9 | 1 | 1 | 21 |
| More Than One Race | 1 | 1 | 0 | 0 | 2 |
| Total | 14 | 12 | 1 | 1 | 28 |
| INTERNATIONAL (including Canadian participants) PLANNED ENROLLMENT REPORT (TREATMENT) | | | | | |
|---|---|---|---|---|---|
| | | Ethnic Cat | egories | | |
| Racial Categories | Not Hispani | c or Latino | Hispanic | or Latino | Total |
| | Female | Male | Female | Male | |
| American Indian/ Alaska<br>Native | 0 | 0 | 0 | 0 | 0 |
| Asian | 0 | 0 | 0 | 0 | 0 |
| Native Hawaiian or<br>Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |
| Black or African<br>American | 0 | 0 | 0 | 0 | 0 |
| White | 1 | 1 | 0 | 0 | 2 |
| More Than One Race | 0 | 0 | 0 | 0 | 0 |
| Total | 1 | 1 | 0 | 0 | 2 |

#### 9.3 Stratification Factors

N/A

# 9.4 Analysis of Secondary Endpoints

#### 9.4.1 PFS

The hypothesis is that the combination of XL184 (cabozantinib), nivolumab, and ipilimumab will improve PFS to more than 4 months. Censored PFS will be determined for all registered patients. the censored time-to-event distributions of PFS will be analyzed with standard Kaplan-Meier methodology. Point and CI estimates of the median and various time point-specific rates will be derived from the K-M life table. Censored PFS will be analyzed for all registered patients

9.4.2 Safety and tolerability of the XL184 (cabozantinib), nivolumab, and ipilimumab combination.

Safety including specific toxicity types, grades, and attributions will be evaluated and summarized. Toxicity will be assessed in all toxicity-evaluable (t-e) patients using the CTCAE

5.0 criteria as defined in Section 12.0. The t-e population is defined as all patients who have received the study treatment. The resulting binary endpoints of each toxicity type at a specific grade(s), will all be summarized with point estimates and 2-sided Wilson type CI estimates. The grade of each type of toxicity will also be summarized with 1-way frequency distributions.

# 9.4.3 DCR

The hypothesis is that the combination of XL184 (cabozantinib), nivolumab, and ipilimumab will improve DCR to more than 50%. The binary endpoint of DCR will be defined as the achievement of either CR, or PR, or SD (yes/no). The resulting binary endpoints of DCR will all be summarized with point estimates and 2-sided Wilson type CI estimates. DCR estimates will be calculated for all r-e patients.

#### 9.4.4 DOR

DOR is measured from the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease, the smallest measurements recorded since the treatment started). The censored time-to-event distributions of DOR will be analyzed with standard Kaplan-Meier methodology. Point and CI estimates of the median and various time point-specific rates will be derived from the Kaplan-Meier life table. Censored DOR will be analyzed for the combination of all patients who achieve either a CR or a PR

#### 9.4.5 Correlative Studies

To determine effects of the combination of XL184 (cabozantinib), nivolumab and ipilimumab on multiple biomarkers of disease or treatment, analysis of available paired tumor biopsy samples will be done using methods that include but are not limited to IHC of intratumoral immune cells and flow cytometry. The antibodies that will be used for the IHC assays are listed below.

| Antigen | Clone | Manufacturer | Cat. No. | Regulatory Status | Target cell |
|---|---|---|---|---|---|
| CD4 | 4B12 | DAKO | M731001-2 | IVD | CD4 T cell |
| CD8a | C8/144B | DAKO | M710301-2 | IVD | CD8 T cell |
| Foxp3 | EP340 | Cell Marque | AC-0304RUOC | IVD | |
| PD-1 | NAT105 | Cell Marque | 315M | IVD | |
| IFN-g | B27 | BD Biosciences | 550011 | RUO | |
| PD-L1 | 22C3 | DAKO | M3653 | IVD | |
| Elastase | NP57 | DAKO | M075201-2 | IVD | TAN |
| CD68 | PG-M1 | DAKO | M087601-2 | IVD | TAM |
| CD163 | MRQ-26 | Cell Marque | 163M | IVD | TAM |
| Arg1 | SP156 | Cell Marque | 380R | IVD | |

For all correlative objectives, the continuously distributed correlative endpoints (CD8+ T lymphocytes, MDSC, and TAM) will be summarized with descriptive statistics (N, mean, standard deviation, median, interquartile range (IQR), minimum, maximum, and a CI for the mean). Statistical graphics (*e.g.*, box plots, dot plots, *etc.*) will also be created to illustrate the distributions of the various correlative endpoints. All of these descriptive statistical analyses and graphical analyses will be performed separately for: a) the pre-treatment biopsy correlatives; b) the on-treatment biopsy correlatives; and c) the pre/post biopsy difference in the correlatives.

# 9.5 Reporting and Exclusions

# 9.5.1 Evaluation of Toxicity

All patients will be evaluable for toxicity from the time of their first treatment with any of the three investigational agents - XL184 (cabozantinib), nivolumab, or ipilimumab.

All toxicities will be graded as per NCI CTCAE version 5.0. Toxicity evaluation will be done at the start of each cycle for as long as the patient is on active treatment.

Patients who experience a Grade 3 or greater toxicity that is attributed to study medication and cannot be ameliorated by the use of adequate medical intervention should have their treatment interrupted until the toxicity improves to a Grade 2 or lower severity. Patients may subsequently be re-started on the study drugs, including at a reduced dose for XL184 (cabozantinib).

# 9.5.2 Evaluation of Response

All patients included in the study must be assessed for response to treatment, even if there are major protocol treatment deviations or if they are ineligible. Each patient will be assigned one of the following categories: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data). [Note: By arbitrary convention, category 9 usually designates the "unknown" status of any type of data in a clinical database.]

All of the patients who met the eligibility criteria (with the possible exception of those who received no study medication) should be included in the main analysis of the response rate. Patients in response categories 4-9 should be considered to have a treatment failure (disease progression). Thus, an incorrect treatment schedule or drug administration does not result in exclusion from the analysis of the response rate. Precise definitions for categories 4-9 will be protocol specific.

All conclusions should be based on all eligible patients. Subanalyses may then be performed on the basis of a subset of patients, excluding those for whom major protocol deviations have been identified (e.g., early death due to other reasons, early discontinuation of treatment, major protocol violations, etc.). However, these subanalyses may not serve as the basis for drawing conclusions concerning treatment efficacy, and the reasons for excluding patients from the analysis should be clearly reported. The 95% confidence intervals should also be provided.

#### 10. ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS

Adverse event (AE) monitoring and reporting is a routine part of every clinical trial. The following list of AEs (Section 10.1) and the characteristics of an observed AE (Sections 10.2 and 10.3) will determine whether the event requires expedited reporting via the Medidata Rave in addition to routine reporting.

# 10.1 Comprehensive Adverse Events and Potential Risks Lists (CAEPRs)

#### 10.1.1 XL184 (cabozantinib)

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements' <a href="http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aeguidelines.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aeguidelines.pdf</a> for further clarification. *Frequency is provided based on 3219 patients*. Below is the CAEPR for XL184 (Cabozantinib).

**NOTE:** Report AEs on the SPEER <u>ONLY IF</u> they exceed the grade noted in parentheses next to the AE in the SPEER. If this CAEPR is part of a combination protocol using multiple investigational agents and has an AE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

Version 2.5, August 29, 20241 Adverse Events with Possible Specific Protocol Relationship to XL184 (Cabozantinib) Exceptions to Expedited (CTCAE 5.0 Term) Reporting (SPEER) [n= 3219] Likely (>20%) Less Likely (<=20%) Rare but Serious (<3%) BLOOD AND LYMPHATIC SYSTEM DISORDERS Anemia ENDOCRINE DISORDERS Endocrine disorders - Other (thyroid dysfunction) Hypothyroidism (Gr 2) Hypothyroidism GASTROINTESTINAL DISORDERS Abdominal pain (Gr 3) Abdominal pain Constipation (Gr 2) Constipation Diarrhea Diarrhea (Gr 3) Dry mouth Drv mouth (Gr 2) Dyspepsia (Gr 2) Dyspepsia Gastrointestinal fistula<sup>2</sup> Gastrointestinal hemorrhage<sup>3</sup> Gastrointestinal perforation4 Mucositis oral (Gr 3) Mucositis oral Nausea (Gr 3) Nausea Oral pain (Gr 2) Oral pain Vomiting (Gr 3) Vomiting

| Re | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | | | |
| GENERAL DISORDERS AN | ID ADMINISTRATION SITE CO | NDITIONS | |
| | Edema limbs | | |
| Fatigue | | | Fatigue (Gr 3) |
| INFECTIONS AND INFEST | | | |
| | Infection <sup>5</sup> | | |
| INJURY, POISONING AND | PROCEDURAL COMPLICATION | | |
| | | Wound complication | |
| INVESTIGATIONS | | | |
| | Alanine aminotransferase increased | | Alanine aminotransferase increased (Gr 3) |
| | Aspartate aminotransferase increased | | Aspartate aminotransferase increased (Gr 3) |
| | Lipase increased | | Lipase increased (Gr 4) |
| | Platelet count decreased | | Platelet count decreased (Gr 3) |
| Weight loss | | | Weight loss (Gr 3) |
| METABOLISM AND NUTRI | TION DISORDERS | | |
| Anorexia | | | Anorexia (Gr 3) |
| | Dehydration | | |
| | Hypocalcemia | | |
| | Hypokalemia | | |
| | Hypomagnesemia | | |
| | Hypophosphatemia | | |
| MUSCULOSKELETAL AND | CONNECTIVE TISSUE DISOR | RDERS | |
| | Arthralgia | | |
| | Generalized muscle weakness | | |
| | Muscle cramp | | |
| | Musculoskeletal and connective tissue disorder - Other (bone metaphyseal dysplasia) | | |
| | | Osteonecrosis of jaw | |
| L<br>NERVOUS SYSTEM DISOF | Pain in extremity | | |
| INERVOUS SYSTEM DISOR | | | |
| Dyegousia | Dizziness | | Dysgeusia (Gr 2) |
| Dysgeusia | Headache | | bysgeusia (Gi Z) |
| | Troductie | Intracranial hemorrhage | |
| | 1 | Ischemia cerebrovascular | |
| | | Reversible posterior leukoencephalopathy syndrome | |
| | 1 | Stroke | |
| | | Transient ischemic attacks | |
| RENAL AND URINARY DIS | ORDERS | | |
| | Hematuria | | |
| | | Proteinuria | |
| RESPIRATORY, THORACIO | C AND MEDIASTINAL DISORD | | |
| | Cough | | |
| | Dyspnea | | |

| Rel | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | | Pneumothorax <sup>6</sup> | |
| | | Respiratory fistula <sup>7</sup> | |
| | Respiratory hemorrhage8 | | |
| | Voice alteration | | Voice alteration (Gr 3) |
| SKIN AND SUBCUTANEOUS | S TISSUE DISORDERS | | |
| | Alopecia | | |
| | Dry skin | | Dry skin (Gr 2) |
| | Hair color changes | | Hair color changes (Gr 1) |
| Palmar-plantar erythrodysesthesia syndrome | | | Palmar-plantar<br>erythrodysesthesia |
| erythodysestriesia syndrome | | | syndrome (Gr 3) |
| | Rash maculo-papular | | Rash maculo-papular (Gr 3) |
| VASCULAR DISORDERS | | • | |
| Hypertension | | | Hypertension (Gr 3) |
| | Thromboembolic event9 | | |

<sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <a href="PIO@CTEP.NCI.NIH.GOV">PIO@CTEP.NCI.NIH.GOV</a>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>2</sup>Gastrointestinal fistula includes Anal fistula, Colonic fistula, Duodenal fistula, Esophageal fistula, Enterovesical fistula, Gastric fistula, Gastrointestinal fistula, Ileal fistula, Jejunal fistula, Oral cavity fistula, Pancreatic fistula, Rectal fistula, and Salivary gland fistula under the GASTROINTESTINAL DISORDERS SOC.

<sup>3</sup>Gastrointestinal hemorrhage includes Anal hemorrhage, Cecal hemorrhage, Colonic hemorrhage, Duodenal hemorrhage, Esophageal hemorrhage, Esophageal varices hemorrhage, Gastric hemorrhage, Hemorrhoidal hemorrhage, Ileal hemorrhage, Intra-abdominal hemorrhage, Jejunal hemorrhage, Lower gastrointestinal hemorrhage, Oral hemorrhage, Pancreatic hemorrhage, Rectal hemorrhage, Retroperitoneal hemorrhage, and Upper gastrointestinal hemorrhage under the GASTROINTESTINAL DISORDERS SOC.

<sup>4</sup>Gastrointestinal perforation includes Colonic perforation, Duodenal perforation, Esophageal perforation, Gastric perforation, Ileal perforation, Jejunal perforation, Rectal perforation, and Small intestinal perforation under the GASTROINTESTINAL DISORDERS SOC.

<sup>5</sup>Infection includes all 75 sites of infection under the INFECTIONS AND INFESTATIONS SOC.

<sup>6</sup>Pneumothorax has been observed at a higher than expected frequency (15-20%) in a study treating patients with relapsed Ewing sarcoma and osteosarcoma all of whom had pulmonary metastases.

<sup>7</sup>Respiratory fistula includes Bronchial fistula, Bronchopleural fistula, Laryngeal fistula, Pharyngeal fistula, Pulmonary fistula, and Tracheal fistula under the RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS SOC.

<sup>8</sup>Respiratory hemorrhage includes Bronchopulmonary hemorrhage, Epistaxis, Hemoptysis, Laryngeal hemorrhage, Mediastinal hemorrhage, Pharyngeal hemorrhage, and Pleural hemorrhage under the RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS SOC.

Adverse events reported on XL184 (Cabozantinib) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that XL184 (Cabozantinib) caused the adverse event:

**BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Blood and lymphatic system disorders - Other (pancytopenia); Disseminated intravascular coagulation; Eosinophilia; Febrile neutropenia; Hemolytic uremic syndrome

**CARDIAC DISORDERS** - Atrial fibrillation; Atrioventricular block complete; Cardiac arrest; Cardiac disorders - Other (hypokinetic cardiomyopathy); Chest pain - cardiac; Heart failure; Left ventricular systolic dysfunction; Myocardial infarction; Myocarditis; Sinus bradycardia; Sinus tachycardia; Supraventricular tachycardia

EAR AND LABYRINTH DISORDERS - Hearing impaired; Vertigo

ENDOCRINE DISORDERS - Endocrine disorders - Other (autoimmune thyroiditis); Endocrine disorders - Other (thyroiditis); Endocrine disorders - Other (thyrotoxicosis); Hyperthyroidism; Hypopituitarism EYE DISORDERS - Blurred vision; Cataract; Eye disorders - Other (corneal epithelium defect)
GASTROINTESTINAL DISORDERS - Abdominal distension; Anal fissure; Anal mucositis; Anal pain; Anal ulcer; Cheilitis; Colitis; Colonic obstruction; Duodenal ulcer; Dysphagia; Enterocolitis; Esophageal ulcer; Esophagitis; Flatulence; Gastric ulcer; Gastroesophageal reflux disease; Gastrointestinal disorders - Other (glossitis); Gastrointestinal disorders - Other (pneumoperitoneum); Gastrointestinal pain; Gingival pain; Hemorrhoids; Ileus; Pancreatitis; Periodontal disease; Rectal pain; Rectal ulcer; Toothache
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Chills; Death NOS; Edema face; Fever; Gait disturbance; General disorders and administration site conditions - Other (general physical health deterioration); General disorders and administration site conditions - Other (implant site inflammation); Hypothermia; Malaise; Multi-organ failure; Non-cardiac chest pain; Pain; Sudden death NOS

**HEPATOBILIARY DISORDERS** - Budd-Chiari syndrome; Cholecystitis; Hepatic failure; Hepatobiliary disorders - Other (cholelithiasis); Hepatobiliary disorders - Other (hepatic cirrhosis); Hepatobiliary disorders - Other (hepatic thrombus); Hepatobiliary disorders - Other (hepatitis toxic); Hepatobiliary disorders - Other (hepatorenal syndrome); Portal vein thrombosis

**IMMUNE SYSTEM DISORDERS** - Allergic reaction; Anaphylaxis; Autoimmune disorder **INJURY, POISONING AND PROCEDURAL COMPLICATIONS** - Fall; Injury, poisoning and procedural complications - Other (post procedural hemorrhage); Injury, poisoning and procedural complications - Other (tendon injury); Wound dehiscence; Wrist fracture

**INVESTIGATIONS** - Alkaline phosphatase increased; Blood bilirubin increased; Blood lactate dehydrogenase increased; CPK increased; Cardiac troponin I increased; Creatinine increased; Ejection fraction decreased; Electrocardiogram QT corrected interval prolonged; GGT increased; Investigations - Other (D-dimer); Investigations - Other (urine ketone body present); Lymphocyte count decreased; Neutrophil count decreased; Serum amylase increased; Thyroid stimulating hormone increased; White blood cell decreased

**METABOLISM AND NUTRITION DISORDERS** - Glucose intolerance; Hyperglycemia; Hypernatremia; Hyperuricemia; Hyponatremia; Metabolism and nutrition disorders - Other (failure to thrive); Metabolism and nutrition disorders - Other (hypoproteinemia)

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Back pain; Buttock pain; Chest wall pain; Flank pain; Muscle weakness lower limb; Musculoskeletal and connective tissue disorder - Other (muscle hemorrhage); Myalgia; Neck pain; Osteonecrosis; Osteoporosis; Rhabdomyolysis

NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (lip and/or oral cavity cancer); Tumor hemorrhage; Tumor pain

<sup>&</sup>lt;sup>9</sup>Thromboembolic event includes pulmonary embolism which may be life-threatening.

NERVOUS SYSTEM DISORDERS - Ataxia; Cognitive disturbance; Concentration impairment; Dysarthria; Dysesthesia; Dysphasia; Encephalopathy; Lethargy; Memory impairment; Nervous system disorders -Other (hemiparesis); Nervous system disorders - Other (vocal cord paralysis); Peripheral motor neuropathy; Peripheral sensory neuropathy; Presyncope; Seizure; Somnolence; Spinal cord compression: Syncope

PSYCHIATRIC DISORDERS - Anxiety; Confusion; Delirium; Depression; Hallucinations; Insomnia; Psychiatric disorders - Other (mental status changes)

RENAL AND URINARY DISORDERS - Acute kidney injury; Chronic kidney disease; Glucosuria; Renal and urinary disorders - Other (hemorrhage urinary tract); Urinary tract obstruction

REPRODUCTIVE SYSTEM AND BREAST DISORDERS - Pelvic pain; Reproductive system and breast disorders - Other (scrotal ulcer/erythema/edema); Scrotal pain; Vaginal fistula; Vaginal inflammation; Vaginal perforation

RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - Adult respiratory distress syndrome; Allergic rhinitis; Atelectasis; Hoarseness; Hypoxia; Laryngeal edema; Oropharyngeal pain; Pharyngeal mucositis; Pleural effusion; Pneumonitis; Productive cough; Pulmonary hypertension; Respiratory failure; Respiratory, thoracic and mediastinal disorders - Other (nasal septum perforation); Respiratory, thoracic and mediastinal disorders - Other (pneumomediastinum); Respiratory, thoracic and mediastinal disorders - Other (rales); Sore throat

SKIN AND SUBCUTANEOUS TISSUE DISORDERS - Erythema multiforme; Nail changes; Pain of skin; Pruritus; Rash acneiform; Skin and subcutaneous tissue disorders - Other (pain, sloughing of skin and erythema); Skin and subcutaneous tissue disorders - Other (psoriasis); Skin hypopigmentation; Skin ulceration

VASCULAR DISORDERS - Hematoma; Hypotension; Superior vena cava syndrome; Vascular disorders - Other (bleeding varicose vein); Vasculitis

Note: XL184 (Cabozantinib) in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

10.1.2 Nivolumab

# Comprehensive Adverse Events and Potential Risks list (CAEPR) for Nivolumab (NSC 748726)

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements' http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aeguidelines.pdf for

further clarification. Frequency is provided based on 2069 patients. Below is the CAEPR for Nivolumab.

**NOTE**: Report AEs on the SPEER **ONLY** IF they exceed the grade noted in parentheses next to the AE in the SPEER. If this CAEPR is part of a combination protocol using multiple investigational agents and has an AE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

**Version 2.4, December 2, 2020**<sup>1</sup> **Adverse Events with Possible Specific Protocol** Relationship to Nivolumab **Exceptions to Expedited** (CTCAE 5.0 Term) Reporting (SPEER) [n=2069]Less Likely (<=20%) Rare but Serious (<3%) Likely (>20%) BLOOD AND LYMPHATIC SYSTEM DISORDERS Anemia Anemia (Gr 3) CARDIAC DISORDERS Cardiac disorders - Other (cardiomyopathy) Myocarditis Pericardial tamponade<sup>2</sup> Pericarditis ENDOCRINE DISORDERS Adrenal insufficiency<sup>3</sup> Hyperthyroidism<sup>3</sup> Hypophysitis<sup>3</sup> Hypothyroidism<sup>3</sup> EYE DISORDERS Blurred vision Dry eye Eye disorders - Other (diplopia)<sup>3</sup> Eve disorders - Other (Graves ophthalmopathy)<sup>3</sup> Eye disorders - Other (optic neuritis retrobulbar)<sup>3</sup> Eve disorders - Other (Vogt-Koyanagi-Harada) Uveitis GASTROINTESTINAL DISORDERS Abdominal pain Abdominal pain (Gr 2) Colitis<sup>3</sup> Colonic perforation<sup>3</sup> Diarrhea Diarrhea (Gr 3) Dry mouth Dry mouth (Gr 2) Enterocolitis Gastritis Mucositis oral

Nausea

Nausea (Gr 2)

| | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Pancreatitis <sup>4</sup> | | |
| | S AND ADMINISTRATION | N SITE CONDITIONS | - (5 A) |
| Fatigue | | | Fatigue (Gr 3) |
| | Fever | | Fever (Gr 2) |
| | Injection site reaction | | Injection site reaction (Gr 2) |
| HEPATOBILIARY DIS | ORDERS | | |
| | | Hepatobiliary disorders -<br>Other (immune-mediated<br>hepatitis) | |
| IMMUNE SYSTEM DI | SORDERS | | |
| | | Allergic reaction <sup>3</sup> | |
| | | Autoimmune disorder <sup>3</sup> | |
| | | Cytokine release<br>syndrome <sup>5</sup> | |
| | | Immune system disorders - Other (GVHD in the setting of allotransplant) <sup>3,6</sup> | |
| | | Immune system disorders - Other (sarcoidosis) <sup>3</sup> | |
| INJURY. POISONING | AND PROCEDURAL COM | | |
| | Infusion related reaction <sup>7</sup> | | |
| INVESTIGATIONS | | | |
| | Alanine aminotransferase increased <sup>3</sup> | | Alanine<br>aminotransferase<br>increased <sup>3</sup> (Gr 3) |
| | Aspartate<br>aminotransferase<br>increased <sup>3</sup> | | Aspartate<br>aminotransferase<br>increased <sup>3</sup> (Gr 3) |
| | Blood bilirubin increased <sup>3</sup> | | Blood bilirubin<br>increased³ (Gr 2) |
| | CD4 lymphocytes decreased | | CD4 lymphocyte<br>decreased (Gr 4) |
| | Creatinine increased | | |
| | Lipase increased Lymphocyte count decreased | | Lymphocyte count<br>decreased (Gr 4) |

| | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Neutrophil count | | |
| | decreased | | |
| | Platelet count decreased | | |
| | Serum amylase increased | | |
| METABOLISM AND N | NUTRITION DISORDERS | 1 | |
| | Anorexia | | |
| | | Hyperglycemia | Hyperglycemia (Gr 2) |
| | | Metabolism and nutrition | |
| | | disorders - Other (diabetes mellitus with | |
| MUSCUI OSVELETAI | L AND CONNECTIVE TISS | ketoacidosis) <sup>3</sup> | |
| MOSCOLOSKELETAL | Arthralgia | OE DISORDERS | |
| | Attiliaigia | Musculoskeletal and | |
| | | connective tissue disorder | |
| | | - Other (polymyositis) | |
| | | Myositis | |
| | | Rhabdomyolysis | |
| NERVOUS SYSTEM D | DISORDERS | 1 | |
| | | Encephalopathy <sup>3</sup> | |
| | | Facial nerve disorder <sup>3</sup> | |
| | | Guillain-Barre syndrome <sup>3</sup> | |
| | | Myasthenia gravis <sup>3</sup> | |
| | | Nervous system disorders | |
| | | - Other (demyelination | |
| | | myasthenic syndrome) | |
| | | Nervous system disorders | |
| | | - Other (encephalitis) <sup>3</sup> | |
| | | Nervous system disorders | |
| | | - Other | |
| | | (meningoencephalitis) | |
| | | Nervous system disorders | |
| | | - Other | |
| | | (meningoradiculitis) <sup>3</sup> | |
| | | Nervous system disorders | |
| | | - Other (myasthenic syndrome) | |

| Adverse Events with Possible Relationship to Nivolumab (CTCAE 5.0 Term) [n= 2069] | | | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | | Peripheral motor | |
| | | neuropathy | |
| | | Peripheral sensory | |
| | | neuropathy | |
| | | Reversible posterior | |
| | | leukoencephalopathy<br>syndrome <sup>3</sup> | |
| RENAL AND URINARY | V DISORDERS | syndrome | |
| REMAL AND URINAR | DISORDERS | Acute kidney injury <sup>3</sup> | |
| | | Renal and urinary | |
| | | disorders - Other | |
| | | (immune-mediated | |
| | | nephritis) | |
| RESPIRATORY, THOR | ACIC AND MEDIASTINA | | |
| , | Pleural effusion <sup>3</sup> | | |
| | Pneumonitis <sup>3</sup> | | |
| | | Respiratory, thoracic and mediastinal disorders - Other (bronchiolitis obliterans with organizing pneumonia) <sup>3</sup> | |
| SKIN AND SUBCUTAN | NEOUS TISSUE DISORDE | • | |
| | | Erythema multiforme <sup>3</sup> | |
| | Pruritus <sup>3</sup> | | Pruritus³ (Gr 2) |
| | Rash maculo-papular <sup>3</sup> | | Rash maculo-papular <sup>3</sup><br>(Gr 2) |
| | | Skin and subcutaneous | |
| | | tissue disorders - Other | |
| | | (bullous pemphigoid) | |
| | Skin and subcutaneous | | |
| | tissue disorders - Other<br>(Sweet's Syndrome) <sup>3</sup> | | |
| | Skin hypopigmentation <sup>3</sup> | | |
| | | Stevens-Johnson<br>syndrome | |
| | | Toxic epidermal necrolysis | |

<sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <u>PIO@CTEP.NCI.NIH.GOV</u>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>2</sup>Pericardial tamponade may be related to possible inflammatory reaction at tumor site.

<sup>3</sup>Nivolumab being a member of class of agents involved in the inhibition of "immune checkpoints", may result in severe and possibly fatal immune-mediated adverse events probably due to T-cell activation and proliferation. This may result in autoimmune disorders that can include (but are not limited to) autoimmune hemolytic anemia, acquired anti-factor VIII immune response, autoimmune aseptic meningitis, autoimmune hepatitis, autoimmune nephritis, autoimmune neuropathy, autoimmune thyroiditis, bullous pemphigoid, exacerbation of Churg-Strauss Syndrome, drug rash with eosinophilia systemic symptoms [DRESS] syndrome, facial nerve disorder (facial nerve paralysis), limbic encephalitis, hepatic failure, pure red cell aplasia, pancreatitis, ulcerative and hemorrhagic colitis, endocrine disorders (e.g., autoimmune thyroiditis, hyperthyroidism, hypothyroidism, autoimmune hypophysitis/hypopituitarism, thyrotoxicosis, and adrenal insufficiency), sarcoid granuloma, myasthenia gravis, polymyositis, and Guillain-Barre syndrome.

<sup>4</sup>Pancreatitis may result in increased serum amylase and/or more frequently lipase.

<sup>5</sup>Cytokine release syndrome may manifest as hemophagocytic lymphohistiocytosis with accompanying fever and pancytopenia.

<sup>6</sup>Complications including hyperacute graft-versus-host disease (GVHD), some fatal, have occurred in patients receiving allo stem cell transplant (SCT) after receiving Nivolumab. These complications may occur despite intervening therapy between receiving Nivolumab and allo-SCT.

<sup>7</sup>Infusion reactions, including high-grade hypersensitivity reactions which have been observed following administration of nivolumab, may manifest as fever, chills, shakes, itching, rash, hypertension or hypotension, or difficulty breathing during and immediately after administration of nivolumab.

Adverse events reported on Nivolumab trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that Nivolumab caused the adverse event:

# **BLOOD AND LYMPHATIC SYSTEM DISORDERS - Leukocytosis**

**CARDIAC DISORDERS** - Atrial fibrillation; Atrioventricular block complete; Heart failure; Ventricular arrhythmia

EAR AND LABYRINTH DISORDERS - Vestibular disorder

**EYE DISORDERS** - Eye disorders - Other (iridocyclitis); Optic nerve disorder; Periorbital edema

**GASTROINTESTINAL DISORDERS** - Constipation; Duodenal ulcer; Flatulence; Gastrointestinal disorders - Other (mouth sores); Vomiting

# $\textbf{GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS} - \textbf{Chills}; \ \textbf{Edema}$

limbs; Malaise; Pain

**HEPATOBILIARY DISORDERS** - Bile duct stenosis

**IMMUNE SYSTEM DISORDERS** - Anaphylaxis; Immune system disorders - Other (autoimmune thrombotic microangiopathy); Immune system disorders - Other (limbic encephalitis)

**INFECTIONS AND INFESTATIONS** - Bronchial infection; Lung infection; Sepsis; Upper respiratory infection

**INVESTIGATIONS** - Blood lactate dehydrogenase increased; GGT increased; Investigations - Other (protein total decreased); Lymphocyte count increased; Weight loss

METABOLISM AND NUTRITION DISORDERS - Dehydration; Hyperuricemia;

Hypoalbuminemia; Hypocalcemia; Hyponatremia; Hypophosphatemia

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Back pain;

Musculoskeletal and connective tissue disorder - Other (musculoskeletal pain); Musculoskeletal and connective tissue disorder - Other (polymyalgia rheumatica); Myalgia; Pain in extremity

NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND

**POLYPS)** - Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Histiocytic necrotizing lymphadenitis)

NERVOUS SYSTEM DISORDERS - Dizziness; Headache; Intracranial hemorrhage PSYCHIATRIC DISORDERS - Insomnia

**RENAL AND URINARY DISORDERS** - Hematuria; Renal and urinary disorders - Other (tubulointerstitial nephritis)

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Bronchospasm; Cough; Dyspnea; Hypoxia

**SKIN AND SUBCUTANEOUS TISSUE DISORDERS** - Alopecia; Dry skin; Hyperhidrosis; Pain of skin; Photosensitivity; Rash acneiform; Skin and subcutaneous tissue disorders - Other (rosacea)

VASCULAR DISORDERS - Flushing; Hypertension; Hypotension; Vasculitis

**Note**: Nivolumab in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

# 10.1.3 Ipilimumab

# Comprehensive Adverse Events and Potential Risks list (CAEPR) for Ipilimumab (MDX-010, NSCs 732442 and 720801)

Frequency is provided based on 2678 patients. Below is the CAEPR for Ipilimumab (MDX-010).

Version 2.10, March 29, 2019<sup>1</sup>

| | Adverse Events with Possible Relationship to Ipilimumab (MDX-010) (CTCAE 5.0 Term) [n= 2678] | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| BLOOD AND LYMP | PHATIC SYSTEM DISORDER | | |
| | | Blood and lymphatic<br>system disorders - Other<br>(acquired hemophilia) | |
| CARDIAC DISORDI | ERS | | |
| | Atrial fibrillation | | |
| | | Myocarditis <sup>2</sup> Pericardial effusion | |
| EAR AND LABYRIN | NTH DISORDERS | | |
| | Hearing impaired | | |
| ENDOCRINE DISOF | RDERS | | |
| | Adrenal insufficiency <sup>2</sup> | | |
| | Hyperthyroidism <sup>2</sup> | | |
| | Hypophysitis <sup>2</sup> | | |
| | Hypopituitarism <sup>2</sup> | | |
| | Hypothyroidism <sup>2</sup> | | |
| | Testosterone deficiency <sup>2</sup> | | |
| EYE DISORDERS | | | |
| | Eye disorders - Other (episcleritis) <sup>2</sup> | | |
| | Uveitis <sup>2</sup> | | |
| GASTROINTESTINA | | | |
| | Abdominal pain | | |
| | Colitis <sup>2</sup> | | Colitis <sup>2</sup> (Gr 3) |
| | | Colonic perforation <sup>3</sup> | |
| | Constipation | | |
| Diarrhea | | | Diarrhea (Gr 3) |
| | Enterocolitis | | |

| Adverse Events with Possible Relationship to Ipilimumab (MDX-010) (CTCAE 5.0 Term) [n= 2678] | | | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| ļ | Esophagitis | | |
| | | Ileus | |
| Nausea | 2 | | Nausea (Gr 3) |
| | Pancreatitis <sup>2</sup> | | |
| | Vomiting | | |
| GENERAL DISORDI | ERS AND ADMINISTRATIO | N SITE CONDITIONS | |
| | Chills | | |
| Fatigue | | | Fatigue (Gr 3) |
| | Fever | | Fever (Gr 2) |
| | | General disorders and | |
| | | administration site | |
| | | conditions - Other | |
| | | (Systemic inflammatory | |
| | | response syndrome [SIRS]) | |
| | | Multi-organ failure | |
| HEPATOBILIARY D | | į. | |
| | Hepatobiliary disorders -<br>Other (hepatitis) <sup>2</sup> | | |
| IMMUNE SYSTEM I | DISORDERS | | |
| | Autoimmune disorder <sup>2</sup> | | |
| | | Immune system disorders -<br>Other (GVHD in the<br>setting of allotransplant) <sup>4</sup> | |
| INFECTIONS AND I | NFESTATIONS | | |
| | | Infections and infestations - Other (aseptic meningitis) <sup>2</sup> | |
| INJURY, POISONING | G AND PROCEDURAL COM | • | |
| | Infusion related reaction | | |
| INVESTIGATIONS | | | |
| | Alanine aminotransferase increased | | |
| | Aspartate aminotransferase increased | | |
| | | Lymphocyte count decreased | |
| | Neutrophil count decreased | | |

| Adverse Events with Possible Relationship to Ipilimumab (MDX-010) (CTCAE 5.0 Term) [n= 2678] | | | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Weight loss | | |
| METABOLISM AND | NUTRITION DISORDERS | | |
| | Anorexia | | |
| | Dehydration | | |
| | Hyperglycemia | | |
| | | Metabolism and nutrition<br>disorders - Other<br>(exacerbation of pre-<br>existing diabetes mellitus) | |
| MUSCULOSKELETA | AL AND CONNECTIVE TISS | | |
| | Arthralgia<br>Arthritis | | |
| | | Generalized muscle<br>weakness | |
| | Musculoskeletal and<br>connective tissue disorder -<br>Other (polymyositis) <sup>2</sup> | | |
| NERVOUS SYSTEM | | | |
| | | Ataxia | |
| | Facial nerve disorder <sup>2</sup> | | |
| | Guillain-Barre syndrome <sup>2</sup> | | |
| | Headache | | |
| | Myasthenia gravis <sup>2</sup> | | |
| | | Nervous system disorders -<br>Other (immune-mediated<br>encephalitis) <sup>2</sup> | |
| | | Peripheral motor neuropathy | |
| | | Peripheral sensory neuropathy | |
| | Trigeminal nerve disorder | | |
| PSYCHIATRIC DISO | RDERS | | |
| | | Psychiatric disorders -<br>Other (mental status<br>changes) | |
| RENAL AND URINA | RY DISORDERS | | |
| | Acute kidney injury | | |

| Re | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Renal and urinary disorders -<br>Other (granulomatous<br>tubulointerstitial nephritis) | | |
| RESPIRATORY, THO | RACIC AND MEDIASTINAL | L DISORDERS | |
| | Pneumonitis | | |
| SKIN AND SUBCUTA | ANEOUS TISSUE DISORDER | 1 | |
| | <br> Pruritus | Erythema multiforme | Pruritus (Gr 3) |
| Rash maculo-papular | 111111111111111111111111111111111111111 | | Rash maculo-papular (Gr 3) |
| Tasa macato papara | Skin and subcutaneous tissue<br>disorders - Other (Sweet's<br>Syndrome) | | instructio paparar (Gr 5) |
| | | Stevens-Johnson syndrome | |
| | | Toxic epidermal necrolysis | |
| | Urticaria | | |
| VASCULAR DISORD | 1 | | |
| | Hypotension | | |

<sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <u>PIO@CTEP.NCI.NIH.GOV</u>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>2</sup>Ipilimumab can result in severe and fatal immune-mediated adverse events probably due to T-cell activation and proliferation. These can include (but are not limited to) autoimmune hemolytic anemia, acquired anti-factor VIII immune response, autoimmune aseptic meningitis, autoimmune hepatitis, autoimmune thyroiditis, hepatic failure, pure red cell aplasia, pancreatitis, ulcerative and hemorrhagic colitis, endocrine disorders (e.g., autoimmune thyroiditis, hyperthyroidism, hypothyroidism, autoimmune hypophysitis/hypopituitarism, and adrenal

insufficiency), ocular manifestations (e.g., uveitis, iritis, conjunctivitis, blepharitis, and episcleritis), sarcoid granuloma, myasthenia gravis, polymyositis, and Guillain-Barre syndrome. The majority of these reactions manifested early during treatment; however, a minority occurred weeks to months after discontinuation of ipilimumab especially with the initiation of additional treatments.

<sup>3</sup>Late bowel perforations have been noted in patients receiving MDX-010 (ipilimumab) in association with subsequent IL-2 therapy.

<sup>4</sup>Complications including hyperacute graft-versus-host disease (GVHD), may occur in patients receiving allo stem cell transplant (SCT) after receiving Ipilimumab (MDX-010). These complications may occur despite intervening therapy between receiving Ipilimumab (MDX-010) and allo-SCT.

<sup>5</sup>In rare cases diplopia (double vision) has occurred as a result of muscle weakness (Myasthenia gravis).

<sup>6</sup>Gastrointestinal hemorrhage includes Anal hemorrhage, Cecal hemorrhage, Colonic hemorrhage, Duodenal hemorrhage, Esophageal hemorrhage, Esophageal varices hemorrhage, Gastric hemorrhage, Hemorrhoidal hemorrhage, Ileal hemorrhage, Intra-abdominal hemorrhage, Jejunal hemorrhage, Lower gastrointestinal hemorrhage, Oral hemorrhage, Pancreatic hemorrhage, Rectal hemorrhage, Retroperitoneal hemorrhage, and Upper gastrointestinal hemorrhage under the GASTROINTESTINAL DISORDERS SOC.

<sup>7</sup>Infection includes all 75 sites of infection under the INFECTIONS AND INFESTATIONS SOC.

Adverse events reported on Ipilimumab (MDX-010) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that Ipilimumab (MDX-010) caused the adverse event:

**BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Anemia; Blood and lymphatic system disorders - Other (pure red cell aplasia)<sup>2</sup>; Febrile neutropenia

**CARDIAC DISORDERS** - Conduction disorder; Restrictive cardiomyopathy **EYE DISORDERS** - Extraocular muscle paresis<sup>5</sup>; Eye disorders - Other (retinal pigment changes)

GASTROINTESTINAL DISORDERS - Colonic ulcer; Dyspepsia; Dysphagia; Gastrointestinal disorders - Other (gastroenteritis); Gastrointestinal hemorrhage<sup>6</sup>; Proctitis GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Flu like symptoms; Non-cardiac chest pain

**HEPATOBILIARY DISORDERS** - Hepatic failure<sup>2</sup>

IMMUNE SYSTEM DISORDERS - Allergic reaction

**INFECTIONS AND INFESTATIONS** - Infection<sup>7</sup>

**INVESTIGATIONS** - Creatinine increased; Investigations - Other (rheumatoid factor); Lipase increased; Platelet count decreased; Serum amylase increased; White blood cell decreased **METABOLISM AND NUTRITION DISORDERS** - Tumor lysis syndrome

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Back pain; Joint range of motion decreased; Myalgia; Pain in extremity

NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - Tumor pain

**NERVOUS SYSTEM DISORDERS** - Dizziness; Dysphasia; Ischemia cerebrovascular; Seizure **PSYCHIATRIC DISORDERS** - Anxiety; Confusion; Depression; Insomnia

**RENAL AND URINARY DISORDERS - Proteinuria** 

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Allergic rhinitis; Cough; Dyspnea; Laryngospasm

**SKIN AND SUBCUTANEOUS TISSUE DISORDERS** - Alopecia; Dry skin; Hyperhidrosis; Skin hypopigmentation

**VASCULAR DISORDERS** - Flushing; Hypertension; Vascular disorders - Other (temporal arteritis)

**Note**: Ipilimumab (BMS-734016; MDX-010 Transfectoma-derived) in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

# 10.2 Adverse Event Characteristics

• CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP website <a href="http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm">http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm</a>.

# • For expedited reporting purposes only:

- AEs for the <u>agent</u> that are **bold and italicized** in the CAEPR (*i.e.*, those listed in the SPEER column, Section 10.1) should be reported through Medidata Rave only if the grade is above the grade provided in the SPEER.

#### • **Attribution** of the AE:

- Definite The AE *is clearly related* to the study treatment.
- Probable The AE *is likely related* to the study treatment.
- Possible The AE *may be related* to the study treatment.
- Unlikely The AE *is doubtfully related* to the study treatment.
- Unrelated The AE *is clearly NOT related* to the study treatment.

# 10.3 Expedited Adverse Event Reporting

10.3.1 Rave-CTEP-AERS Integration

The Rave Cancer Therapy Evaluation Program Adverse Event Reporting System (CTEP-AERS) integration enables evaluation of Adverse Events (AEs) entered in Rave to

determine whether they require expedited reporting and facilitates entry in CTEP-AERS for those AEs requiring expedited reporting. Sites must initiate all AEs for this study in Medidata Rave.

Treatment-emergent AEs: All AEs that occur after start of treatment are collected in Medidata Rave using the Adverse Event form, which is available for entry at each treatment course or reporting period and is used to collect AEs that start during the period or persist from the previous reporting period. AEs that occur 30 days after the last administration of the investigational agent/intervention are collected using the Late Adverse Event form.

Prior to sending AEs through the rules evaluation process, site staff should verify the following on the Adverse Event form in Rave:

- The reporting period (course/cycle) is correct, and
- AEs are recorded and complete (no missing fields) and the form is query free.

The CRA reports AEs in Rave at the time the Investigator learns of the event. If the CRA modifies an AE, it must be re-submitted for rules evaluation.

Upon completion of AE entry in Medidata Rave, the CRA submits the AE for rules evaluation by completing the Expedited Reporting Evaluation form (*i.e.*, checking the box *Send All AEs for Evaluation* and save the form). Both NCI and protocol-specific reporting rules evaluate the AEs submitted for expedited reporting. A report is initiated in CTEP-AERS using information entered in Medidata Rave for AEs that meet reporting requirements. The CRA completes the report by accessing CTEP-AERS via a direct link on the Medidata Rave Expedited Reporting Evaluation form. Contact the CTSU Help Desk at 1-888-823-5923 or by email at ctsucontact@westat.com if you have any issues submitting an expedited report in CTEP-AERS.

In the rare occurrence that internet connectivity is lost, a 24-hour notification is to be made to CTEP by telephone at 301-897-7497. Once internet connectivity is restored, the 24-hour notification that was phoned in must be entered immediately into CTEP-AERS using the direct link from Medidata Rave.

Additional information about the CTEP-AERS integration is available on the CTSU members' website:

- Study specific documents: *Protocols > Documents> Protocol Related Documents> Adverse Event Reporting*, and
- Additional resources: Resources > CTSU Operations Information > User Guides & Help Topics.

NCI requirements for SAE reporting are available on the CTEP website:

• NCI Guidelines for Investigators: Adverse Event Reporting Requirements is

available at

https://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf.

# 10.3.2 <u>Distribution of Adverse Event Reports</u>

CTEP-AERS is programmed for automatic electronic distribution of reports to the following individuals: Principal Investigator and Adverse Event Coordinator(s) (if applicable) of the Corresponding Organization or Lead Organization, the local treating physician, and the Reporter and Submitter. CTEP-AERS provides a copy feature for other e-mail recipients.

# 10.3.3 Expedited Reporting Guidelines

Use the NCI protocol number and the protocol-specific patient ID assigned during trial registration on all reports.

Note: A death on study requires <u>both</u> routine and expedited reporting, regardless of causality. Attribution to treatment or other cause must be provided.

Death due to progressive disease should be reported as **Grade 5 "Disease progression"** in the system organ class (SOC) "General disorders and administration site conditions." Evidence that the death was a manifestation of underlying disease (*e.g.*, radiological changes suggesting tumor growth or progression: clinical deterioration associated with a disease process) should be submitted.

Phase 1 and Early Phase 2 Studies: Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND/IDE within 30 Days of the Last Administration of the Investigational Agent/Intervention <sup>1, 2</sup>

#### FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

NOTE: Investigators MUST immediately report to the sponsor (NCI) ANY SAEs, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64).

An AE is considered serious if it results in ANY of the following outcomes:

- 1) Death
- 2) A life-threatening AE
- 3) An AE that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours.
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SAEs</u> that meet the above criteria <u>MUST</u> be immediately reported to the NCI via CTEP-AERS within the timeframes detailed in the table below.

| Grade 1-2 Timeframes | Grade 3-5 Timeframes |
|---|---|
| 24-Hour notification, 10 Calendar Days | 24-Hour notification, 5 Calendar Days |

**NOTE:** Protocol-specific exceptions to expedited reporting of SAEs are found in the Specific Protocol Exceptions to Expedited Reporting (SPEER) portion of the CAEPR.

#### **Expedited AE reporting timeframes are defined as:**

- "24-Hour notification, 5 Calendar Days" The SAE must initially be reported via CTEP-AERS within 24 hours of learning of the SAE, followed by a complete expedited report within 5 calendar days of the initial 24-hour report.
- "24-Hour notification, 10 Calendar Days" The SAE must initially be reported via CTEP-AERS within 24 hours of learning of the SAE, followed by a complete expedited report within 10 calendar days of the initial 24-hour report.

<sup>1</sup>SAEs that occur more than 30 days after the last administration of investigational agent/intervention and have an attribution of possible, probable, or definite require reporting as follows:

#### Expedited 24-Hour notifications are required for all SAEs followed by a complete report

- Within 5 calendar days for Grade 3-5 SAEs
- Within 10 calendar days for Grade 1-2 SAEs

<sup>2</sup>For studies using nuclear medicine or molecular imaging IND agents (NM, SPECT, or PET), the SAE reporting period is limited to 10 radioactive half-lives, rounded UP to the nearest whole day, after the agent/intervention was last administered. Footnote "1" above applies after this reporting period.

Effective Date: August 30, 2024

#### 10.4 Routine Adverse Event Reporting

All Adverse Events must be reported in routine study data submissions. AEs reported expeditiously through Medidata Rave must <u>also</u> be reported in routine study data submissions.

Adverse event data collection and reporting, which are required as part of every clinical trial, are done to ensure the safety of patients enrolled in the studies as well as those who will enroll in future studies using similar agents. AEs are reported in a routine manner at scheduled times during the trial using Medidata Rave. For this trial the Adverse Event CRF is used for routine AE reporting in Rave.

# 10.5 Pregnancy

Although not an adverse event in and of itself, pregnancy as well as its outcome must be documented via **Medidata Rave**. In addition, the *Pregnancy Information Form* included within the NCI Guidelines for Adverse Event Reporting Requirements must be completed and submitted to CTEP. Any pregnancy occurring in a patient or patient's partner from the time of consent to 90 days after the last dose of study drug must be reported and then followed for outcome. Newborn infants should be followed until 30 days old. Please see the "NCI Guidelines for Investigators: Adverse Event Reporting Requirements for DCTD (CTEP and CIP) and DCP INDs and IDEs" (at <a href="http://ctep.cancer.gov/protocolDevelopment/adverse\_effects.htm">http://ctep.cancer.gov/protocolDevelopment/adverse\_effects.htm</a>) for more details on how to report pregnancy and its outcome to CTEP.

# **10.6 Secondary Malignancy**

A secondary malignancy is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A secondary malignancy is not considered a metastasis of the initial neoplasm.

CTEP requires all secondary malignancies that occur following treatment with an agent under an NCI IND/IDE be reported expeditiously via Medidata Rave. Three options are available to describe the event:

- Leukemia secondary to oncology chemotherapy (e.g., acute myelocytic leukemia [AML])
- Myelodysplastic syndrome (MDS)
- Treatment-related secondary malignancy

Any malignancy possibly related to cancer treatment (including AML/MDS) should also be reported via the routine reporting mechanisms outlined in each protocol.

Indicate form for reporting in Rave, timeframes, and if loading of the pathology report is required.

# 10.7 Second Malignancy

A second malignancy is one unrelated to the treatment of a prior malignancy (and is **NOT** a metastasis from the initial malignancy). Second malignancies require **ONLY** routine AE reporting unless otherwise specified.

# 11. STUDY CALENDAR

Following registration, patients should begin protocol treatment within a minimum of 7 days and no more than 14 days. Baseline evaluations are to be conducted within 1 week prior to start of protocol therapy. Scans and x-rays must be done  $\leq 4$  weeks prior to the start of therapy. In the event that the patient's condition is deteriorating, laboratory evaluations should be repeated within 48 hours prior to initiation of the next cycle of therapy.

| | Pre-study<br>(≤30 days<br>prior to | Cycles 1 - 4: Cycle length = 3 weeks | | | | | | | | | Cycles 5+:<br>Cycle length = 4 weeks | At disease | 4 weeks after last dose of | Long term follow-up off | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | registration) | Week | Cycle 1<br>Week | Week | Week | Cycle 2<br>Week | | Week | Cycle 3<br>Week | Week | Week | Cycle 4<br>Week | Week | Cycle 5+ Day | progression | study drug <sup>D</sup> | study treatment <sup>E</sup> |
| | | 1 | 2 | 3 | 1 | 2 | 3 | 1 | 2 | 3 | 1 | 2 | 3 | 1 1 | | | |
| XL184 (cabozantinib) <sup>A</sup> | | Х— | | | | | | | | | | | | X | | | |
| Nivolumab <sup>B</sup> | | X | | | X | | | X | | | X | | | X | | | |
| Ipilimumab <sup>C</sup> | | X | | | X | | | X | | | X | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics, Medical history | X | | | | | | | | | | | | | | | | |
| Concurrent meds | X | X | | | | | | | | | | | | X | | | |
| Physical exam, Vital signs, Weight,<br>Performance status | X | X | | | X | | | X | | | X | | | X | X | X | |
| Height | X | | | | | | | | | | | | | | | | |
| CBC w/differential and platelets | X | X | | | X | | | X | | | X | | | X | X | X <sup>M</sup> | |
| Serum Chemistry <sup>F</sup> | X | X | | | X | | | X | | | X | | | X | X | $X^{M}$ | |
| PT/INR, PTT | X | | | | | | | | | | | | | | X | X <sup>M</sup> | |
| Urine protein to creatinine ratio | X | X | | | X | | | X | | | X | | | X | X | X <sup>M</sup> | |
| Amylase and lipase | X | X | | | X | | | X | | | X | | | X | X | $X^{M}$ | |
| Pregnancy test <sup>G</sup> | X | X | | | X | | | X | | | X | | | X | | | |
| TSH (with reflex T3/T4, if abnormal) | X | X | | | X | | | X | | | X | | | X | X | X <sup>M</sup> | |
| Adrenocorticotropic hormone (ACTH) <sup>H</sup> | | X | | | | | | X | | | | | | X | X | X <sup>M</sup> | |
| Serum cortisol (AM measurement preferred) <sup>H</sup> | | X | | | | | | X | | | | | | X | X | $X^{M}$ | |
| Troponin, 2D echocardiogram, and cardiac history <sup>I</sup> | X | | | | | | | | | | | | | | | | |
| EKG <sup>J</sup> | X | X | | | X | | | X | | | X | | | X | X | X <sup>M</sup> | |
| Adverse event evaluation | | X | | | | | | | | | | | | X | X | X | |
| Radiologic evaluation K | X | | | | | | | X | | | | | | $X^N$ | X | | |

| | Pre-study<br>(≤30 days | Cycles 1 - 4: Cycle length = 3 weeks | | | | | | | | | Cycles 5+:<br>Cycle length = 4 weeks | At disease | 4 weeks after | Long term | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | prior to<br>registration) | Cycle 1 | | | Cycle 2 | | | Cycle 3 | | | Cycle 4 | | | Cycle 5+ | progression | last dose of<br>study drug <sup>D</sup> | follow-up off study treatment <sup>E</sup> |
| | | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>1 | Week<br>2 | Week<br>3 | Day<br>1 | | study drug | study ireatment |
| Ki-67 index | X | | | | | | | | | | | | | | | | |
| Tumor Biopsy for correlative studies <sup>L</sup> | X | | | | | X | | | | | | | | | | | |
| Blood collection in cfDNA streck tubes <sup>L</sup> | X | | | | | | | | | | | | | | | | |
| Follow-up (via phone is allowed in case the patient cannot make the clinic visit) | | | | | | | | | | | | | | | | | X |

- A: XL184 (cabozantinib): 40 mg PO once daily until disease progression or death.
- B: Nivolumab: 3 mg/kg IV on Day 1 of Cycles 1-4 and 480 mg IV on Day 1 of Cycle 5 and subsequent cycles until disease progression or death. May be given ±3 days from a scheduled start of dosing.
- C: Ipilimumab: 1 mg/kg IV on Day 1 of Cycles 1-4 (total of four doses). May be given ±3 days from a scheduled start of dosing. When scheduled for the same day, ipilimumab should be given immediately following nivolumab administration.
- D: Patients will need to come in for an initial clinical follow up at 4 weeks after the last dose of the study drug.
- E: Off-study evaluation: Patients will be followed every 12 weeks after the 4-week clinical visit for 2 years after discontinuation of study treatment or until death, whichever occurs first. In addition, patients removed from study for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event. Follow-up may be by phone interview.
- F: To include albumin, alkaline phosphatase, ALT, AST, bicarbonate, BUN, calcium, chloride, creatinine, GGT, glucose, lactate dehydrogenase, magnesium, phosphorus, potassium, sodium, total bilirubin, and total protein.
- G: Serum pregnancy test (women of childbearing potential only) will be performed at least seven days before beginning study therapy. A negative serum or urine pregnancy test is also required at the beginning of each treatment cycle.
- H: ACTH and serum cortisol will be tested at C1D1 and C3D1 prior to ipilimumab and nivolumab administration, C5D1 prior to nivolumab administration, and every other cycle thereafter.
- I: Troponin assessment and cardiac history should be obtained at baseline and subsequently as clinically indicated. A 2D echocardiogram should be obtained at baseline for patients with a history of CHF and at the investigator's discretion, and may be repeated as clinically indicated.
- J: EKG will be performed at baseline, on Day 1 of Cycles 1 to 5, and then every 8 weeks (every other cycle).
- K: CT or MRI scans of chest, abdomen, and pelvis will be done at baseline and to assess the response per RECIST v1.1 criteria. CTs or MRIs with IV contrast are encouraged but will be done at the investigator's discretion. CT imaging of the neck could be added at the investigator's discretion. IV Contrast enhanced CT imaging of chest, abdomen, and pelvis should occur every 2 cycles for the first 6 months and every 3 cycles thereafter until disease progression.
- L: Mandatory
- M: Should be done if clinically indicated.
- N: Tumor measurements are to be repeated every 2 cycles for the first 6 months and every 3 cycles thereafter.

ALT=alanine aminotransferase, AST=aspartate aminotransferase, BUN=blood urea nitrogen, CBC=complete blood count, CT=computed tomography, EKG=electrocardiogram, GGT=γ-glutamyl transferase,

IV=intravenous, MRI=magnetic resonance imaging, PO=orally, TSH=thyroid stimulating hormone.

# 12. MEASUREMENT OF EFFECT

#### 12.1 Antitumor Effect – Solid Tumors

For the purposes of this study, patients should be re-evaluated for response every 2 cycles for the first 6 months on treatment and every 3 cycles thereafter. In addition to a baseline scan, confirmatory scans should also be obtained in case of suspected psuedoprogression at 6 weeks following initial documentation of objective response. If clear progression is observed *i.e.* new lesions *etc.*, no additional scan is needed for confirmation. CT scan of the chest, abdomen, and pelvis with contrast will be used for evaluation of disease at baseline, every 2 cycles for the first 6 months and every 3 cycles thereafter until disease progression. MRI of the brain may be used in addition, if prior brain involvement is known and should coincide with the CT scan schedule.

Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

#### 12.1.1 Definitions

<u>Evaluable for toxicity</u>. All patients will be evaluable for toxicity from the time of their first treatment with XL184 (cabozantinib), nivolumab, and ipilimumab.

<u>Evaluable for objective response.</u> All eligible patients who have measurable disease present at baseline, have received at least one dose of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated below. (Note: Patients who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.)

<u>Evaluable Non-Target Disease Response</u>. Patients who have lesions present at baseline that are evaluable but do not meet the definitions of measurable disease, have received at least one dose of therapy, and have had their disease re-evaluated will be considered evaluable for non-target disease. The response assessment is based on the presence, absence, or unequivocal progression of the lesions.

#### 12.1.2 Disease Parameters

<u>Measurable disease</u>. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as  $\geq$ 20 mm ( $\geq$ 2 cm) by chest x-ray or as  $\geq$ 10 mm ( $\geq$ 1 cm) with CT scan, MRI, or calipers by clinical exam. All tumor measurements must be recorded in <u>millimeters</u> (or decimal fractions of centimeters).

Note: Tumor lesions that are situated in a previously irradiated area might or might not be considered measurable. *If the investigator thinks it appropriate to include them, the conditions under which such lesions should be considered must be defined in the protocol.* 

Malignant lymph nodes. To be considered pathologically enlarged and measurable, a lymph node must be  $\ge 15$  mm ( $\ge 1.5$  cm) in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm [0.5 cm]). At baseline and in follow-up, only the short axis will be measured and followed.

Non-measurable disease. All other lesions (or sites of disease), including small lesions (longest diameter <10 mm [<1 cm] or pathological lymph nodes with ≥10 to <15 mm [≥1 to <1.5 cm] short axis), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT or MRI), are considered as non-measurable.

Note: Cystic lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.

'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions.

<u>Target lesions.</u> All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as **target lesions** and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement in which circumstance the next largest lesion which can be measured reproducibly should be selected. A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters. If lymph nodes are to be included in the sum, then only the short axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the disease.

<u>Non-target lesions</u>. All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as **non-target lesions** and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow-up.

# 12.1.3 Methods for Evaluation of Measurable Disease

All measurements should be taken and recorded in metric notation using a ruler or calipers. All baseline evaluations should be performed as closely as possible to the beginning of treatment and never more than 4 weeks before the beginning of the treatment.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is

preferred to evaluation by clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam.

Clinical lesions. Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes) and  $\geq 10$  mm ( $\geq 1$  cm) diameter as assessed using calipers (e.g., skin nodules). In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.

<u>Chest x-ray.</u> Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.

Conventional CT and MRI. This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm (0.5 cm) or less. If CT scans have slice thickness greater than 5 mm (0.5 cm), the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable in certain situations (*e.g.* for body scans).

Use of MRI remains a complex issue. MRI has excellent contrast, spatial, and temporal resolution; however, there are many image acquisition variables involved in MRI, which greatly impact image quality, lesion conspicuity, and measurement. Furthermore, the availability of MRI is variable globally. As with CT, if an MRI is performed, the technical specifications of the scanning sequences used should be optimized for the evaluation of the type and site of disease. Furthermore, as with CT, the modality used at follow-up should be the same as was used at baseline and the lesions should be measured/assessed on the same pulse sequence. It is beyond the scope of the RECIST guidelines to prescribe specific MRI pulse sequence parameters for all scanners, body parts, and diseases. Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior scans. Body scans should be performed with breath-hold scanning techniques, if possible.

<u>PET-CT</u>. At present, the low dose or attenuation correction CT portion of a combined PET-CT is not always of optimal diagnostic CT quality for use with RECIST measurements. Hence it should not be used for tumor response assessment in the evaluation of patients enrolled in the study.

<u>Ultrasound</u>. Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement. Ultrasound examinations cannot be reproduced in their entirety for independent review at a later date and, because they are operator dependent, it cannot be guaranteed that the same technique and measurements will be taken from one assessment to the next. If new lesions are identified by ultrasound in the course of the study, confirmation by CT or MRI is advised. If there is concern about radiation exposure at CT, MRI may be used instead of CT in selected instances.

<u>Endoscopy</u>, <u>Laparoscopy</u>. The utilization of these techniques for objective tumor evaluation is not advised. However, such techniques may be useful to confirm complete pathological response when biopsies are obtained or to determine relapse in trials where recurrence following complete response (CR) or surgical resection is an endpoint.

<u>Tumor markers.</u> Tumor markers alone cannot be used to assess response. If markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response. Specific guidelines for both CA-125 response (in recurrent ovarian cancer) and PSA response (in recurrent prostate cancer) have been published [*JNCI* 96:487-488, 2004; *J Clin Oncol* 17, 3461-3467, 1999; *J Clin Oncol* 26:1148-1159, 2008]. In addition, the Gynecologic Cancer Intergroup has developed CA-125 progression criteria which are to be integrated with objective tumor assessment for use in first-line trials in ovarian cancer [*JNCI* 92:1534-1535, 2000].

<u>Cytology</u>, <u>Histology</u>. These techniques can be used to differentiate between partial responses (PR) and complete responses (CR) in rare cases (*e.g.*, residual lesions in tumor types, such as germ cell tumors, where known residual benign tumors can remain).

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease (an effusion may be a side effect of the treatment) and progressive disease.

<u>FDG-PET</u>. While FDG-PET response assessments need additional study, it is sometimes reasonable to incorporate the use of FDG-PET scanning to complement CT scanning in assessment of progression (particularly possible 'new' disease). New lesions on the basis of FDG-PET imaging can be identified according to the following algorithm:

- a. Negative FDG-PET at baseline, with a positive FDG-PET at follow-up is a sign of PD based on a new lesion.
- b. No FDG-PET at baseline and a positive FDG-PET at follow-up: If the positive FDG-PET at follow-up corresponds to a new site of disease confirmed by CT, this is PD. If the positive FDG-PET at follow-up is not confirmed as a new site of disease on CT, additional follow-up CT scans are needed to determine if there is truly progression occurring at that site (if so, the date of PD will be the date of the initial abnormal FDG-PET scan). If the positive FDG-PET at follow-up corresponds to a pre-existing site of disease on CT that is not progressing on the basis of the anatomic images, this is not PD.
- c. FDG-PET may be used to upgrade a response to a CR in a manner similar to a biopsy in cases where a residual radiographic abnormality is thought to represent fibrosis or scarring. The use of FDG-PET in this circumstance should be prospectively described in the protocol and supported by disease-specific medical literature for the indication. However, it must be acknowledged that both approaches may lead to false positive CR due to limitations of FDG-PET and biopsy resolution/sensitivity.

Note: A 'positive' FDG-PET scan lesion means one which is FDG avid with an uptake greater than twice that of the surrounding tissue on the attenuation corrected image.

# 12.1.4 Response Criteria

# 12.1.4.1 Evaluation of Target Lesions

<u>Complete Response (CR)</u>: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm).

<u>Partial Response (PR)</u>: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

<u>Progressive Disease (PD)</u>: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). (Note: the appearance of one or more new lesions is also considered progressions).

<u>Stable Disease (SD)</u>: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

# 12.1.4.2 Evaluation of Non-Target Lesions

<u>Complete Response (CR)</u>: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm [<1 cm] short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.

<u>Non-CR/Non-PD:</u> Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.

<u>Progressive Disease (PD)</u>: Appearance of one or more new lesions and/or <u>unequivocal</u> <u>progression</u> of existing non-target lesions. <u>Unequivocal progression</u> should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator).

#### 12.1.4.3 Evaluation of Best Overall Response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

#### For Patients with Measurable Disease (i.e., Target Disease)

| Target<br>Lesions | Non-Target<br>Lesions | New<br>Lesions | Overall<br>Response | Best Overall Response when Confirmation is Required* |
|---|---|---|---|---|
| CR | CR | No | CR | ≥4 wks. Confirmation** |
| CR | Non-CR/Non-<br>PD | No | PR | |
| CR | Not evaluated | No | PR | 1 vylsa Canfirmation** |
| PR | Non-CR/Non- | No | PR | ≥4 wks. Confirmation** |
| | PD/not<br>evaluated | | | |
| SD | Non-CR/Non-<br>PD/not<br>evaluated | No | SD | Documented at least once ≥4 wks. from baseline** |
| PD | Any | Yes or No | PD | |
| Any | PD*** | Yes or No | PD | no prior SD, PR or CR |
| Any | Any | Yes | PD | |

<sup>\*</sup> See RECIST 1.1 manuscript for further details on what is evidence of a new lesion.

Note: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

# For Patients with Non-Measurable Disease (i.e., Non-Target Disease)

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

<sup>\* &#</sup>x27;Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised

# 12.1.5 Duration of Response

<u>Duration of overall response</u>: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

<sup>\*\*</sup> Only for non-randomized trials with response as primary endpoint.

<sup>\*\*\*</sup> In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression.

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.

<u>Duration of stable disease</u>: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.

# **12.1.6** Progression-Free Survival

PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

# 12.1.7 Response Review

**TBD** 

# 12.2 Other Response Parameters

N/A

# 13. STUDY OVERSIGHT AND DATA REPORTING / REGULATORY REQUIREMENTS

Adverse event lists, guidelines, and instructions for AE reporting can be found in Section 10 (Adverse Events: List and Reporting Requirements).

# 13.1 Study Oversight

This protocol is monitored at several levels, as described in this section. The Protocol Principal Investigator is responsible for monitoring the conduct and progress of the clinical trial, including the ongoing review of accrual, patient-specific clinical and laboratory data, and routine and serious adverse events; reporting of expedited adverse events; and accumulation of reported adverse events from other trials testing the same drug(s). The Protocol Principal Investigator and statistician have access to the data at all times through the CTMS web-based reporting portal.

The Protocol Principal Investigator will have, at a minimum, quarterly conference calls with the Study Investigators and the CTEP Medical Officer(s) to review accrual, progress, and pharmacovigilance. Decisions to proceed to the second stage of a Phase 2 trial will require sign-off by the Protocol Principal Investigator and the Protocol Statistician.

All Study Investigators at participating sites who register/enroll patients on a given protocol are responsible for timely submission of data via Medidata Rave and timely reporting of adverse events for that particular study. This includes timely review of data collected on the electronic CRFs submitted via Medidata Rave.

All studies are also reviewed in accordance with the enrolling institution's data safety monitoring plan.

#### 13.2 Data Reporting

Medidata Rave is the clinical data management system being used for data collection for this trial/study. Access to the trial in Rave is controlled through the CTEP-IAM system and role assignments.

Requirements to access Rave via iMedidata:

- Active CTEP registration with the credentials necessary to access secure NCI/CTSU IT systems; and
- Assigned a Rave role on the LPO or PO roster at the enrolling site of: Rave CRA, Rave Read Only, Rave CRA (LabAdmin), Rave SLA, or Rave Investigator.
  - o Rave role requirements:
    - Rave CRA or Rave CRA (Lab Admin) role must have a minimum of an Associate Plus (AP) registration type,
    - Rave Investigator role must be registered as a Non-Physician Investigator (NPIVR) or Investigator (IVR), and

- Rave Read Only or Rave SLA role must have at a minimum an Associate
   (A) registration type.
- o Refer to <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a> for registration types and documentation required.
- DTL Rave CRA task assignment requirements (for write access):
  - o Corresponding role (Rave CRA or Rave CRA (Lab Admin)) on the site roster; and
  - Completion of the Theradex Specimen Tracking System (STS) Training course in CLASS (see Section 4.2.3 – Delegation of Tasks Log (DTL)).

# 13.2.1 Protocol Specific Requirements For Rave Access

- Specimen Tracking System Training Requirement for full read/write Rave access:
  - All site staff assigned the Rave CRA task on the DTL must complete the online specimen tracking training, which is administered via the Compliance, Learning, and SOP Solutions (CLASS) system.
  - O Completion of the training will be automatically communicated to the CTSU Regulatory application and to Medidata Rave, and the individual will receive an invitation to [protocol #] in Rave. There is no need to submit a training completion certificate to the CTSU through the Regulatory Submission Portal.
  - O The training is a one-time only requirement per individual. If an individual has previously completed the training for another ETCTN study (either within CLASS, or via the procedure in place prior to CLASS), the training does not need to be completed again. However, new versions of the Specimen Tracking System training course may require new training.
  - o For questions about the training content or the tracking system itself, please contact STS Support at Theradex (STS.Support@theradex.com).
  - o For questions or concerns about accessing the training in CLASS, please contact the CLASS Help Desk <u>CLASSHelpDesk@westat.com</u>.

Upon initial site registration approval for the study in the Regulatory application, all persons with Rave roles assigned on the appropriate roster will be sent a study invitation email from iMedidata. No action will be required; each study invitation will be automatically accepted and study access in Rave will be automatically granted. Site staff will not be able to access the study in Rave until all required Medidata and study specific trainings are completed. Trainings will be in the form of electronic learnings (eLearnings) and can be accessed by clicking on the eLearning link in the *Tasks* pane located in the upper right corner of the iMedidata screen. If an eLearning is required for a study and has not yet been taken, the link to the eLearning will appear under the study name in the *Studies* pane located in the center of the iMedidata screen; once the successful completion of the eLearning has been recorded, access to the study in Rave will be granted, and a *Rave EDC* link will replace the eLearning link under the study name.

Action will be required by site staff (to activate their account) who have not previously activated their iMedidata/Rave account at the time of initial site registration approval for the study in the Regulatory application. Account activation instructions are located on the CTSU website in the Data Management section under the Data Management Help Topics > Rave Resources >
Medidata Account Activation and Study Invitation (to activate your iMedidata account). Additional information on iMedidata/Rave is available on the CTSU members' website in the Data Management Rave Resources section or by contacting the CTSU Help Desk at 1-888-823-5923 or by email at <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>.

### 13.2.2 Method

This study will be monitored by the Clinical Trials Monitoring Service (CTMS). Data will be submitted to CTMS at least once every two weeks via Medidata Rave (or other modality if approved by CTEP). Information on CTMS reporting is available at <a href="http://www.theradex.com/clinicalTechnologies/?National-Cancer-Institute-NCI-11">http://www.theradex.com/clinicalTechnologies/?National-Cancer-Institute-NCI-11</a>. On-site audits will be conducted three times annually (one annual site visit and two data audits). For CTMS monitored studies, after users have activated their accounts, please contact the Theradex Help Desk at (609) 619-7862 or by email at <a href="https://ctms.com/ct

### 13.2.3 Responsibility for Data Submission

For ETCTN trials, it is the responsibility of the PI(s) at the site to ensure that all investigators at the ETCTN Sites understand the procedures for data submission for each ETCTN protocol and that protocol specified data are submitted accurately and in a timely manner to the CTMS via the electronic data capture system, Medidata Rave.

Data are to be submitted via Medidata Rave to CTMS on a real-time basis, but no less than once every 2 weeks. The timeliness of data submissions and timeliness in resolving data queries will be tracked by CTMS. Metrics for timeliness will be followed and assessed on a quarterly basis. For the purpose of Institutional Performance Monitoring, data will be considered delinquent if it is greater than 4 weeks past due.

Data from Medidata Rave and CTEP-AERS is reviewed by the CTMS on an ongoing basis as data is received. Queries will be issued by CTMS directly within Rave. The queries will appear on the Task Summary Tab within Rave for the CRA at the ETCTN to resolve. Monthly web-based reports are posted for review by the Drug Monitors in the IDB, CTEP. Onsite audits will be conducted by the CTMS to ensure compliance with regulatory requirements, GCP, and NCI policies and procedures with the overarching goal of ensuring the integrity of data generated from NCI-sponsored clinical trials, as described in the ETCTN Program Guidelines, which may be found on the CTEP

(<u>http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/adverse\_events.htm</u>) and CTSU websites.

An End of Study CRF is to be completed by the PI, and is to include a summary of study endpoints not otherwise captured in the database, such as (for phase 1 trials) the recommended phase 2 dose (RP2D) and a description of any dose-limiting toxicities (DLTs). CTMS will utilize a core set of eCRFs that are Cancer Data Standards Registry and Repository (caDSR) compliant (<a href="http://cbiit.nci.nih.gov/ncip/biomedical-informatics-resources/interoperability-and-semantics/metadata-and-models">http://cbiit.nci.nih.gov/ncip/biomedical-informatics-resources/interoperability-and-semantics/metadata-and-models</a>). Customized eCRFs will be included when appropriate to meet

unique study requirements. The PI is encouraged to review the eCRFs, working closely with CTMS to ensure prospectively that all required items are appropriately captured in the eCRFs prior to study activation. CTMS will prepare the eCRFs with built-in edit checks to the extent possible to promote data integrity.

CDUS data submissions for ETCTN trials activated after March 1, 2014, will be carried out by the CTMS contractor, Theradex. CDUS submissions are performed by Theradex on a monthly basis. The trial's lead institution is responsible for timely submission to CTMS via Rave, as above.

Further information on data submission procedures can be found in the ETCTN Program Guidelines

(http://ctep.cancer.gov/protocolDevelopment/electronic applications/adverse events.htm).

### 13.3 Data Quality Portal

The Data Quality Portal (DQP) provides a central location for site staff to manage unanswered queries and form delinquencies, monitor data quality and timeliness, generate reports, and review metrics.

The DQP is located on the CTSU members' website under Data Management. The Rave Home section displays a table providing summary counts of Total Delinquencies and Total Queries. DQP Queries, DQP Delinquent Forms, DQP Form Status and the DQP Reports modules are available to access details and reports of unanswered queries, delinquent forms, forms with current status, and timeliness reports. Site staff should review the DQP modules on a regular basis to manage specified queries and delinquent forms.

The DQP is accessible by site staff who are rostered to a site and have access to the CTSU website. Staff who have Rave study access can access the Rave study data via direct links available on the DQP modules.

CTSU Delinquency Notification emails are sent to primary contacts at sites twice a month. These notifications serve as alerts that queries and/or delinquent forms require site review, providing a summary count of queries and delinquent forms for each Rave study that a site is participating in. Additional site staff can subscribe and unsubscribe to these notifications using the CTSU Report and Information Subscription Portal on the CTSU members' website.

To learn more about DQP use and access, click on the Help Topics button displayed on the Rave Home, DQP Queries, DQP Delinquent Forms, DQP Form Status, and DQP Reports modules.

13.4 CTEP Multicenter Guidelines

N/A

### 13.5 Collaborative Agreements Language

The agent(s) supplied by CTEP, DCTD, NCI used in this protocol is/are provided to the NCI under a Collaborative Agreement (CRADA, CTA, CSA) between the Pharmaceutical Company(ies) (hereinafter referred to as "Collaborator(s)") and the NCI Division of Cancer Treatment and Diagnosis. Therefore, the following obligations/guidelines, in addition to the provisions in the "Intellectual Property Option to Collaborator" (<a href="http://ctep.cancer.gov/industryCollaborations2/intellectual property.htm">http://ctep.cancer.gov/industryCollaborations2/intellectual property.htm</a>) contained within the terms of award, apply to the use of the Agent(s) in this study:

- 1. Agent(s) may not be used for any purpose outside the scope of this protocol, nor can Agent(s) be transferred or licensed to any party not participating in the clinical study. Collaborator(s) data for Agent(s) are confidential and proprietary to Collaborator(s) and shall be maintained as such by the investigators. The protocol documents for studies utilizing Agents contain confidential information and should not be shared or distributed without the permission of the NCI. If a copy of this protocol is requested by a patient or patient's family member participating on the study, the individual should sign a confidentiality agreement. A suitable model agreement can be downloaded from: http://ctep.cancer.gov.
- 2. For a clinical protocol where there is an investigational Agent used in combination with (an)other Agent(s), each the subject of different Collaborative Agreements, the access to and use of data by each Collaborator shall be as follows (data pertaining to such combination use shall hereinafter be referred to as "Multi-Party Data"):
  - a. NCI will provide all Collaborators with prior written notice regarding the existence and nature of any agreements governing their collaboration with NCI, the design of the proposed combination protocol, and the existence of any obligations that would tend to restrict NCI's participation in the proposed combination protocol.
  - b. Each Collaborator shall agree to permit use of the Multi-Party Data from the clinical trial by any other Collaborator solely to the extent necessary to allow said other Collaborator to develop, obtain regulatory approval or commercialize its own Agent.
  - c. Any Collaborator having the right to use the Multi-Party Data from these trials must agree in writing prior to the commencement of the trials that it will use the Multi-Party Data solely for development, regulatory approval, and commercialization of its own Agent.
- 3. Clinical Trial Data and Results and Raw Data developed under a Collaborative Agreement will be made available to Collaborator(s), the NCI, and the FDA, as appropriate and unless additional disclosure is required by law or court order as described in the IP Option to Collaborator (<a href="http://ctep.cancer.gov/industryCollaborations2/intellectual\_property.htm">http://ctep.cancer.gov/industryCollaborations2/intellectual\_property.htm</a>). Additionally, all Clinical Data and Results and Raw Data will be collected, used and disclosed consistent with all applicable federal statutes and regulations for the protection of human subjects, including, if applicable, the *Standards for Privacy of Individually Identifiable Health Information* set forth in 45 C.F.R. Part 164.

4. When a Collaborator wishes to initiate a data request, the request should first be sent to the NCI, who will then notify the appropriate investigators (Group Chair for Cooperative Group studies, or PI for other studies) of Collaborator's wish to contact them.

- 5. Any data provided to Collaborator(s) for Phase 3 studies must be in accordance with the guidelines and policies of the responsible Data Monitoring Committee (DMC), if there is a DMC for this clinical trial.
- 6. Any manuscripts reporting the results of this clinical trial must be provided to CTEP by the Group office for Cooperative Group studies or by the principal investigator for non-Cooperative Group studies for immediate delivery to Collaborator(s) for advisory review and comment prior to submission for publication. Collaborator(s) will have 30 days from the date of receipt for review. Collaborator shall have the right to request that publication be delayed for up to an additional 30 days in order to ensure that Collaborator's confidential and proprietary data, in addition to Collaborator(s)'s intellectual property rights, are protected. Copies of abstracts must be provided to CTEP for forwarding to Collaborator(s) for courtesy review as soon as possible and preferably at least three (3) days prior to submission, but in any case, prior to presentation at the meeting or publication in the proceedings. Press releases and other media presentations must also be forwarded to CTEP prior to release. Copies of any manuscript, abstract and/or press release/ media presentation should be sent to:

Email: ncicteppubs@mail.nih.gov

The Regulatory Affairs Branch will then distribute them to Collaborator(s). No publication, manuscript or other form of public disclosure shall contain any of Collaborator's confidential/proprietary information.

#### 14. REFERENCES

AACR Press release. (2019). Immune checkpoint inhibitor combination efficacious for patients with high-grade neuroendocrine carcinoma. 31 March 2019.

Andreyev, H.J., P. Scott-Mackie, D. Cunningham, *et al.* (1995). Phase II study of continuous infusion fluorouracil and interferon alfa-2b in the palliation of malignant neuroendocrine tumors. *J Clin Oncol.* 13:1486-1492.

Ansell, S.M., S.A. Hurvitz, P.A. Koenig, *et al.* (2009). Phase I study of ipilimumab, an anti-CTLA-4 monoclonal antibody, in patients with relapsed and refractory B-cell non-Hodgkin lymphoma. *Clin Cancer Res.* 15:6446-53.

Antonia, S.J., J.A. Lopez-Martin, J. Bendell, et al. (2016). Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. *Lancet Oncol.* 17:883-895.

Apolo, A.B., A. Mortazavi, M. Stein, *et al.* (2016). A phase I study of cabozantinib plus nivolumab (CaboNivo) in patients (pts) refractory metastatic urothelial carcinoma (mUC) and other genitourinary (GU) tumors. *Ann Oncol.* 27:266-295.

Apolo, A.B., A. Mortazavi, M.N. Stein, *et al.* (2017). A phase I study of cabozantinib plus nivolumab (CaboNivo) and ipilimumab (CaboNivoIpi) in patients (pts) with refractory metastatic urothelial carcinoma (mUC) and other genitourinary (GU) tumors. *J Clin Oncol.* 35:293.

Apolo, A.B., Y. Tomita, M.J. Lee, *et al.* (2014). Effect of cabozantinib on immunosuppressive subsets in metastatic urothelial carcinoma. *J Clin Oncol.* 32:4501.

Basu, B., B. Sirohi, and P. Corrie. (2010). Systemic therapy for neuroendocrine tumours of gastroenteropancreatic origin. *Endocr Relat Cancer*. 17:R75-90.

Bentzien, F., Zuzow, M., Heald, N., *et al.* (2013). In vitro and in vivo activity of XL184 (cabozantinib) (XL184), an inhibitor of RET, MET, and VEGFR2, in a model of medullary thyroid cancer. *Thyroid*. 23:1569-1577.

Birchmeier, C., Birchmeier, W., Gherardi, E., and Vande Woude, G.F. (2003). Met, metastasis, motility and more. *Nat Rev Mol Cell Biol.* 4:915-925.

Boccaccio, C., and Comoglio, P.M. (2006). Invasive growth: a MET-driven genetic programme for cancer and stem cells. *Nat Rev Cancer*. 6:637-645.

Bosman, F.T., World Health Organization., International Agency for Research on Cancer. (2010). WHO classification of tumours of the digestive system. *Lyon: International Agency for Research on Cancer*. 4th ed. 417.

NCI Protocol #: 10315

Version Date: June 3, 2025

Chan, J.A., J.E. Faris, J.E. Murphy, et al. (2017). Phase II trial of cabozantinib in patients with carcinoid and pancreatic neuroendocrine tumors (pNET). J Clin Oncol. 4 suppl:228

Chauhan, A., Q. Yu, N. Ray, et al. (2018). Global burden of neuroendocrine tumors and changing incidence in Kentucky. *Oncotarget*. 9:19245-54.

Chen, Q., T. Li, and W. Yue. (2018). Drug response to PD-1/PD-L1 blockade: based on biomarkers. *Onco Targets Ther*. 11:4673-4683.

Christensen, J.G., Burrows, J., and Salgia, R. (2005). MET as a target for human cancer and characterization of inhibitors for therapeutic intervention. *Cancer Lett.* 225:1-26.

Comoglio, P.M., Giordano, S., and Trusolino, L. (2008). Drug development of MET inhibitors: targeting oncogene addiction and expedience. *Nat Rev Drug Discov.* 7:504-516.

Coudriet, G.M., J. He, M. Trucco, *et al.* (2010). Hepatocyte growth factor modulates interleukin-6 production in bone marrow derived macrophages: implications for inflammatory mediated diseases. *PLoS One.* 5:e15384.

Curran, M.A., Montalvo, W., Yagita, H., *et al.* (2010). PD-1 and CTLA-4 combination blockade expands infiltrating T cells and reduces regulatory T and myeloid cells within B16 melanoma tumors. *Proc Natl Acad Sci USA*. 107:4275-4280.

Dasari, A., C. Shen, D. Halperin, *et al.* (2017). Trends in the incidence, prevalence, and survival outcomes in patients with neuroendocrine tumors in the United States. *JAMA oncology*. 3:1335-1342.

Dong, H., and Chen, L. (2003). B7-H1 pathway and its role in the evasion of tumor immunity. *J Mol Med (Berl)*. 81:281-287.

Eisenhauer, E.A., P. Therasse, J. Bogaerts, *et al.* (2009). New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). *Eur J Cancer*. 45:228-247.

Eriksson, B., B. Skogseid, G. Lundqvist, Wide L, *et al.* (1990). Medical treatment and long-term survival in a prospective study of 84 patients with endocrine pancreatic tumors. *Cancer*. 65:1883-1890.

Ferris, R.L., Blumenschein, Jr., G., Fayette, J., et al. (2016). Nivolumab for recurrent squamous-cell carcinoma of the head and neck. N Engl J Med. 375:1856-1867.

Green, R.C., J.S. Berg, W.W. Grody, *et al.* (American College of Medical Genetics and Genomics). (2013). ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. *Genet Med.* 15:565-574.

Hadoux, J., D. Malka, D. Planchard, et al. (2015). Post-first-line FOLFOX chemotherapy for grade 3 neuroendocrine carcinoma. Endocr Relat Cancer. 22:289-298.

Hentic, O., P. Hammel, A. Couvelard, *et al.* (2012). FOLFIRI regimen: an effective second-line chemotherapy after failure of etoposide-platinum combination in patients with neuroendocrine carcinomas grade 3. *Endocr Relat Cancer*. 19:751-757.

Imai, H., H. Shirota, A. Okita, *et al.* (2016). Efficacy and safety of carboplatin and etoposide combination chemotherapy for extrapulmonary neuroendocrine carcinoma: A retrospective case series. *Chemotherapy*. 61:111-116.

Investigator's Brochure. (2018). Cabozantinib (XL184). Version 14, 14 June 2018. Exelixis, Inc. Alameda, CA.

Investigator's Brochure. (2018). Ipilimumab, BMS-734016, MDX010. Version 21, 14 March 2018. Bristol-Myers Squibb. Wallingford, CT.

Investigator's Brochure. (2018). Nivolumab, BMS-936558, MDX1106. Version 17, 27 June 2018. Bristol-Myers Squibb. Lawrenceville, NJ.

Iwasa, S., C. Morizane, T. Okusaka, et al. (2010). Cisplatin and etoposide as first-line chemotherapy for poorly differentiated neuroendocrine carcinoma of the hepatobiliary tract and pancreas. *J Clin Oncol.* 40:313-318.

Jeffers, M., Schmidt, L., Nakaigawa, N., et al. (1997). Activating mutations for the met tyrosine kinase receptor in human cancer. *Proc Natl Acad Sci U S A*. 94:11445-11450.

Kalia, S.S., K. Adelman, S.J. Bale, *et al.* (2016). Recommendations for reporting of secondary findings in clinical exome and genome sequencing, 2016 update (ACMG SF v2.0): a policy statement of the American College of Medical Genetics and Genomics. *Genet Med.* 19:249-255.

Kang, H., J.B. O'Connell, M.J. Leonardi, *et al.* (2007). Rare tumors of the colon and rectum: a national review. *Int J Colorectal Dis.* 22:183-189.

Kaufman, H.L., J. Russell, O. Hamid, *et al.* (2016). Avelumab in patients with chemotherapy-refractory metastatic Merkel cell carcinoma: a multicentre, single-group, open-label, phase 2 trial. *Lancet Oncol.* 17:1374-1385.

Kim, J.Y., S.M. Hong and J.Y. Ro. (2017). Recent updates on grading and classification of neuroendocrine tumors. *Ann Diagn Pathol.* 29:11-16.

Kolby, L., G. Persson, S. Franzen, and B. Ahren. (2003). Randomized clinical trial of the effect of interferon alpha on survival in patients with disseminated midgut carcinoid tumours. *Br J Surg.* 90:687-693.

Kwilas, A.R., A. Ardiani, R.N. Donahue, *et al.* (2014). Dual effects of a targeted small-molecule inhibitor (cabozantinib) on immune-mediated killing of tumor cells and immune tumor

microenvironment permissiveness when combined with a cancer vaccine. *J Translat Med*. 12:294.

Liu, X., Newton, R.C., and Scherle, P.A. (2010). Developing c-MET pathway inhibitors for cancer therapy: progress and challenges. *Trends Mol Med.* 16:37-45.

Lu, X., J.W. Horner, E. Paul, *et al.* (2017). Effective combinatorial immunotherapy for castration-resistant prostate cancer. *Nature*. 543:728-732.

Maggard, M.A., J.B. O'Connell and C.Y. Ko. (2004). Updated population-based review of carcinoid tumors. *Ann Surg.* 240:117-122.

Mitry, E., E. Baudin, M. Ducreux, et al. (1999). Treatment of poorly differentiated neuroendocrine tumours with etoposide and cisplatin. Br J Cancer. 81:1351-1355.

Moertel, C.G., J. Rubin and L.K. Kvols. (1989). Therapy of metastatic carcinoid tumor and the malignant carcinoid syndrome with recombinant leukocyte A interferon. *J Clin Oncol.* 7:865-868.

Moertel, C.G., L.K. Kvols, M.J. O'Connell, and J. Rubin. (1991). Treatment of neuroendocrine carcinomas with combined etoposide and cisplatin. Evidence of major therapeutic activity in the anaplastic variants of these neoplasms. *Cancer*. 68:227-232.

Nghiem, P.T., S. Bhatia, E.J. Lipson, *et al.* (2016). PD-1 Blockade with pembrolizumab in advanced Merkel-cell carcinoma. *N Engl J Med.* 374:2542-2552

Nivolumab [package insert]. New York, NY: BMS; 2014. [Available from: <a href="https://www.accessdata.fda.gov/drugsatfda">https://www.accessdata.fda.gov/drugsatfda</a> docs/label/2017/125554s055lbl.pdf.]

Nomi, T., Sho, M., Akahori, T., *et al.* (2007). Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. *Clin Cancer Res.* 13:2151-2157.

Oberg, K., and B. Eriksson. (1991). The role of interferons in the management of carcinoid tumours. *Br J Haematol*. 79 Suppl 1:74-77.

Oberg, K., I. Norheim I, E. Lind, *et al.* (1986). Treatment of malignant carcinoid tumors with human leukocyte interferon: long-term results. *Cancer Treat Rep.* 70:1297-1304.

Oberg, K., K. Funa and G. Alm. (1983). Effects of leukocyte interferon on clinical symptoms and hormone levels in patients with mid-gut carcinoid tumors and carcinoid syndrome. *N Engl J Med.* 309:129-133.

Ohigashi, Y., Sho, M., Yamada, Y., *et al.* (2005). Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. *Clin Cancer Res.* 11:2947-2953.

Okunishi, K., M. Dohi, K. Nakagome, *et al.* (2005). A novel role of hepatocyte growth factor as an immune regulator through suppressing dendritic cell function. *J Immunol.* 175:4745-4753.

Olsen, I.H., U. Knigge, B. Federspiel, *et al.* (2014). Topotecan monotherapy in heavily pretreated patients with progressive advanced stage neuroendocrine carcinomas. *J Cancer*. 5:628-632.

Ott, P.A., E. Elez, S. Hiret, *et al.* (2017). Pembrolizumab in patients with extensive-stage small-cell lung cancer: results from the phase Ib KEYNOTE-028 Study. *J Clin Oncol.* 35:3823-3829.

Overman, M.J., McDermott, R., Leach, J.L., *et al.* (2017). Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. *Lancet Oncol.* 18:1182-1191.

Pàez-Ribes, M., Allen, E., Hudock, J., *et al.* (2009). Antiangiogenic therapy elicits malignant progression of tumors to increased local invasion and distant metastasis. *Cancer Cells*. 15(3):220-231.

PASS 2019: Power and Analysis Sample Size Software. NCSS, LLC. Kaysville, Utah, USA. 2019 [Available from: <a href="https://www.ncss.com/software/pass">www.ncss.com/software/pass</a>].

Patta, A., and M. Fakih. (2011). First-line cisplatin plus etoposide in high-grade metastatic neuroendocrine tumors of colon and rectum (MCRC NET): review of 8 cases. *Anticancer Res*. 31:975-978.

Rindi, G, D.S. Klimstra, B. Abedi-Ardekani, *et al.* (2018). A common classification framework for neuroendocrine neoplasms: an International Agency for Research on Cancer (IARC) and World Health Organization (WHO) expert consensus proposal. *Mod Pathol.* 31:1770-1786.

Roberts, J.A., R.S. Gonzalez, S. Das, et al. (2017). Expression of PD-1 and PD-L1 in poorly differentiated neuroendocrine carcinomas of the digestive system: a potential target for anti-PD-1/PD-L1 therapy. *Hum Pathol.* 70:49-54.

Roskoski, Jr., R. (2008). VEGF receptor protein-tyrosine kinases: structure and regulation. *Biochem Biophys Res Commun.* 375:287-291.

Schmidt, L., Duh, F.M., Chen, F., *et al.* (1997). Germline and somatic mutations in the tyrosine kinase domain of the MET proto-oncogene in papillary renal carcinomas. *Nat Genet.* 16:68-73.

Schultheis, A.M., A.H. Scheel, L. Ozretic, *et al.* (2015). PD-L1 expression in small cell neuroendocrine carcinomas. *Eur J Cancer*. 51:421-426.

Sharma, P., and J.P. Allison. (2015). The future of immune checkpoint therapy. *Science*. 348:56-61.

Sorbye, H., S. Welin, S.W. Langer, *et al.* (2013). Predictive and prognostic factors for treatment and survival in 305 patients with advanced gastrointestinal neuroendocrine carcinoma (WHO G3): the NORDIC NEC study. *Ann Oncol.* 24:152-160.

Spranger, S., and T. Gajewski. (2013). Rational combinations of immunotherapeutics that target discrete pathways. *J ImmunoTher Cancer*. 1:1-14.

Taal, B.G. and O. Visser (2004). Epidemiology of neuroendocrine tumours. *Neuroendocrinology.* 80 Suppl 1:3-7.

Taube, J.M., Anders, R.A., Young, G.D., *et al.* (2012). Colocalization of inflammatory response with B7-H1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. *Sci Transl Med.* 4:127ra137.

Thompson, R.H., Gillett, M.D., Cheville, J.C., *et al.* (2004). Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. *Proc Natl Acad Sci USA*. 101:17174-17179.

Thompson, R.H., Gillett, M.D., Cheville, J.C., *et al.* (2005). Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. *Cancer.* 104:2084-2091.

Thompson, R.H., Kuntz, S.M., Leibovich, B.C., *et al.* (2006). Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. *Cancer Res.* 66:3381-3385.

Topalian, S.L., Hodi, F.S., Brahmer, J.R., et al. (2012). Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 366:2443-2454.

Tugues, S., Koch, S., Gualandi, L., et al. (2011). Vascular endothelial growth factors and receptors: anti-angiogenic therapy in the treatment of cancer. Mol Aspects Med. 32:88-111.

Weber, J.S., D'Angelo, S.P., Minor, D., *et al.* (2015). Nivolumab versus chemotherapy in patients with advanced melanoma who progressed after anti-CTLA-4 treatment (CheckMate 037): a randomised, controlled, open-label, phase 3 trial. *Lancet Oncol.* 16:375-384.

Wolchok, J.D., Kluger, H., Callahan, M.K., *et al.* (2013). Nivolumab plus ipilimumab in advanced melanoma. *N Engl J Med.* 369:122-133.

Woo, S.R., Turnis, M.E., Goldberg, M.V., *et al.* (2012). Immune inhibitory molecules LAG-3 and PD-1 synergistically regulate T-cell function to promote tumoral immune escape. *Cancer Res.* 72:917-927.

Wu, C., Zhu, Y., Jiang, J., *et al.* (2006). Immunohistochemical localization of programmed death-1 ligand-1 (PD-L1) in gastric carcinoma and its clinical significance. *Acta Histochem*. 108:19-24.

Yakes, F.M., Chen, J., Tan, J., *et al.* (2011). XL184 (cabozantinib) (XL184), a novel MET and VEGFR2 inhibitor, simultaneously suppresses metastasis, angiogenesis, and tumor growth. *Mol Cancer Ther.* 10:2298-2308.

Yao, J.C., M. Hassan, A. Phan, *et al.* (2008). One hundred years after "Carcinoid": Epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. *J Clin Oncol.* 26:3063-3072.

Yi, M., D. Jiao, H. Xu, et al. (2018). Biomarkers for predicting efficacy of PD-1/PD-L1 inhibitors. *Mol Cancer*. 17:129.

Zitvogel, L., Tesniere, A., and Kroemer, G. (2006). Cancer despite immunosurveillance: immunoselection and immunosubversion. *Nat Rev Immunol*. 6:715-727.

### APPENDIX A PERFORMANCE STATUS CRITERIA

| ECO | ECOG Performance Status Scale | | Carnofsky Performance Scale |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| 0 | Normal activity. Fully active, able to carry on all pre-disease | 100 | Normal, no complaints, no evidence of disease. |
| U | performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| 1 | to carry out work of a light or sedentary nature ( <i>e.g.</i> , light housework, office work). | 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| | any work activities. Up and about more than 50% of waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. | 40 | Disabled, requires special care and assistance. |
| S | | 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| 4 | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |

# APPENDIX B FORMULA TO ESTIMATE RENAL FUNCTION USING SERUM CREATININE

Formulas to estimate renal function using serum creatinine provided by the NCI's Investigational Drug Steering Committee (IDSC) Pharmacological Task Force in table below.

 Estimated glomerular filtration rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) (Levey et al., 2009).

#### Formulae:

| Race and<br>Sex<br>Black | Serum Creatinine (SCr), | Equation |
|---|---|---|
| Female | ≤62 (≤0.7)<br>>62 (>0.7) | GFR = $166 \times (SCr/0.7)^{-0.329} \times (0.993)^{Age}$<br>GFR = $166 \times (SCr/0.7)^{-1.209} \times (0.993)^{Age}$ |
| Male<br>White or | ≤80 (≤0.9)<br>>80 (>0.9) | GFR = $163 \times (SCr/0.9)^{-0.411} \times (0.993)^{Age}$<br>GFR = $163 \times (SCr/0.9)^{-1.209} \times (0.993)^{Age}$ |
| other | | |
| Female | ≤62 (≤0.7)<br>>62 (>0.7) | GFR = $144 \times (SCr/0.7)^{-0.329} \times (0.993)^{Age}$<br>GFR = $144 \times (SCr/0.7)^{-1.209} \times (0.993)^{Age}$ |
| Male | ≤80 (≤0.9)<br>>80 (>0.9) | GFR = $141 \times (SCr/0.9)^{-0.411} \times (0.993)^{Age}$<br>GFR = $141 \times (SCr/0.9)^{-1.209} \times (0.993)^{Age}$ |

SCr in mg/dL; Output is in mL/min/1.73 m<sup>2</sup> and needs no further conversions.

2. eGFR using the Modification of Diet in Renal Disease (MDRD) Study (Levey et al., 2006).

$$175 \text{ x SCr}^{-1.154} \times \text{age}^{-0.203} \times 0.742$$
 (if female)  $\times$  1.212 (if black) Output is in mL/min/1.73 m<sup>2</sup> and needs no further conversions.

3. Estimated creatinine clearance (ClCr) by the Cockcroft-Gault (C-G) equation (Cockcroft and Gault, 1976).

$$CLcr (mL/min) = \frac{[140 - age (years)] \times weight (kg)}{72 \times serum \ creatinine \ (mg/dL)} \{ \times 0.85 \ for \ female \ patients \}$$

Followed by conversion to a value normalized to 1.73 m<sup>2</sup> with the patient's body surface area (BSA).

#### References

- Levey, A.S., L.A. Stevens, C.H. Schmid, et al. (2009). A new equation to estimate glomerular filtration rate. Ann Inter Med. 150:604-612.
- Levey, A.S., J. Coresh, T. Greene, et al. (2006). Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 145:247-254.
- 3. Cockcroft, D.W. and M.H. Gault. (1976). Prediction of creatinine clearance from serum creatinine. *Nephron.* 16:31-41.

### APPENDIX C PATIENT CLINICAL TRIAL WALLET CARD



#### APPENDIX D PRE-BIOPSY ASSESSMENT

A pre-biopsy lesion assessment can increase trial safety and efficiency. By agreement between all investigators, an attempt at biopsy will be made if the clinical trial team determines that a biopsy poses minimal relative risk, provides potential clinical gain to the participant, and will likely yield sufficient tissue for analysis.

Pre-biopsy assessments will be reported and tracked through a trial-specific CRF within the CTEP Medidata Rave system. Additional information can be found in the Investigational Radiology SOP available at:

https://ctep.cancer.gov/initiativesPrograms/docs/ETCTN IR Research Biopsy SOP.pdf.

**Individual Patient Pre-Biopsy Assessment.** IR co-investigators are encouraged to apply this pre-biopsy scoring and correlation system to assist in the determination of biopsy appropriateness.

- IR co-investigators assign a subjective score of 1-3 based on likelihood of success due to lesion characteristics.
  - 1. Biopsy should not be done
    - A. Due to safety concerns
    - B. Due to lack of suitable lesion for biopsy
  - 2. Uncertainty about success
    - A. Due to access path to lesion
    - B. Due to lesion characteristics
  - 3. Likely successful
- Lesion characteristics to be considered
  - Size (small) (<2 cm)
  - Location/path to lesion
  - Morphologic features (necrosis, sub-solid, sclerosis, ill-defined/infiltrative)
  - PET (+/-), avidity
  - Organ/site (sclerotic bone is low yield; fine needle aspiration to be used)

NCI Protocol #: 10315

Version Date: November 25, 2024

### APPENDIX E PATIENT MEDICATION DIARY

| CTEP-assigned Protocol # 10315 |
|--------------------------------|
| Local Protocol # TBD |

| | PATIENT'S MEDICATION DIARY – XL184 (cab | ozantinib) – For Cycles 1-4 |
|---|---|---|
| Today's date: | | Agent: XL184 (cabozantinib) |
| <b>Patient Name:</b> | (initials acceptable) | Patient Study ID: |

#### INSTRUCTIONS TO THE PATIENT:

- 1. Complete one form for each cycle.
- 2. You will take your dose of XL184 (cabozantinib) at the same time each day:
  - $\square$  2 (20 mg) tablets every day; (or)  $\square$  1 (20 mg) tablet every day; (or)  $\square$  1 (20 mg) tablet every other day.
  - You should swallow the tablets as a whole. **Do not crush or chew**. You should take XL184 (cabozantinib) on an empty stomach, and at least 2 hours after and 1 hour before eating.
- 3. Store XL184 (cabozantinib) tablets in the original bottle and not in weekly pill boxes. Record the date, the number of tablets you took, and when you took them.
- 4. If you forget to take a dose at the scheduled time, you can still take that dose as long as it is within 12 hours of the scheduled time. You should not take the missed dose if it is within 12 hours of your next scheduled dose. Take your next dose at the regularly scheduled time.
- 5. If you vomit after taking a dose, do not retake the dose. Take the next dose at the regularly scheduled time.
- 6. Notify your doctor at the first sign of poorly formed or loose stools, or an increased frequency of bowel movements. Loperamide (Imodium) should be kept on hand and should be taken as recommended by your doctor.
- 7. If you have any comments or notice any side effects, please record them in the Comments column.

8. Please return the forms to your physician when you go for your next appointment.

| Day | | ate | What time was dose taken? | | Comments |
|---|---|---|---|---|---|
| 1. | | | | | |
| 2. | | | | | |
| 3. | | | | | |
| 4. | | | | | |
| 5. | | | | | |
| 6. | | | | | |
| 7. | | | | | |
| 8. | | | | | |
| 9. | | | | | |
| 10. | | | | | |
| 11. | | | | | |
| 12. | | | | | |
| 13. | | | | | |
| 14. | | | | | |
| 15. | | | | | |
| 16. | | | | | |
| 17. | | | | | |
| 18. | | | | | |
| 19. | | | | | |
| 20. | | | | | |
| 21. | <u> </u> | O 001 | | | |
| Phy | | | will complete this section: | | |
| | | | ient started protocol treatment | | |
| | | | ient was removed from study | | |
| | | | planned total daily dose | | |
| | | | mber of pills taken this month (e | | |
| | 5. ] | rnysicia: | n/Nurse/Data Manager's Signatu | ıre | |

| Patient's signature: |
|----------------------|
| _ |

NCI Protocol #: 10315

Version Date: June 3, 2025

CTEP-assigned Protocol # 10315 Local Protocol # TBD

| PATIENT'S MEDICAT | ION DIARY – XL184 (cabozantinib) – For Cycles 5 and beyond |
|---|---|
| Today's date: | Agent: XL184 (cabozantinib) |
| Patient Name: | (initials acceptable) Patient Study ID: |

#### INSTRUCTIONS TO THE PATIENT:

- 5. Complete one form for each cycle.
- 6. You will take your dose of XL184 (cabozantinib) at the same time each day:
  - □ 2 (20 mg) tablets every day; (or) □ 1 (20 mg) tablet every day; (or) □ 1 (20 mg) tablet every other day.
  - You should swallow the tablets as a whole. **Do not crush or chew**. You should take XL184 (cabozantinib) on an empty stomach, and at least 2 hours after and 1 hour before eating.
- 7. Store XL184 (cabozantinib) tablets in the original bottle and not in weekly pill boxes. Record the date, the number of tablets you took, and when you took them.
- 8. If you forget to take a dose at the scheduled time, you can still take that dose as long as it is within 12 hours of the scheduled time. You should not take the missed dose if it is within 12 hours of your next scheduled dose. Take your next dose at the regularly scheduled time.
- 9. If you vomit after taking a dose, do not retake the dose. Take the next dose at the regularly scheduled time.
- 10. Notify your doctor at the first sign of poorly formed or loose stools, or an increased frequency of bowel movements. Loperamide (Imodium) should be kept on hand and should be taken as recommended by your doctor.
- 11. If you have any comments or notice any side effects, please record them in the Comments column.
- 12. Please return the forms to your physician when you go for your next appointment.

| Day | Date | What time was dose taken? | | |
|-----|------|-----------------------------|--------------------|----------|
| 1. | Dutt | THE UNITED THE WOSE CARCILL | " of tubicts taken | Commency |
| 2. | | | | |
| 3. | | | | |
| 4. | | | | |
| 5. | | | | |
| 6. | | | | |
| 7. | | | | |
| 8. | | | | |
| 9. | | | | |
| 10. | | | | |
| 11. | | | | |
| 12. | | | | |
| 13. | | | | |
| 14. | | | | |
| 15. | | | | |
| 16. | | | | |
| 17. | | | | |
| 18. | | | | |
| 19. | | | | |
| 20. | | | | |
| 21. | | | | |
| 22. | | | | |
| 23. | | | | |
| 24. | | | | |
| 25. | | | | |
| 26. | | | | |
| 27. | | | | |
| 28. | | | | |

| BATCH | INITIALS: | DATE: |
|-------|-----------|-------|

| INSTR | UCTION | OT 2V | THE | PATIENT: |
|-------|--------|-------|-----|----------|

- 5. Complete one form for each cycle.
- 6. You will take your dose of XL184 (cabozantinib) at the same time each day:
  - $\square$  2 (20 mg) tablets every day; (or)  $\square$  1 (20 mg) tablet every day; (or)  $\square$  1 (20 mg) tablet every other day. You should swallow the tablets as a whole. **Do not crush or chew**. You should take XL184 (cabozantinib) on an empty stomach, and at
- least 2 hours after and 1 hour before eating. 7. Store XL184 (cabozantinib) tablets in the original bottle and not in weekly pill boxes. Record the date, the number of tablets you took, and when you took them.
- 8. If you forget to take a dose at the scheduled time, you can still take that dose as long as it is within 12 hours of the scheduled time. You should not take the missed dose if it is within 12 hours of your next scheduled dose. Take your next dose at the regularly scheduled time.
- 9. If you vomit after taking a dose, do not retake the dose. Take the next dose at the regularly scheduled time.
- 10. Notify your doctor at the first sign of poorly formed or loose stools, or an increased frequency of bowel movements. Loperamide (Imodium) should be kept on hand and should be taken as recommended by your doctor.
- 11. If you have any comments or notice any side effects, please record them in the Comments column.

| 12. P | lease re | eturn the fo | orms to your physician when you go | for your next appoint | ment. |
|---|---|---|---|---|---|
| Day | D | <b>Date</b> | What time was dose taken? | # of tablets taken | Comments |
| Phys | ician' | s Office v | will complete this section: | | |
| | 1. | Date pati | ient started protocol treatment | | |
| | 2. | Date pati | ient was removed from study | | |
| | 3. | Patient's | planned total daily dose | | |
| | 4. | Total nu | mber of pills taken this month (e | ach size) | |
| | 5. | Physician | n/Nurse/Data Manager's Signatu | ire | |

| ıy | Date | What time was dose taken? | # of tablets taken | Comments |
|---|---|---|---|---|
| hysiciai | n's Office | will complete this section: | | |
| 1. | Date pat | ient started protocol treatment | | |
| 2. | Date pat | ient was removed from study | | |
| 3. | Patient's | planned total daily dose | | |
| 4. | Total nu | mber of pills taken this month (e | each size) | |
| 5. | Physicia | n/Nurse/Data Manager's Signatu | ure | |

| BATCH | INITIALS: | DATE: |
|-------|-----------|-------|

NCI Protocol #: 10315

Version Date: November 25, 2024

APPENDIX F: NIVOLUMAB AND IPILIMUMAB MANAGEMENT ALGORITHMS FOR ENDOCRINOPATHY,

GASTROINTESTINAL, HEPATIC, NEUROLOGICAL, PULMONARY, RENAL, AND SKIN

ADVERSE EVENTS

## **Endocrinopathy Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue immuno-oncology (I-O) therapy. Consider visual field testing, endocrinology consultation, and imaging.



## GI Adverse Event Management Algorithm

Rule out non-inflammatory causes. If non-inflammatory cause is identified, treat accordingly and continue I-O therapy. Opiates/narcotics may mask symptoms of perforation. Infliximab should not be used in cases of perforation or sepsis.



# **Hepatic Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy. Consider imaging for obstruction.



<sup>\*</sup>I-O therapy may be delayed rather than discontinued if AST/ALT ≤ 8 x ULN and T.bili ≤ 5 x ULN.

<sup>\*\*</sup>The recommended starting dose for grade 4 hepatitis is 2 mg/kg/day methylprednisolone IV.

# **Neurological Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy.



# **Pulmonary Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy. Evaluate with imaging and pulmonary consultation.



# Renal Adverse Event Management Algorithm

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy



# Skin Adverse Event Management Algorithm

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy.

